A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Official Title:

Controlled Pilot and Dose-Ranging Study of GDC-0853 in Patients With Refractory Chronic Spontaneous Urticaria (CSU)

NCT Number: NCT03137069

**Document Date:** Protocol Version 4: 09-August-2018

#### **PROTOCOL**

TITLE: A PHASE II, MULTICENTER, RANDOMIZED,

DOUBLE-BLIND, PLACEBO-CONTROLLED PILOT AND DOSE-RANGING STUDY OF GDC-0853 IN PATIENTS WITH REFRACTORY CHRONIC

**SPONTANEOUS URTICARIA (CSU)** 

PROTOCOL NUMBER: GS39684

**VERSION NUMBER:** 4

**EUDRACT NUMBER:** 2016-004624-35

**TEST PRODUCT:** Fenebrutinib (GDC-0853, RO7010939)

**MEDICAL MONITOR:** , M.D.

**SPONSOR:** Genentech, Inc.

**DATE FINAL:** Version 1: 13 December 2016

Version 2 (Germany Only): 11 April 2017

Version 3: 19 December 2017

Version 4: See electronic date stamp below.

FINAL PROTOCOL APPROVAL

**Approver's Name** 



**Date and Time (UTC)** 09-Aug-2018 23:42:38

#### **CONFIDENTIAL**

The information contained in this document, especially any unpublished data, is the property of Genentech, Inc. (or under its control) and therefore is provided to you in confidence as an investigator, potential investigator, or consultant, for review by you, your staff, and an applicable Ethics Committee or Institutional Review Board. It is understood that this information will not be disclosed to others without written authorization from Genentech except to the extent necessary to obtain informed consent from persons to whom the drug may be administered.

# PROTOCOL AMENDMENT, VERSION 4: RATIONALE

Protocol GS39684 has been amended to allow patients the option to enter an open-label extension (OLE) Study GS40868 after completing the 8-week treatment period. Language has been updated throughout the protocol to include the OLE (Sections 3.1, 3.1.2, and 4.3.2.1 and Appendix 1).

The following additional changes have been made:

- The name of the study drug has been updated from GDC-0853 to fenebrutinib throughout the document.
- The Medical Monitor has changed.
- General enrollment update for subjects who received fenebrutinib or placebo (Section 1.2.3).
- Safety data regarding hepatotoxicity has been updated (Section 1.2.3, 1.3.4, and 5.1.1.6).
- Clarification regarding the use of rescue medication (Section 3.1).
- Clarification of contradictory language regarding tubal ligation since bilateral tubal ligation is an example of a contraceptive method with a failure rate of < 1% per year (Section 4.1.1).
- The inclusion criterion that women must refrain from donating eggs during the treatment period and for at least 4 weeks after the last dose of study drug has been added (Section 4.1.1)
- Clarification of fasting before morning clinic visits (Section 4.3.2.1)
- Bilastine dose range has been updated based on daily-recommended dose of 20 mg (Section 4.3.2.3).
- Recommendations have been updated regarding the maximum dose of several lipid-lowering agents (statins) that are metabolized by CYP3A (simvastatin, lovastatin) and/or transported by BCRP (rosuvastatin, atorvastatin), and thus may be affected by drug-drug interaction with fenebrutinib (Section 4.4.2.2 and Appendix 5).
- Clarification regarding the effect of ethinyl estradiol with fenebrutinib has been added (Section 4.4.2.3).
- Clarification regarding the use of prohibited therapies and corticosteroids for exacerbations has been added (Section 4.4.3).
- Eligibility criteria for re-screening have been clarified (Section 4.5.2.2).
- Added language to clarify use of samples after withdrawal of patient consent (Section 4.5.7).
- Contradictory language between Section 4.5.8 and the Schedule of Activities regarding electrocardiograms has been corrected.
- Clarification of the UAS7 definition (Section 4.5.9.2).

- Additional information around infections has been added (Section 5.1.1.1).
- Additional information around bleeding has been added (Section 5.1.1.3).
- Additional information around gastrointestinal effects has been added (Section 5.1.1.5).
- Language has been revised to account for the fact that some sites may not allow follow-up on partner pregnancies (Section 5.4.3.2).
- Language has been added for consistency with Roche's current data retention policy and to accommodate more stringent local requirements (if applicable) (Section 7.6).
- The process for reviewing and handling protocol deviations has been updated per internal standard operating procedures (Section 9.2).

Additional minor changes have been made to improve clarity and consistency. Substantive new information appears in italics. This amendment represents cumulative changes to the original protocol.

## **TABLE OF CONTENTS**

| PR | OTOCOL AC | CEPTANCE FORM | 11 |
|---|---|---|---|
| PR | OTOCOL SY | NOPSIS | 12 |
| 1. | BACKGRO | UND | 25 |
| | 1.1 | Background on Chronic Spontaneous Urticaria | 25 |
| | 1.2 | Background on Bruton's Tyrosine Kinase and fenebrutinib | 26 |
| | 1.2.1 | Bruton's Tyrosine Kinase | 26 |
| | 1.2.2 | Nonclinical Experience with Fenebrutinib | 27 |
| | 1.2.3 | Clinical Experience with Fenebrutinib | 28 |
| | 1.3 | Study Rationale and Benefit-Risk Assessment | 30 |
| | 1.3.1 | Infections | 31 |
| | 1.3.2 | Bleeding | 31 |
| | 1.3.3 | Cytopenias | 31 |
| | 1.3.4 | Hepatotoxicity | 32 |
| | 1.3.5 | Cardiovascular Effects | 32 |
| | 1.3.6 | Malignancy | 32 |
| 2. | OBJECTIVE | ES AND ENDPOINTS | 33 |
| 3. | STUDY DE | SIGN | 34 |
| | 3.1 | Description of the Study | 34 |
| | 3.1.1 | Internal Monitoring Committee | |
| | 3.1.2 | Open-Label Extension Study GS40868 | 38 |
| | 3.2 | End of Study and Length of Study | 38 |
| | 3.3 | Rationale for Study Design | 38 |
| | | | 38 |
| | 3.3.2 | Rationale for Patient Population | 39 |
| | 3.3.3 | Rationale for Control Group | 40 |
| | | | 40 |
| | 3.3.5 | Rationale for Pharmacokinetic Sample Collection Schedule | 40 |
| | 3.3.6 | Rationale for Efficacy Endpoints | 40 |

| 4. | MATERIALS | AND METHODS | 41 |
|---|---|---|---|
| | 4.1 | Patients | 41 |
| | 4.1.1 | Inclusion Criteria | 41 |
| | 4.1.2 | Exclusion Criteria | 43 |
| | 4.2 | Method of Treatment Assignment and Blinding | 46 |
| | 4.2.1 | Randomization and Blinding | 46 |
| | 4.2.2 | Unblinding | 47 |
| | 4.3 | Study Treatment | 48 |
| | 4.3.1 | Formulation, Packaging, and Handling | 48 |
| | 4.3.1.1 | Fenebrutinib and Placebo | 48 |
| | 4.3.1.2 | Background Therapy: Standard-of-Care H1 Antihistamines for CSU | 48 |
| | 4.3.2 | Dosage, Administration, and Compliance of Fenebrutinib and Placebo | 48 |
| | 4.3.2.1 | Fenebrutinib and Placebo Dose and Administration | 48 |
| | 4.3.2.2 | Fenebrutinib and Placebo Compliance | 49 |
| | 4.3.2.3 | Background Therapy: Standard-of-Care H1 Antihistamines for CSU | 50 |
| | 4.3.3 | Investigational Medicinal Product Accountability | 50 |
| | 4.3.4 | Post-Trial Access to Fenebrutinib | 51 |
| | 4.4 | Concomitant Therapy and Additional Restrictions | 51 |
| | 4.4.1 | Permitted Therapy | 51 |
| | 4.4.2 | Cautionary Therapy | 51 |
| | 4.4.2.1 | Acid-Reducing Agents | 51 |
| | 4.4.2.2 | Statins | 52 |
| | 4.4.2.3 | CYP3A and BCRP-Mediated Drug Interactions | 52 |
| | 4.4.3 | Prohibited Therapy | 54 |
| | 4.4.3.1 | Live or Attenuated Vaccinations | 54 |
| | 4.4.4 | Prohibited Food | 54 |
| | 4.4.5 | Additional Restrictions | 54 |
| | 4.5 | Study Assessments | 54 |
| | 4.5.1 | Informed Consent Forms and Screening Log | 54 |
| | 4.5.2 | Eligibility at Screening | 55 |

| | 4.5.2.1 | Retesting: Laboratory Inclusion/Exclusion | 55 |
|---|---|---|---|
| | 4.5.2.2 | Re-screening | 55 |
| | 4.5.3 | Medical History and Demographic Data | 55 |
| | 4.5.4 | Physical Examinations | 55 |
| | 4.5.5 | Vital Signs | 56 |
| | 4.5.6 | FricTest | 56 |
| | 4.5.7 | Laboratory, and Other Biological Samples. | 56 |
| | 4.5.8 | Electrocardiograms | 58 |
| | 4.5.9 | Patient-Reported Outcomes | 59 |
| | 4.5.9.1 | Urticaria Patient Daily eDiary | 59 |
| | 4.5.9.2 | Urticaria Activity Score | 60 |
| | | | 60 |
| | | | 60 |
| | 4.6 | Patient, Treatment, Study, and Site Discontinuation | 61 |
| | 4.6.1 | Patient Discontinuation | 61 |
| | 4.6.2 | Study Treatment Discontinuation | 62 |
| | 4.6.3 | Study and Site Discontinuation | 62 |
| 5. | ASSESSME | NT OF SAFETY | 63 |
| | 5.1 | Safety Plan | 63 |
| | 5.1.1 | Safety Plan for Potential Risks Associated with Fenebrutinib | 63 |
| | 5.1.1.1 | Infections | 63 |
| | 5.1.1.2 | Vaccinations | 65 |
| | 5.1.1.3 | Bleeding | 65 |
| | 5.1.1.4 | Cytopenias | 66 |
| | 5.1.1.5 | Gastrointestinal Effects | 67 |
| | 5.1.1.6 | Hepatotoxicity | 67 |
| | 5.1.1.7 | Cardiovascular Effects | 68 |
| | 5.1.1.8 | Vascular Inflammation | 69 |
| | 5.1.1.9 | Malignancy | 69 |
| | 5.1.2 | Management of Patients Who Experience Specific Adverse Events | 70 |

| 5.1.2.1 | Management of Specific Adverse Events | 70 |
|---|---|---|
| 5.1.2.2 | Management of Increases in QT Interval | 71 |
| 5.2 | Safety Parameters and Definitions | 72 |
| 5.2.1 | Adverse Events | 72 |
| 5.2.2 | Serious Adverse Events (Immediately Reportable to the Sponsor) | 72 |
| 5.2.3 | Adverse Events of Special Interest (Immediately Reportable to the Sponsor) | 73 |
| 5.3 | Methods and Timing for Capturing and Assessing Safety Parameters | 74 |
| 5.3.1 | Adverse Event Reporting Period | 74 |
| 5.3.2 | Eliciting Adverse Event Information | 74 |
| 5.3.3 | Assessment of Severity of Adverse Events | 74 |
| 5.3.4 | Assessment of Causality of Adverse Events | 75 |
| 5.3.5 | Procedures for Recording Adverse Events | 76 |
| 5.3.5.1 | Diagnosis versus Signs and Symptoms | 76 |
| 5.3.5.2 | Adverse Events That Are Secondary to Other Events | 76 |
| 5.3.5.3 | Persistent or Recurrent Adverse Events | 76 |
| 5.3.5.4 | Abnormal Laboratory Values | 77 |
| 5.3.5.5 | Abnormal Vital Sign Values | 78 |
| 5.3.5.6 | Abnormal Liver Function Tests | 78 |
| 5.3.5.7 | Deaths | 78 |
| 5.3.5.8 | Preexisting Medical Conditions | 79 |
| 5.3.5.9 | Lack of Efficacy or Worsening of Chronic Spontaneous Urticaria | 79 |
| 5.3.5.10 | Hospitalization or Prolonged Hospitalization | 79 |
| 5.3.5.11 | Adverse Events Associated with an Overdose or Error in Drug Administration | 80 |
| 5.3.5.12 | Patient-Reported Outcome Data | 80 |
| 5.4 | Immediate Reporting Requirements from Investigator to Sponsor | 80 |
| 5.4.1 | Emergency Medical Contacts | |
| 5.4.2 | Reporting Requirements for Serious Adverse Events and Adverse Events of Special Interest | |

| | 5.4.2.1 | Events That Occur prior to Study Drug Initiation | 81 |
|---|---|---|---|
| | 5.4.2.2 | Events That Occur after Study Drug Initiation | 81 |
| | 5.4.3 | Reporting Requirements for Pregnancies | 82 |
| | 5.4.3.1 | Pregnancies in Female Patients | 82 |
| | 5.4.3.2 | Pregnancies in Female Partners of Male Patients | 82 |
| | 5.4.3.3 | Congenital Anomalies/Birth Defects and Abortions | 83 |
| | 5.5 | Follow-Up of Patients after Adverse Events | 83 |
| | 5.5.1 | Investigator Follow-Up | 83 |
| | 5.5.2 | Sponsor Follow-Up | 83 |
| | 5.6 | Adverse Events That Occur after the Adverse Event Reporting Period | 83 |
| | 5.7 | Expedited Reporting to Health Authorities,<br>Investigators, Institutional Review Boards, and<br>Ethics Committees | 84 |
| 6. | STATISTICA | AL CONSIDERATIONS AND ANALYSIS PLAN | 84 |
| | 6.1 | Determination of Sample Size | 84 |
| | 6.1.1 | Cohort 1: Pilot Assessment | 84 |
| | 6.1.2 | Cohort 2: Dose-Ranging Assessment | 85 |
| | 6.2 | Summaries of Conduct of Study | 85 |
| | 6.3 | Summaries of Treatment Group Comparability | 86 |
| | 6.4 | Efficacy Analyses | 86 |
| | 6.4.1 | Primary Efficacy Endpoint | 86 |
| | 6.4.2 | Secondary Efficacy Endpoints | 87 |
| | 6.4.3 | Exploratory Efficacy Endpoints | 87 |
| | 6.5 | Safety Analyses | 88 |
| | 6.6 | Pharmacokinetic Analyses | 88 |
| | | | 88 |
| | 6.8 | Interim Analysis | 89 |
| | 6.8.1 | Cohort 1: Planned Interim Analysis | 89 |
| | 6.8.2 | Cohort 2: Optional Interim Analysis | 89 |
| 7. | DATA COLL | LECTION AND MANAGEMENT | 89 |
| | 7.1 | Data Quality Assurance | 89 |
| | 7.2 | Electronic Case Report Forms | 90 |

| | 7.3 | Electronic Patient-Reported Outcome Data | 90 |
|---|---|---|---|
| | 7.4 | Source Data Documentation | 90 |
| | 7.5 | Use of Computerized Systems | 91 |
| | 7.6 | Retention of Records | 91 |
| 8. | ETHICA | AL CONSIDERATIONS | 92 |
| | 8.1 | Compliance with Laws and Regulations | 92 |
| | 8.2 | Informed Consent | 92 |
| | 8.3 | Institutional Review Board or Ethics Committee | 93 |
| | 8.4 | Confidentiality | 93 |
| | 8.5 | Financial Disclosure | 94 |
| 9. | | DOCUMENTATION, MONITORING, AND STRATION | 94 |
| | 9.1 | Study Documentation | 94 |
| | 9.2 | Protocol Deviations | 94 |
| | 9.3 | Site Inspections | 94 |
| | 9.4 | Administrative Structure | 95 |
| | 9.5 | Publication of Data and Protection of Trade Secrets | 95 |
| | 9.6 | Protocol Amendments | 96 |
| 10. | REFER | ENCES | 97 |
| | | LIST OF TABLES | |
| Tab | ole 1<br>ole 2 | Objectives and Corresponding Endpoints Twice Daily Patient Assessment of CSU Disease Activity | 33 |
| Tub | 10 2 | (UAS Scale) | |
| Tab | le 3 | Fenebrutinib Dosing Regimen by Treatment Arm (Cohort 2) | 49 |
| | | | 57 |
| Tab | le 5 | Guidelines for Management of Patients Who Experience Specific Adverse Events | 70 |
| Tab | le 6 | Adverse Event Severity Grading Scale | 75<br>75 |
| Tab | le 7 | Causal Attribution Guidance | |

# **LIST OF FIGURES**

| Figure 1 | Study Schema | 37 |
|---|---|---|
| | LIST OF APPENDICES | |
| Appendix 1<br>Appendix 2 | Schedule of Activities (Cohorts 1 and 2) | 101 |
| • | Contraception | 106 |
| Appendix 3 | Urticaria Patient Daily eDiary | 108 |
| | | 113 |
| Appendix 5 | Concomitant Medications (Including Foods and Herbal | |
| | Products) | 114 |

## PROTOCOL ACCEPTANCE FORM

| TITLE: | A PHASE II, MULTICENTER, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED PILOT AND DOSE-RANGING STUDY OF GDC-0853 IN PATIENTS WITH REFRACTORY CHRONIC SPONTANEOUS URTICARIA (CSU) |
|---|---|
| PROTOCOL NUMBER: | GS39684 |
| VERSION NUMBER: | 4 |
| EUDRACT NUMBER: | 2016-004624-35 |
| TEST PRODUCT: | Fenebrutinib (GDC-0853, RO7010939) |
| MEDICAL MONITOR: | , M.D. |
| SPONSOR: | Genentech, Inc. |
| I agree to conduct the stud | dy in accordance with the current protocol. |
| Principal Investigator's Name | (print) |
| Principal Investigator's Signatu | ure Date |

Please return a copy of the signed form as instructed by the CRO. Please retain the original for your study files.

#### PROTOCOL SYNOPSIS

TITLE: A PHASE II, MULTICENTER, RANDOMIZED, DOUBLE-BLIND,

PLACEBO-CONTROLLED PILOT AND DOSE-RANGING STUDY OF GDC-0853 IN PATIENTS WITH REFRACTORY CHRONIC

**SPONTANEOUS URTICARIA (CSU)** 

PROTOCOL NUMBER: GS39684

VERSION NUMBER: 4

**EUDRACT NUMBER**: 2016-004624-35

**TEST PRODUCT:** Fenebrutinib (GDC-0853, RO7010939)

PHASE: Phase II

INDICATION: Refractory Chronic Spontaneous Urticaria (CSU)

**SPONSOR:** Genentech, Inc.

#### **Objectives and Endpoints**

This pilot and dose-ranging study will evaluate the efficacy, safety, and pharmacokinetics of fenebrutinib compared with placebo in patients with chronic spontaneous urticaria (CSU) refractory to anti-histamines (up to 4 times the approved dose per local treatment guidelines). Specific objectives and corresponding endpoints for the study are outlined below.

#### **Objectives and Corresponding Endpoints**

| Objectives | Corresponding Endpoints |
|---|---|
| Efficacy Objective: | |
| To evaluate the efficacy of fenebrutinib | Primary Endpoint: |
| compared with placebo in patients with | Change from baseline in the UAS7 at Day 57 (Week 8) |
| CSU who are refractory to anti-histamines | Secondary Endpoints: |
| anti-nistanines | <ul> <li>Proportion of patients who are well controlled (UAS7 ≤ 6) at<br/>Day 57</li> </ul> |
| | Change from baseline in the UAS7 at Day 29 (Week 4) |
| | Exploratory Endpoints: |
| | Change from baseline in the weekly itch score at Day 29 |
| | Change from baseline in the weekly itch score at Day 57 |
| | Change from baseline in the weekly hives score at Day 57 |
| | <ul> <li>Proportion of patients who are well controlled (UAS7 ≤ 6) at<br/>Day 29</li> </ul> |
| | <ul> <li>Proportion of patients who achieve complete response<br/>(UAS7 = 0) at Day 29</li> </ul> |
| | <ul> <li>Proportion of patients who achieve complete response<br/>(UAS7 = 0) at Day 57</li> </ul> |
| | <ul> <li>Proportion of patients achieving MID in UAS7 at Day 57<br/>(reduction from baseline ≥ 11 points)</li> </ul> |
| | <ul> <li>Proportion of patients achieving MID in the weekly itch score at<br/>Day 57 (reduction from baseline ≥ 5 points)</li> </ul> |

#### Objectives and Corresponding Endpoints (Continued)

| Objectives | Corresponding Endpoints |
|---|---|
| | Exploratory Endpoints (Continued): |
| | Time to achieving MID in UAS7 (reduction from baseline ≥ 11 points) |
| Safety Objective: | |
| To evaluate the safety of fenebrutinib<br>compared with placebo | The nature, frequency, timing, and severity of adverse events Change from baseline in targeted vital signs, physical examination findings, ECGs, and clinical laboratory results following fenebrutinib administration |
| Pharmacokinetic Objective: | |
| To characterize the pharmacokinetics of fenebrutinib in patients | Plasma concentrations of fenebrutinib at specified timepoints |

AUC<sub>0-t</sub> = area under the concentration–time curve from time 0 to time t; BTK= Bruton's tyrosine kinase CL/F = apparent clearance; C<sub>max</sub> = maximum concentration observed; C<sub>trough</sub> = steady-state concentration at the end of a dosing interval; CSU = chronic spontaneous urticaria; MID = minimally important difference; PK = pharmacokinetic; t<sub>1/2</sub> = half-life; t<sub>max</sub> = time to maximum concentration; UAS7 = Urticaria Activity Score over 7 days;

#### **Study Design**

#### **Description of Study**

This pilot and dose-ranging study is a multicenter, randomized, double-blind, placebo-controlled, parallel-group study of the efficacy and safety of fenebrutinib as add-on therapy for the treatment of adult patients 18–75 years old who have been diagnosed with CSU and who remain symptomatic despite treatment with H1 antihistamines (including doses up to 4 times the approved dose per local treatment guidelines). The study will consist of two cohorts. Cohort 1

will enroll approximately 45 patients across multiple sites. After screening, eligible patients will be randomly allocated in a 2:1 ratio to receive fenebrutinib 200 mg orally (PO) twice daily (BID) or matching placebo for 8 weeks and will maintain stable doses of standard-of-care H1 antihistamine therapy throughout the study. On the basis of results from an interim analysis of Cohort 1, a dose-ranging cohort, Cohort 2, will be opened and approximately 120 patients will be randomly allocated in a 1:1:1:1 ratio to receive 50 mg PO daily (QD), 150 mg PO QD, 200 mg PO BID of fenebrutinib, or placebo, respectively, for 8 weeks and will maintain stable doses of standard-of-care H1 antihistamine therapy (background therapy) throughout the study. Both cohorts will consist of 3 distinct study periods over a time-period of 14 weeks as outlined below:

Screening period: Day –14 to Day –1

Treatment Period: Day 1 to Day 57 (Week 0 to Week 8)

Follow-Up Period: Day 57 to Day 85 (Week 8 to Week 12)

Patients in both cohorts will have a screening period of approximately 2 weeks to establish their eligibility for the study and baseline symptom scores. For the duration of the screening period, patients must maintain stable doses of their pre-screening combination therapy with standard-of-care H1 antihistamines (i.e., up to 4 times the approved dose per local treatment guidelines). The screening period will consist of visits at Day –14 and Day –7. Patients must meet all of the following criteria to enter the screening period:

- Documented treatment with a regimen that includes standard-of-care H1 antihistamine for CSU at Day -14 and for at least the 3 consecutive days immediately prior to Day -14
- Willing and able to complete a symptom electronic diary (Urticaria Patient Daily eDiary) twice daily throughout the screening period to establish the patient's Urticaria Activity Score over 7 days (UAS7) score.

To be eligible for randomization in both cohorts, for the 7 days prior to randomization, patients must meet all of the following:

- Seven consecutive days of entries in the Urticaria Patient Daily eDiary, and
- UAS7 symptom score of ≥ 16 (range: 0-42)

Only in exceptional circumstances, when information concerning eligibility is outstanding (e.g., delayed laboratory results), will a longer screening period be permitted up to 3 business days. Upon approval from the Medical Monitor, patients may be re-screened or may be retested during the screening period. Circumstances that may permit re-screening or retesting include, but are not limited to, a laboratory test result that does not meet eligibility requirements.

On Day 1, eligible patients in Cohort 1 will be randomly allocated in a 2:1 ratio to receive fenebrutinib 200 mg orally (PO) twice daily (BID) or placebo for 8 weeks. Eligible patients in Cohort 2 will be will be randomly allocated in a 1:1:1:1 ratio to receive 50 mg PO daily (QD), 150 mg PO QD, 200 mg PO BID of fenebrutinib, or placebo, respectively, for 8 weeks. The primary efficacy endpoint will be at Day 57 (Week 8). Throughout the treatment period, patients must maintain stable doses of their pre-randomization H1 antihistamine therapy.

After completion of the 8-week treatment period, all patients in both cohorts will either enter a 4-week safety follow-up period to allow for further characterization of the pharmacokinetics and pharmacodynamics of fenebrutinib, and collection of additional efficacy and safety or they will have the opportunity to participate in the open-label extension Study GS40868. During safety follow-up period, no study treatment will be given; patients must maintain stable doses of their pre-randomization CSU H1 antihistamine treatment (background therapy). In the safety follow-up period, patients may add up to one additional H1 antihistamine therapy in case of worsened symptoms. The goal of allowing additional H1 antihistamine therapy after the treatment period is to reduce patient dropout for improved safety evaluation.

In addition to their daily background therapy, for the duration of the study all patients will be able to use a single approved dose of loratadine (10 mg maximum) or cetirizine (10 mg maximum) within a 24-hour period as rescue medication if symptoms worsen. If a patient needs rescue therapy and is already on background treatment with cetirizine or loratadine, the patient may receive 10 mg more of the same drug only if the total daily dose remains below 4 times the

approved dose. *Otherwise*, the alternate rescue medication *may be used*. Patients should record the use of this medication in their eDiary. Patients receiving proton-pump inhibitors (PPIs) or H2 receptor antagonists (H2RAs) should be stabilized on a regimen beginning at least 2 weeks prior to randomization and continuing throughout the study.

#### **Internal Monitoring Committee**

For Cohort 2, periodic safety reviews and any interim analysis will be performed by the Sponsor's internal monitoring committee (IMC) as outlined in the IMC charter. This committee will be unblinded to treatment assignments and will include Sponsor representatives from the following functions: Clinical Science, Drug Safety, Biostatistics, and Statistical Programming and Analysis. The IMC members will not have direct contact with investigational staff or site monitors. The IMC may decide to unblind the study team to enable decision-making and potential interactions with regulatory bodies. The IMC may invite representatives from other functional areas on an ad-hoc basis when additional expertise is required (e.g., Clinical Pharmacology, Research, etc.) or additional Sponsor scientists to participate in data analyses and review.

At any time during the study, the Sponsor may choose to inactivate and suspend enrollment and further dosing for a given treatment arm (in Cohort 2) or reduce the dose due to safety concerns and as guided by the IMC. In Cohort 2, subsequently enrolled patients will be randomly allocated to the remaining active arms.

#### Open-Label Extension Study GS40868

After completing the 8-week treatment period (at Day 57), eligible patients from Cohort 1 and 2 will have the option to enter the OLE Study GS40868 and receive open-label fenebrutinib treatment. Patients who do not enter the OLE after completing the treatment period will undergo assessments at 4 weeks after the last dose of study drug (safety follow-up).

Patients who completed the treatment period and 4-week safety follow-up period may also enroll in the OLE study if eligible.

#### **Number of Patients**

Approximately 45 patients, aged 18 to 75 years old who have been diagnosed with refractory CSU and who remain symptomatic despite standard-of-care H1 antihistamine (i.e., up to 4 times the approved dose per local treatment guidelines), will be enrolled in Cohort 1. On the basis of results from an interim analysis of Cohort 1, a dose-ranging cohort, Cohort 2, will be opened and approximately 120 patients will be enrolled.

#### **Target Population**

#### Inclusion Criteria

Patients in Cohort 1 and 2 must meet the following criteria for study entry:

- Willing to give written informed consent, adhere to the visit schedules, comply with the study drug regimen, and meet other study requirements
- Aged 18 75 years, inclusive
- Diagnosis of CSU refractory to H1 antihistamines at the time of randomization, as defined by all of the following:
  - The presence of itch and hives for > 6 consecutive weeks at any time prior to enrollment despite current use of H1 antihistamine, consistent with standard of care (i.e., up to 4 times the approved dose per local treatment guidelines) during this time period
  - UAS7 score ≥ 16 during the 7 days prior to randomization (Day 1)
  - Patients must have been on daily stable doses of H1 antihistamine, consistent with standard of care (i.e., up to 4 times the approved dose per local treatment guidelines) treatment for CSU starting at least 3 consecutive days immediately prior to the screening visit through Day 1 and must document current use on all visits.
  - CSU diagnosis for ≥ 6 months
- Willing and able to complete an Urticaria Patient Daily eDiary for the duration of the study

- Completion of 7 days of the Urticaria Patient Daily eDiary entries in the 7 days prior to randomization (7 of 7 days must be completed [i.e., must complete an entry every day] with up to 2 non-consecutive entries missed)
- No evidence of active or latent or inadequately treated infection with tuberculosis (TB) as defined by the following:
  - A negative QuantiFERON-TB-Gold® (QFT) performed at the screening visit or within the 3 months prior to screening (for German sites only: QFT is the preferred test)

If QFT is unavailable, a negative Mantoux purified protein derivative (PPD) skin test as defined by the Centers for Disease Control and Prevention guidelines, may be performed at the screening visit or within the 3 months prior to screening -AND-

Any additional procedures (e.g., chest X-Ray) required per local guidelines to rule out latent or active TB

NOTE: A documented negative screening for TB via the PPD test or a negative QFT within 3 months prior to screening (and if required per local standard of care, a chest X-ray), is sufficient and no further screening with QFT is required.

Patients with a history of Bacille Calmette-Guérin (BCG) vaccination should be screened using the QFT test, only.

- An indeterminate QFT test should be repeated.
- A positive QFT test or two successive indeterminate QFT results should be considered a positive diagnostic TB test.
- An indeterminate QFT test followed by a negative QFT test should be considered a negative diagnostic TB test.
- Only for patients currently receiving PPIs or H2RAs: Treatment must be at a stable dose during the 2 week screening period prior to randomization and with a plan to remain at a stable dose for the duration of the study
- For women of childbearing potential: Agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 4 weeks after the last dose of study drug. Women must refrain from donating eggs during this same period.

A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).

Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, established proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. Women using estrogen-containing hormonal contraceptives as a method of contraception <u>must</u> also use a barrier, such as a male condom, in conjunction with the hormonal contraceptives.

The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception.

• For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm, as defined below:

With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 4 weeks after the last dose of study treatment to avoid exposing the embryo. Men must refrain from donating sperm during this same period.

The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence

(e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception.

#### **Exclusion Criteria**

Patients in Cohort 1 and 2 who meet any of the following criteria will be excluded from study entry:

- Treatment with omalizumab or other monoclonal antibody therapies used to treat CSU within 4 months prior to screening or primary nonresponse to omalizumab
- Use of a non-biologic investigational drug or participation in an investigational study with a non-biologic drug within 30 days prior to study drug administration on Day 1 (or within 5 half-lives of the investigational product, whichever is greater)
- Use of a biologic investigational therapy or participation in an investigational study involving biologic therapy within 90 days or 5 half-lives, whichever is greater, prior to study drug administration on Day 1
- Previous treatment with fenebrutinib or other Bruton's tyrosine kinase (BTK) inhibitors
- · Patients whose urticaria is solely due to physical urticaria
- Other diseases with symptoms of urticaria or angioedema, including urticarial vasculitis, urticaria pigmentosa, erythema multiforme, mastocytosis, hereditary or acquired angioedema, lymphoma, or leukemia
- Atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, or other skin disease associated with itch such as psoriasis
- Routine (daily or every other day during 5 or more consecutive days) doses of the following medications within 30 days prior to screening: systemic or cutaneous (topical) corticosteroids (prescription or over the counter), hydroxychloroquine, methotrexate, cyclosporine, or cyclophosphamide
- Prior utilization of intravenous (IV) steroids for treatment of laryngeal angioedema
- IV immunoglobulin G (IVIG) or plasmapheresis within 30 days prior to screening
- History of anaphylactic shock without clearly identifiable avoidable antigen (e.g., due to food allergy)
- Hypersensitivity to fenebrutinib or any component of the formulation
- Major surgery, within 8 weeks prior to screening or surgery planned prior to end of study (12 weeks after randomization)
- Require any prohibited concomitant medications
- History of live attenuated vaccine within 6 weeks prior to randomization or requirement to receive these vaccinations at any time during study drug treatment
  - Seasonal influenza and H1N1 vaccination is permitted if the inactivated vaccine formulation is administered.
- Evidence of clinically significant cardiac, neurologic, psychiatric, pulmonary, renal, hepatic, endocrine (including uncontrolled diabetes mellitus), metabolic, or gastrointestinal (GI) disease that, in the investigator's opinion, would compromise the safety of the patient, interfere with the interpretation of the study results, or otherwise preclude patient participation.

Any items that are cause for uncertainty must be reviewed with the Medical Monitor.

- Uncontrolled disease states, such as asthma, psoriasis, or inflammatory bowel disease, where flares are commonly treated with oral or parenteral corticosteroids
- History of vasculitis
- Current liver disease
- Any known active infection (with the exception of fungal nail infections or oral herpes)

- History of recurrent bacterial, viral, mycobacterial or fungal infections (defined as >2 similar episodes requiring anti-microbial treatment within the previous 12 months), with the exception of recurrent oral or genital herpes (herpes simplex virus 1/herpes simplex virus 2) or uncomplicated urinary tract infections in females.
- Any history of opportunistic infections that, in the investigator or Sponsor's judgment, would raise safety concerns regarding the patient's participation in the study
- Any major episode of infection requiring hospitalization or treatment with IV antimicrobials within 8 weeks prior to and during screening or treatment with oral antimicrobials within 2 weeks prior to and during screening

Antimicrobials include antifungal, antibacterial, and antiviral agents.

- History of or currently active primary or secondary immunodeficiency, including known history of HIV infection
- Evidence of chronic and/or active hepatitis B or C

Positive hepatitis B surface antigen (HBsAg) or hepatitis C serology (regardless of treatment status)

Positive hepatitis B core antibody (HBcAb)

 History of cancer, including hematologic malignancy and solid tumors, within 10 years before screening

Basal or squamous cell carcinoma of the skin that has been excised and is considered cured and in situ carcinoma of the cervix treated with apparent success by curative therapy > 1 year prior to screening are not exclusionary.

- Women who are pregnant, nursing (breastfeeding), or intending to become pregnant during the study or within 4 weeks after completion of the study
- For women of childbearing potential (including those who have had a tubal ligation): positive serum pregnancy test result at screening or on Day 1.

A serum pregnancy test is needed on Day 1 only if the urine pregnancy test is positive.

- History of alcohol, drug(e.g., tetrahydrocannabinol [THC], marijuana), or chemical abuse within the 12 months prior to screening as determined by the investigator
- Need for systemic anti-coagulation with warfarin, other oral or injectable anti-coagulants, or anti-platelet agents other than non-steroidal anti-inflammatory drugs (NSAIDs), aspirin, and other salicylates
- History of non-gallstone-related pancreatitis or chronic pancreatitis
- History of hospitalizations or transfusion for a GI bleed
- History of cerebrovascular accident (CVA) within 10 years or any history of hemorrhagic CVA
- History of spontaneous intracranial hemorrhage or history of traumatic intracranial hemorrhage within 10 years
- Known bleeding diathesis
- Screening 12-lead ECG that demonstrates clinically relevant abnormalities that may affect patient safety or interpretation of study results, including

QT interval corrected using Fridericia's formula (QTcF) > 440 ms demonstrated by at least two ECGs > 30 minutes apart

History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias such as long QT syndrome and other genetic risk factors (e.g., Brugada syndrome), structural heart disease (e.g., severe left ventricular systolic dysfunction, severe left ventricular hypertrophy), coronary heart disease (symptomatic, or with ischemia demonstrated by diagnostic testing, prior coronary artery bypass grafting, or coronary lesions > 70% diameter stenosis that have not been or cannot be re-vascularized), clinically significant electrolyte abnormalities (e.g., hypokalemia, hypomagnesemia, hypocalcemia), or family history of sudden unexplained death or cardiac ion channel mutations (e.g., congenital long QT syndrome)

- Current treatment with medications that are well known to prolong the QT interval (see https://crediblemeds.org/index.php/login/dlcheck) at doses that have a clinically meaningful effect on QT, as determined by the investigator; the investigator may contact the Sponsor for confirmation if needed
- Current treatment with astemizole, terfenadine, and/or ebastine
- Any condition possibly affecting oral drug absorption (e.g., gastrectomy, clinically significant diabetic gastroenteropathy, or certain types of bariatric surgery such as gastric bypass)
  - Procedures such as gastric banding, that simply divide the stomach into separate chambers, are not exclusionary.
- Any uncontrolled clinically significant laboratory abnormality that would affect safety, interpretation of study data, or the patient's participation in the study
- For German sites only: Subjects who live in detention on court order or on regulatory action as per local and national law (see §40 subSection 1 sentence 3 no. 4 Arzneimittelgesetz).

The following exclusion criteria are based on screening laboratory tests. Laboratory tests may be repeated once during the screening period unless otherwise indicated:

- Creatinine > 1.5 times the upper limit of normal (ULN; may be repeated if 1.5–2×ULN)
- Creatinine clearance < 70 mL/min (may be repeated if 60–69 mL/min) as estimated by the Cockcroft-Gault Equation
- ALT or AST > 1.5 times ULN (may be repeated if 1.5–3 × ULN)
- Total bilirubin > ULN (may be repeated if 1–3 × ULN)
- Hemoglobin < 11 g/dL (may be repeated if 10–10.9 g/dL)</li>
- ANC  $< 1.5 \times 10^9$ /L (may be repeated if  $1.2-1.5 \times 10^9$ /L)
- Platelet count  $< 100 \times 10^9$ /L (may be repeated if  $80-100 \times 10^9$ /L)
- IgG < 500 mg/dL (should not be repeated)</li>
- Abnormalities in hepatic synthetic function tests (e.g., PT, INR, PTT, albumin) judged by the investigator to be clinically significant

#### **End of Study**

The end of this study is defined as the date when all patients have completed the study completion visit or early termination visit or have otherwise been discontinued from the study.

#### Length of Study

The total duration of this study for each subject is approximately 14 weeks, including screening, treatment, and safety follow-up periods.

The total length of the study, from screening of the first patient to the end of the study, is expected to be approximately 19 months.

#### **Investigational Medicinal Products**

The investigational medicinal product for this study is fenebrutinib. For Cohort 1, patients will receive fenebrutinib 200 mg PO BID or placebo for 8 weeks. For Cohort 2, will receive fenebrutinib 50 mg QD, 150 mg QD, 200 mg BID, or placebo for 8 weeks.

#### **Non-Investigational Medicinal Products**

Throughout the treatment period, patients must maintain stable doses of their pre-randomization H1 antihistamine therapy. In addition to their daily background therapy, for the duration of the study all patients will be able to use a single approved dose of loratadine (10 mg maximum) or cetirizine (10 mg maximum) within a 24-hour period as rescue medication if symptoms worsen. If a patient needs rescue therapy and is already on background treatment with cetirizine or loratadine, the patient may receive 10 mg more of the same drug only if the total daily dose remains below 4 times the approved dose. Otherwise, the alternate rescue medication may be used.

#### **Statistical Methods**

#### **Primary Analysis**

The primary efficacy endpoint is the change from baseline in the UAS7 at Day 57 (Week 8).

The Urticaria Activity Score (UAS) is to be recorded twice daily (i.e., morning and evening) using an eDiary that will be provided to each patient. Scores ranging from 0 (none) to 3 (severe) will be entered for each of the two UAS domains consisting of number of wheals (hives) and intensity of pruritis (itch) resulting in a total possible score of 0 to 6. The daily UAS is calculated as the average of the morning and evening scores. When either the morning or evening score is missing, the non-missing UAS for that day (morning or evening) will be used as the daily UAS, and when both the morning and evening UAS are missing, the daily UAS will be deemed missing. The UAS7 is the sum of the daily UAS over the 7 days prior to the time point of interest. The baseline UAS7 will be calculated as the sum of daily UAS values over the week (7 days) prior to Day 1.

When one or more daily UAS values is missing, over the week prior to a timepoint of interest, rules for deriving UAS7 will be as follows:

- If a patient has at least 4 completed daily scores on the UAS (both domains) over the 7 days prior to the time point of interest, the UAS7 will be defined as the average of the available daily scores, multiplied by 7.
- If a patient has fewer than 4 completed daily scores on the UAS over the 7 days prior to the time point of interest, then the UAS7 will be considered missing for that time point.

The primary endpoint will be analyzed using a mixed model for repeated measures model. Additional model covariates will include baseline UAS7 and its interaction with visit. Missing data will be handled by the model under the missing-at-random assumption without need for imputation. As a sensitivity analysis, an analysis of covariance (ANCOVA) model adjusted for country and baseline UAS7 will be fit, and missing Day 57 data will be imputed by last observation carried forward.

## **Determination of Sample Size**

#### **Cohort 1: Pilot Assessment**

The purpose of this cohort is to evaluate the efficacy of fenebrutinib compared with placebo in improving the UAS7. Point and interval estimates of the change from baseline of the UAS7 within each treatment group as well as of the difference in change from baseline of the UAS7 between treatment groups will be presented.

The cohort will enroll approximately 45 patients. Patients will be randomized in a 2:1 ratio to receive treatment with either fenebrutinib or placebo. The sample size of approximately 30 patients in the fenebrutinib arm and 15 patients in the placebo arm provides approximately 80% power to detect an 11-point difference in the UAS7 change from baseline at Day 57 between treatment groups under the following assumptions:

- The absolute change from baseline at Day 57 is normally distributed with a standard deviation of 13.
- Two-sided alpha is 0.10.
- Drop out at Day 57 is 10%, leading to a 10% loss of information.

#### **Cohort 2: Dose-Ranging Assessment**

The purpose of this cohort is estimation and hypothesis generation regarding the dose-ranging effects of fenebrutinib compared with placebo in improving the UAS7. Point and interval estimates of the change from baseline of the UAS7 within each treatment group as well as of the difference in change from baseline of the UAS7 between treatment groups vs placebo will be presented.

The cohort will enroll approximately 120 patients. Patients will be randomly allocated in a 1:1:1:1 ratio to receive treatment with one of three dose levels of fenebrutinib or placebo. The sample size of approximately 30 in each arm provides approximately 90% power to detect an 11-point difference in the UAS7 change from baseline at Day 57 between treatment groups, under the following assumptions:

- The absolute change from baseline at Day 57 is normally distributed with a standard deviation of 13
- Two-sided alpha is 0.10
- Dropout rate at Day 57 is 10%, leading to a 10% loss of information.

The overall sample size may be adjusted depending on the outcome of a planned interim analysis for Cohort 1, which will include an evaluation of these assumptions.

#### **Interim Analysis**

#### **Cohort 1: Planned Interim Analysis**

An interim analysis will be performed after approximately 33 patients have completed their 8–week treatment period. The purpose of this analysis is to assess the efficacy of the 200mg fenebrutinib BID daily arm compared with the placebo, to guide internal decision-making around issues such as ungating of Cohort 2, adequacy of sample sizes for safety and/or efficacy analyses in Cohort 2, or to inform further development decisions. Summaries of safety and efficacy data by treatment groups will be prepared and reviewed by Sponsor personnel who do not have direct contact with investigational staff, monitors, and patients. Further details of the interim analysis will be specified in the data analysis plan (DAP) prior to the conduct of the interim analysis. Access to treatment assignment information will follow the Sponsor's standard procedures.

#### **Cohort 2: Optional Interim Analysis**

Given the hypothesis-generating nature of this study, the Sponsor may choose to conduct up to two interim efficacy analyses. The decision to conduct an optional interim analysis and the timing of the analysis will be documented in the Sponsor's trial master file prior to the conduct of the interim analysis. The interim analysis will be performed and interpreted by members of the IMC. Access to treatment assignment information will follow the Sponsor's standard procedures.

## **LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS**

| Abbreviation | Definition |
|---|---|
| ANCOVA | analysis of covariance |
| AUC | area under the concentration-time curve |
| AUC <sub>0-t</sub> | area under the concentration-time curve from time 0 to time t |
| BCG | Bacille Calmette-Guérin |
| BCR | B-cell receptor |
| BCRP | breast cancer resistance protein |
| BID | twice a day |
| BTK | Bruton's tyrosine kinase |
| $C_{max}$ | maximum observed concentration |
| $C_{\text{trough}}$ | steady-state concentration at the end of a dosing interval |
| CIU | chronic idiopathic urticaria |
| CL/F | apparent clearance |
| CRP | C-reactive protein |
| CSR | clinical study report |
| CSU | chronic spontaneous urticaria |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CVA | cerebrovascular accident |
| DAP | data analysis plan |
| DLAE | dose-limiting adverse events |
| DLT | dose-limiting toxicity |
| EC | Ethics Committee |
| eCRF | electronic Case Report Form |
| EDC | electronic data capture |
| FcεRI | high affinity IgE receptor |
| FDA | Food and Drug Administration |
| GI | gastrointestinal |
| H2RA | H2 receptor antagonist |
| HBcAb | hepatitis B core antibody |
| HBsAg | hepatitis B surface antigen |
| ICH | International Conference on Harmonisation |

| Abbreviation | Definition |
|------------------|--------------------------------------------------|
| IL-1 | interleukin 1 |
| IL-6 | interleukin 6 |
| IMC | Internal monitoring committee |
| IMP | investigational medicinal product |
| IND | Investigational New Drug (application) |
| IRB | Institutional Review Board |
| IV | intravenous |
| IVIG | intravenous immunoglobulin G |
| IxRS | interactive voice or web-based response system |
| LTRA | leukotriene receptor antagonist |
| MAD | multiple-ascending dose |
| MID | minimally important difference |
| mITT | modified intent-to-treat |
| MMRM | mixed model for repeated measures |
| NCI | National Cancer Institute |
| NOAEL | no observed adverse effect level |
| NSAID | non-steroidal anti-inflammatory drug |
| PD | pharmacodynamic |
| PK | pharmacokinetic |
| PO | by mouth, orally |
| PPD | Purified Protein Derivative |
| PPI | proton-pump inhibitor |
| PRO | patient-reported outcome |
| QD | once a day |
| QFT | QuantiFERON-TB-Gold |
| QTcF | QT interval corrected using Fridericia's formula |
| RA | rheumatoid arthritis |
| SAD | single-ascending dose |
| SLE | systemic lupus erythematosus |
| t <sub>1/2</sub> | half-life |
| t <sub>max</sub> | time to maximum concentration |
| ТВ | tuberculosis |
| THC | tetrahydrocannabinol |
| TNF-α | tumor necrosis factor alpha |
| UAS | Urticaria Activity Score |
| UAS7 | Urticaria Activity Score over 7 days |

| Abbreviation | Definition |
|--------------|-----------------------------|
| XLA | X-linked agammaglobulinemia |

## 1. <u>BACKGROUND</u>

#### 1.1 BACKGROUND ON CHRONIC SPONTANEOUS URTICARIA

Chronic spontaneous urticaria (CSU, also referred to as chronic idiopathic urticaria [CIU]) is defined by the presence of wheals (hives), angioedema, or both for at least 6 weeks without an obvious cause (Greaves 2003). Previous estimates of the prevalence of CSU were approximately 0.1%, which persists in 20% of CSU patients 2 decades after diagnosis (Greaves 2000; Saini 2014). More recent evidence indicates that the point prevalence of the disease is approximately 1% (Maurer et al. 2011). Affected patients experience frequent pruritic hives with associated erythema and/or episodes of angioedema. CSU is reported to be associated with angioedema in approximately 50% of cases (McGirt et al. 2006). The classic urticaria description is a wheal and flare with a pale elevated lesion and surrounding erythema, ranging in size from a few millimeters to a few centimeters across, usually occurring in groups and often coalescing to form large confluent lesions.

The etiology of CSU is not clear. There are several theories including one proposing an infectious origin and another related to an autoimmune origin (Kaplan 2002). Some studies have found that approximately 30%–60% of patients with CSU have an autoimmune component as evidenced by the presence of a positive autologous serum skin test (Fiebiger et al. 1995; Tong et al. 1997; Zweiman et al. 1998). Another hypothesis regarding the etiology of CSU is that of a specific IgE antibody targeted to an endogenous antigen (Altrichter et al. 2011). Crosslinking of this IgE antibody docked in the high affinity IgE receptor (FcɛRI) could result in the activation of skin mast cells and release of chemical mediators, such as histamine, that lead to the wheal and flare formation of a hive. In fact, recent findings in a study of more than 450 patients with CSU indicate that greater than 50% of CSU patients have IgE antibodies directed against thyroperoxidase (Altrichter et al. 2011). While an autoimmune etiology can be found in a large percentage of patients, many patients do not have an identified autoimmune etiology despite having a similar disease presentation (Ferrer 2015).

The final common pathway in CSU is the abnormal activation of mast cells and basophils in the skin. In patients with CSU, increased numbers of mast cells can be found in both affected and unaffected skin (Kay et al. 2014). Furthermore, mast cells from CSU patients are more sensitive, have lower thresholds for activation, and respond more robustly by releasing more histamine and other inflammatory mediators. Similarly, increased numbers of basophils have been seen in the lesional and non-lesional skin of patients with CSU (Ying et al. 2002). In patients with CSU, there is a paradoxical basopenia thought to be due to increased recruitment of basophils to diseased skin. The peripheral basopenia is inversely correlated with severity of disease activity. In comparison with healthy controls, studies have shown that blood basophils of CSU patients have a reduced capacity to release histamine following IgE stimulation. This paradoxical reduction is attributed to prior in vivo activation in the skin (Kern and Lichtenstein 1976). However, when basophils from CSU patients are incubated with

serum from other CSU patients or even normal sera, they release more histamine than basophils from healthy donors. Collectively, these data suggest that basophil signaling and activation are dysregulated in patients with CSU (Luquin et al. 2005).

Roughly half of patients with CSU achieve symptomatic control with H1 antihistamine therapy at approved doses. In some cases, the dose of antihistamine is increased (up to 4 times the approved dose per local treatment guidelines) and additional therapies, such as leukotriene receptor antagonists (LTRAs), are used although increased doses of antihistamines and LTRAs are not approved for the treatment of CSU. CSU can be a debilitating condition because of a lack of clinical response as well as the unpredictable course of the disease, both of which can have a profound negative influence on the patient's quality of life (Tilles 2005).

Patients may remain symptomatic despite ongoing H1 antihistamine treatment (up to 4 times the approved dose per local treatment guidelines; Powell et al. 2015), and for this group of patients, therapies such as immunosuppressants (including cyclosporine, corticosteroids, intravenous immunoglobulin G [IVIG], and methotrexate) and plasmapheresis have been used (Kozel and Sabroe 2004). These agents have variable success and may be associated with severe adverse effects. More recently, omalizumab was approved for treatment of refractory CSU/CIU.

#### 1.2 **BACKGROUND ON BRUTON'S TYROSINE KINASE AND FENEBRUTINIB**

#### 1.2.1 **Bruton's Tyrosine Kinase**

Discovery of the genetic basis for primary immunodeficiencies has been the source of new therapeutic targets in immunomodulatory therapies (Puri et al. 2013; Bugatti et al. 2014; Whang and Chang 2014). In humans, mutations in the gene for Bruton's tyrosine kinase (BTK), which is located on the X chromosome, can result in the development of an immunodeficiency state characterized by a significant absence of circulating B cells (Bruton 1952; Tsukada et al. 1993; Vetrie et al. 1993; Conley et al. 2005) and very low immunoglobulin levels due to a defect in B-cell differentiation at the pro- to pre-B cell stage that precludes assembly of the B-cell receptor (BCR) complex and immunoglobulin gene expression (Reth and Nielsen 2014). Affected male patients have a primary immune deficiency, X-linked agammaglobulinemia (XLA), and are susceptible to recurrent infections starting shortly after birth. Patients with XLA can live relatively normal lives on a standard therapy of intravenous (IV) immunoglobulin, which suggests that BTK can be safely inhibited, especially in people with established immune systems. IV immunoglobulin replacement therapy lowers the rate of infection, reduces hospitalization rates for patients with XLA, and has greatly improved the long-term prognosis of these patients.

BTK is essential for the differentiation and activity of B cells during immune system ontogeny and normal adaptive immune responses. BTK is activated by phosphatidylinositol 3-kinase-dependent plasma membrane recruitment and

Fenebrutinib (GDC-0853)—Genentech, Inc.

phosphorylation on tyrosine Y551 by the Src-family kinase Lyn. Autophosphorylation and activation also occurs on tyrosine Y223 in a BTK-specific manner. Once activated, BTK induces PLC $\gamma$ 2- and Ca<sup>2+</sup>-dependent signaling, which leads to the activation of NF- $\kappa$ B- and NFAT-dependent pathways leading to cellular activation and differentiation (Niiro and Clark 2002). In addition, BTK is important in Fc $\epsilon$ RI signaling in both basophils and mast cells, the key cell types in the pathogenesis of CSU. BTK null mice have impaired Fc $\epsilon$ RI signaling resulting in decreased histamine and inflammatory cytokine release (Hata et al. 1998; Iyer et al. 2011).

## 1.2.2 <u>Nonclinical Experience with Fenebrutinib</u>

Fenebrutinib (also referred to as GDC-0853 or RO7010939) is a highly selective, orally administered, reversible inhibitor of BTK that is being developed by Genentech, Inc. as a potential therapeutic for autoimmune diseases, including CSU. Fenebrutinib has undergone extensive investigation in nonclinical in vitro and in vivo studies to characterize its pharmacological, metabolic, and toxicological properties (see the Fenebrutinib Investigator's Brochure for further details).

In vitro cell-based experiments suggest that antagonism of BTK leads to inhibition of BCR-dependent B-cell proliferation and a reduction of inflammatory cytokine production from myeloid cells (including tumor necrosis factor alpha [TNF- $\alpha$ ], interleukin 1 [IL-1], and interleukin 6 [IL-6]) by preventing signaling through the Fc $\gamma$ RIII receptor (Di Paolo et al. 2011; Liu et al. 2011). Fenebrutinib effectively blocks BCR- and CD40-mediated activation and proliferation of B cells. BTK in B cells also plays a role in TLR4-mediated B-cell proliferation and class switching. In monocytes, fenebrutinib inhibits TLR4- and immune complex-mediated inflammatory cytokine production, including TNF- $\alpha$ , which contributes to disease pathogenesis in rheumatoid arthritis (RA).

As described above, the pathophysiology of CSU is not completely understood. A key step is  $Fc_ERI$ -activation and release of histamine and inflammatory cytokines from mast cells and basophils, leading to the wheal and flare formation of a hive as well as angioedema. In support of the importance of BTK in  $Fc_ERI$  signaling and the pathogenesis of CSU, BTK null mice have impaired  $Fc_ERI$  signaling, resulting in decreased histamine and inflammatory cytokine release (Hata et al. 1998; Iyer et al. 2011).

Consistent with these findings, in vitro experiments with human mast cell lines demonstrated that fenebrutinib could effectively inhibit the release of histamine induced by cross-linking of IgE bound to Fc $\epsilon$ RI on the surface of mast cells. In addition, in a Phase Ib study in healthy volunteers, oral administration of fenebrutinib inhibited ex vivo basophil activation as measured by diminished cell surface expression of CD63 after cross-linking of IgE. As such, fenebrutinib inhibits the activity of two specific cell types that play key roles in disease pathology in CSU.

The fenebrutinib safety profile has been assessed in repeat-dose, general toxicology studies (once a day [QD] oral dosing) ranging from 1 week to 9 months in rats and dogs; in vitro and in vivo genetic toxicology studies; in vitro phototoxicity evaluation; in vitro and in vivo safety pharmacology studies of the central nervous, respiratory, and cardiovascular systems; and embryo-fetal development (Seg II) studies in rats and rabbits. Overall, fenebrutinib was well tolerated for up to 6 months in rats (up to 104  $\mu$ M • hr) and up to 9 months in dogs (up to 36  $\mu$ M • hr). Notable findings identified in nonclinical toxicology studies include vascular inflammation ( $\geq$  56  $\mu$ M • hr) in dogs, hepatotoxicity (180  $\mu$ M • hr) in dogs and rats, and a minimal increase in corrected QT interval (QTc; 7 ms or 3%; extrapolated unbound maximum observed concentration [Cmax] of 3.17  $\mu$ M) in dogs. Fetal malformations in rats (at 627  $\mu$ M • hr) and rabbits ( $\geq$  10.6  $\mu$ M • hr) warrant the continued use of highly effective contraception in clinical trials. On the basis of the nonclinical and clinical safety data to date, fenebrutinib is expected to be well tolerated at the doses and duration administered in the current study.

## 1.2.3 <u>Clinical Experience with Fenebrutinib</u>

As of 12 March 2018, fenebrutinib or placebo has been administered to 1099 subjects (i.e., 333 healthy subjects, 24 patients with hematological malignancies, 576 patients with rheumatoid arthritis, 129 patients with systemic lupus erythematosus, and 37 patients with chronic spontaneous urticaria) at doses with a range of 0.5–600 mg and has been generally well tolerated with no safety concerns that have led to a change in the conduct of the studies.

Study GO29089 is a Phase I, open-label study in which fenebrutinib has been evaluated in patients with relapsed or refractory B-cell non-Hodgkin's lymphoma or chronic lymphocytic leukemia. In order to focus on the autoimmune indications, Genentech elected to stop development of fenebrutinib in oncology, and the Phase I study is continuing without further patient enrollment. Enrollment was stopped after completion of the 400-mg dose level at which time 24 patients had been enrolled in 3 cohorts: 100 mg, 200 mg, and 400 mg fenebrutinib daily. Seven patients remain in the study, and all have undergone intrapatient dose escalation to 400 mg QD fenebrutinib. The mean duration of daily dosing for these 7 patients has been 21 months (range of 18–23 months). Fenebrutinib was well tolerated with no dose-limiting toxicities (DLTs), maximum tolerated dose was not reached, and adverse events have been generally non-serious National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (NCI CTCAE v4.0) Grade 1 or Grade 2 events that have been clinically manageable. The adverse events regardless of causality reported in ≥ 15% of patients include fatique, nausea, diarrhea, headache, abdominal pain, dizziness, cough, and thrombocytopenia. As of August 2016, 11 serious adverse events had been reported in 5 patients, of whom 2 had a fatal outcome (i.e., complications of H1N1 influenza and influenza pneumonia).

Study GP29318 was a two-part, single-ascending dose (SAD) study to assess the safety, tolerability, and pharmacokinetics of fenebrutinib administered to 93 healthy subjects. In Part 1, the single-dose–escalation portion, 71 subjects were randomized to panels of 8 subjects (6:2 active:placebo ratio) per dose group (0.5-600 mg), with 53 subjects receiving active fenebrutinib. In Part 2, 100 mg fenebrutinib was administered to 40 subjects in the open-label food and pilot rabeprazole effect study. There were no serious adverse events and no withdrawals due to adverse events during the conduct of Study GP29318. In Part 1 of the study, there were no dose-limiting adverse events (DLAEs) at single doses up to 600 mg fenebrutinib. All adverse events were mild in intensity (Grade 1; Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials) and transient. No adverse events increased in intensity or frequency with dose escalation. There were two treatment-emergent adverse events of mild self-limited headache reported as related to fenebrutinib administration. There were no trends in safety laboratory findings, vital sign changes, physical examination findings, or ECG changes. There were no trends in hepatic laboratory changes following single doses of fenebrutinib in healthy subjects. Administration of fenebrutinib inhibited ex vivo basophil activation as demonstrated by diminished CD63 cell surface expression after cross-linking of IgE. Refer to the Fenebrutinib Investigator's Brochure for further information on Study GP29318, including pharmacokinetics.

Study GA29347 was a multiple-ascending dose (MAD) study to assess the safety, tolerability, and pharmacokinetics of multiple doses of fenebrutinib administered to 30 healthy subjects for 14 days. Forty subjects were randomized to panels of 8 subjects (6:2 active:placebo) per dose group, at doses of 20 mg twice a day (BID), 60 mg BID, 150 mg BID, 250 mg BID, or 500 mg QD for 14 days, with 30 subjects receiving active fenebrutinib. The study drug was well tolerated. There were no serious adverse events and no withdrawals due to adverse events during the conduct of the study. All adverse events were mild in intensity (Grade 1) and transient, with no relationship to dose. Adverse events included skin reactions (i.e., rash, contact dermatitis, and skin irritation from ECG leads), nausea, headache, insomnia, toothache, tinnitus, and asymptomatic bacteriuria. There were no trends in safety laboratory, vital sign, physical examination, or ECG findings. Similar to the SAD study, dose-dependent inhibition of CD63 expression was observed following fenebrutinib administration, with sustained inhibition over the duration of dosing.

Study GP29832 was a relative bioavailability study designed to evaluate the effects of formulation, food, and proton-pump inhibitor (PPI) or methotrexate co-administration on the pharmacokinetics of fenebrutinib in healthy subjects. Fenebrutinib was well tolerated when administered to 48 healthy subjects at the 200-mg dose level.

Study GA29350 is a multicenter Phase II dose ranging study comparing the efficacy and safety of fenebrutinib versus placebo and adalimumab in patients with RA who have had an inadequate response to previous methotrexate therapy and versus placebo in

Fenebrutinib (GDC-0853)—Genentech, Inc. 29/Protocol GS39684, Version 4

patients with an inadequate response to previous tumor necrosis factor therapy. The study began enrollment in September 2016, and the total planned enrollment is approximately 580 patients.

Study GA30044 is the first study investigating fenebrutinib in systemic lupus erythematosus (SLE). This is a multicenter, Phase II, randomized, double-blind, placebo-controlled, parallel-group, dose-ranging study designed to evaluate the efficacy and safety of fenebrutinib in patients with moderate-to-severe active SLE in combination with standard-of-care therapy.

The drug-drug interaction Study GP39616 has recently concluded. While final results are not yet available, preliminary data suggests:

• Fenebrutinib is a Breast Cancer Resistance Protein (BCRP) inhibitor. Consequently, fenebrutinib may alter transport of BCRP substrates and result in increased plasma concentrations of BCRP substrates.

The study also confirmed the following:

- Fenebrutinib is a mild inhibitor of CYP3A at clinically relevant doses. Consequently, fenebrutinib may alter metabolism of CYP3A substrates and result in increased plasma concentrations of CYP3A substrates.
- Fenebrutinib is a moderately sensitive substrate of CYP3A at clinically relevant doses. There is a moderate potential for levels of fenebrutinib to increase in patients taking concomitant medications that inhibit CYP3A and decrease in patients taking medications that induce CYP3A.

Refer to the Fenebrutinib Investigator's Brochure for detailed background information on fenebrutinib as well as for additional details on nonclinical and clinical studies.

#### 1.3 STUDY RATIONALE AND BENEFIT-RISK ASSESSMENT

Omalizumab, an anti-IgE monoclonal antibody, has demonstrated efficacy in treating patients with CSU, highlighting the key role of IgE in CSU pathogenesis. Inhibition of IgE-mediated FcERI signaling by BTK inhibition offers a promising mechanism for the treatment of CSU. In preclinical in vitro studies, BTK inhibition was able to prevent the release of histamine and inflammatory cytokines from mast cells after FcERI engagement and cross-linking. In addition, in the healthy volunteer SAD and MAD studies, oral administration of fenebrutinib was able to inhibit ex vivo basophil activation as demonstrated by diminished CD63 cell surface expression. As such, fenebrutinib inhibits two key pathogenic cell types in CSU. The aim of this study is to determine if fenebrutinib can effectively treat patients with CSU, as measured by reduction in disease activity.

Humans with XLA lack functional BTK but can live relatively normal lives on a standard therapy of IV immunoglobulin (Kaveri et al. 2011), suggesting that BTK can be safely inhibited in patients with CSU who have functional immune systems. Clinical experience

with fenebrutinib to date has not generated safety concerns that would preclude further evaluation in patients with CSU. In the SAD (Study GP29318), MAD (Study GA29347), relative bioavailability (Study GP29832), and oncology (Study GO29089) studies, fenebrutinib was well tolerated with no DLAEs or DLTs. In the oncology study, there were 2 deaths due to complications of confirmed influenza (i.e., H1N1 influenza and influenza pneumonia).

Several measures will be taken to ensure the safety of patients participating in this study based on the potential risks for fenebrutinib based on nonclinical and clinical studies and published literature (see Section 5.1.1). Eligibility criteria have been designed to exclude patients at higher risk for potential toxicities. In addition, the sites selected for this study will be specialty dermatology and immunology clinics with experience in treating CSU.

#### 1.3.1 Infections

Fenebrutinib is a targeted immunomodulator; however, as a reversible inhibitor, the degree to which fenebrutinib antagonism of BTK signaling may suppress immune activity is unknown. Patients participating in this study may be at risk for infections, including opportunistic infections. Therefore, patients at high risk for infection will be excluded (see Section 5.1.1.1). Patients will be carefully monitored throughout the study for infections. Fenebrutinib will be discontinued in any patient who develops a serious infection, opportunistic infection, or any infection requiring treatment with an IV antimicrobial agent.

## 1.3.2 Bleeding

BTK is expressed in platelets and is involved in platelet function via GPVI/collagen receptor signaling and GP1b receptor signaling. Platelets from patients with XLA demonstrate decreased activation in response to submaximal collagen stimulation but normal response to thrombin; clinically, there is no reported bleeding propensity in patients with XLA. In the fenebrutinib clinical study involving oncology patients (GO29089), 2 patients experienced Grade ≥3 gastrointestinal (GI) bleeding. These events were not dose related and occurred in patients on non-steroidal anti-inflammatory drugs (NSAIDs)/acetylsalicylic acid with a history of gastroesophageal or peptic ulcer disease.

It is unknown whether fenebrutinib will increase the risk of bleeding in patients with CSU who receive antiplatelet or anticoagulant therapies. Therefore, the eligibility criteria exclude patients at high risk for bleeding complications.

### 1.3.3 <u>Cytopenias</u>

Neutropenia, anemia, and thrombocytopenia have been observed in patients with hematologic malignancies who received fenebrutinib. No clinically significant changes in cell counts were observed in the healthy volunteer studies. Events have been

monitorable and clinically manageable. Cell counts will be monitored regularly throughout the study.

## 1.3.4 <u>Hepatotoxicity</u>

Evidence of hepatobiliary injury was observed in animals administered relatively high doses of fenebrutinib in repeat-dose toxicity studies. In clinical studies to date, in autoimmune indications, enrolling over 800 patients, multiple cases of treatment emergent Grade 3 (or severe) elevations of ALT, some of which were considered serious adverse events, have been observed in the randomized clinical studies, which remain blinded to the Sponsor in terms of treatment assignment, as well as in open label extensions of fenebrutinib. These cases have been seen in blinded studies in CSU. None of the cases of transaminase elevations resulted in clinical jaundice or bilirubin >2 × ULN (Hy's Law). All transaminase elevations have been reversible when dosing of blinded study medication/placebo was withheld. These findings have not been seen in single dose and multiple dosing for 14 days in healthy subjects and QD dosing in patients with hematological malignancies. To minimize this risk, exclusion criteria have been defined for abnormal liver enzyme and function tests and current liver disease (see Section 4.1.2). For further information on nonclinical and clinical findings of hepatotoxicity, please see the Fenebrutinib Investigator's Brochure.

## 1.3.5 <u>Cardiovascular Effects</u>

Fenebrutinib is considered to have a low potential to cause QT interval prolongation or to directly affect other cardiovascular parameters at therapeutic exposures. A minimal increase in corrected QT (QTc; 7 ms or 3%) interval was noted at 45 mg/kg in the single-dose cardiovascular safety pharmacology study in telemetry-instrumented dogs. Cardiac safety will be evaluated in all patients at baseline and throughout the study, with routine monitoring of vital signs, including heart rate and blood pressure, collection of ECGs, and reporting of cardiac adverse events.

### 1.3.6 Malignancy

The impact of BTK inhibition on the development of malignancies is not known; however, malignancies are considered a potential concern for all immunomodulatory agents. Patients with a history of cancer within 10 years of screening will be excluded from study participation, except for basal or squamous cell carcinoma of the skin that has been excised and is considered cured and in situ carcinoma of the cervix treated with apparent success by curative therapy more than 1 year prior to screening.

Overall, fenebrutinib has been well tolerated in Phase I healthy subjects and an oncology study. On the basis of the compelling mechanism for BTK inhibition in CSU, the benefit-risk ratio for this study is deemed acceptable. The safety profile of fenebrutinib will be further characterized in this Phase II study. A robust safety monitoring plan that describes the potential risks for fenebrutinib and the risk-mitigation strategies to minimize risks for the patients in this trial is provided in Section 5.

Please refer to the most recent Fenebrutinib Investigator's Brochure for additional details on clinical and nonclinical studies and additional safety information.

## 2. <u>OBJECTIVES AND ENDPOINTS</u>

This pilot and dose-ranging study will evaluate the efficacy, safety, and pharmacokinetics of fenebrutinib compared with placebo in patients with CSU refractory to anti-histamines (up to 4 times the approved dose per local treatment guidelines). Specific objectives and corresponding endpoints for the study are outlined in Table 1.

Table 1 Objectives and Corresponding Endpoints

| Objectives | Corresponding Endpoints |
|---|---|
| Efficacy Objective: | |
| To evaluate the efficacy of<br>fenebrutinib compared with placebo | Primary Endpoint: |
| | Change from baseline in the UAS7 at Day 57 (Week 8) |
| in patients with CSU who are | Secondary Endpoints: |
| refractory to anti-histamines | <ul> <li>Proportion of patients who are well controlled (UAS7 ≤6)<br/>at Day 57</li> </ul> |
| | <ul> <li>Change from baseline in the UAS7 at Day 29 (Week 4)</li> </ul> |
| | Exploratory Endpoint: |
| | Change from baseline in the weekly itch score at Day 29 |
| | Change from baseline in the weekly itch score at Day 57 |
| | Change from baseline in the weekly hives score at Day 57 |
| | <ul> <li>Proportion of patients who are well controlled (UAS7 ≤ 6)<br/>at Day 29</li> </ul> |
| | <ul> <li>Proportion of patients who achieve complete response<br/>(UAS7=0) at Day 29</li> </ul> |
| | <ul> <li>Proportion of patients who achieve complete response<br/>(UAS7=0) at Day 57</li> </ul> |
| | <ul> <li>Proportion of patients achieving MID in UAS7 at Day 57<br/>(reduction from baseline ≥ 11 points)</li> </ul> |
| | <ul> <li>Proportion of patients achieving MID in the weekly itch<br/>score at Day 57 (reduction from baseline ≥ 5 points)</li> </ul> |
| | <ul> <li>Time to achieving MID in UAS7 (reduction from baseline<br/>≥11 points)</li> </ul> |

Table 1 Objectives and Corresponding Endpoints (cont.)

| Objectives | Corresponding Endpoints |
|---|---|
| Safety Objective: | |
| To evaluate the safety of<br>fenebrutinib compared with<br>placebo | <ul> <li>The nature, frequency, timing, and severity of adverse events</li> <li>Change from baseline in targeted vital signs, physical examination findings, ECGs, and clinical laboratory results following fenebrutinib administration</li> </ul> |
| Pharmacokinetic Objective: | |
| To characterize the<br>pharmacokinetics of fenebrutinib<br>in patients | Plasma concentrations of fenebrutinib at specified timepoints |

AUC<sub>0-t</sub>= area under the concentration–time curve from time 0 to time t; BTK=Bruton's tyrosine kinase CL/F = apparent clearance; C<sub>max</sub>= maximum concentration observed; C<sub>trough</sub>= steady-state concentration at the end of a dosing interval; CSU = chronic spontaneous urticaria; MID = minimally important difference;

PK = pharmacokinetic; t<sub>1/2</sub> = half-life; t<sub>max</sub> = time to maximum concentration; UAS7 = Urticaria Activity Score over 7 days;

### 3. STUDY DESIGN

## 3.1 DESCRIPTION OF THE STUDY

This pilot and dose-ranging study is a multicenter, randomized, double-blind, placebo-controlled, parallel-group study of the efficacy and safety of fenebrutinib as add-on

Fenebrutinib (GDC-0853)—Genentech, Inc.

34/Protocol GS39684, Version 4

therapy for the treatment of adult patients 18–75 years old who have been diagnosed with CSU and who remain symptomatic despite treatment with H1 antihistamines (including doses up to 4 times the approved dose per local treatment guidelines). The study will consist of two cohorts. Cohort 1 will enroll approximately 45 patients across multiple sites. After screening, eligible patients will be randomly allocated in a 2:1 ratio to receive fenebrutinib 200 mg orally (PO) twice daily (BID) or matching placebo for 8 weeks and will maintain stable doses of standard-of-care H1 antihistamine therapy throughout the study. On the basis of results from an interim analysis of Cohort 1, a dose-ranging cohort, Cohort 2, will be opened and approximately 120 patients will be randomly allocated in a 1:1:1:1 ratio to receive 50 mg PO daily (QD), 150 mg PO QD, 200 mg PO BID of fenebrutinib, or placebo, respectively, for 8 weeks and will maintain stable doses of standard-of-care H1 antihistamine therapy (background therapy) throughout the study.

Both cohorts will consist of 3 distinct study periods over a time-period of 14 weeks as outlined below (see Figure 1):

Screening period: Day –14 to Day –1

• Treatment Period: Day 1 to Day 57 (Week 0 to Week 8)

Follow-Up Period: Day 57 to Day 85 (Week 8 to Week 12)

Patients in both cohorts will have a screening period of approximately 2 weeks to establish their eligibility for the study and baseline symptom scores. For the duration of the screening period, patients must maintain stable doses of their pre-screening combination therapy with standard-of-care H1 antihistamines (i.e., up to 4 times the approved dose per local treatment guidelines). The screening period will consist of visits at Day –14 and Day –7. Patients must meet all of the following criteria to enter the screening period:

- Documented treatment with a regimen that includes standard-of-care H1
   antihistamine for CSU at Day –14 and for at least the 3 consecutive days
   immediately prior to Day –14 (see Section 4.4.1 for list of H1 antihistamines available
   for use in this study)
- Willing and able to complete a symptom electronic diary (Urticaria Patient Daily eDiary) twice daily throughout the screening period to establish the patient's Urticaria Activity Score over 7 days (UAS7) score.

To be eligible for randomization in both cohorts, for the 7 days prior to randomization, patients must meet all of the following:

- Seven consecutive days of entries in the Urticaria Patient Daily eDiary, and
- UAS7 symptom score of ≥ 16 (range: 0-42)

Only in exceptional circumstances, when information concerning eligibility is outstanding (e.g., delayed laboratory results), will a longer screening period be permitted up to
3 business days. Upon approval from the Medical Monitor, patients may be re-screened or maybe retested during the screening period (see Section 4.5.2.2 and Section 4.5.2.1, respectively). Circumstances that may permit re-screening or retesting include, but are not limited to, a laboratory test result that does not meet eligibility requirements.

The primary efficacy endpoint will be at Day 57 (Week 8). Throughout the treatment period, patients must maintain stable doses of their pre-randomization H1 antihistamine therapy.

After completion of the 8-week treatment period, all patients in both cohorts will either enter a 4-week safety follow-up period to allow for further characterization of the pharmacokinetics and pharmacodynamics of fenebrutinib and collection of additional efficacy and safety data or they will have the opportunity to participate in the OLE Study GS40868 (see Section 3.1.2). During safety follow-up period, no study treatment will be given; patients must maintain stable doses of their pre-randomization CSU H1 antihistamine treatment (background therapy). In the safety follow-up period, patients may add up to one additional H1 antihistamine therapy in case of worsened symptoms (see Section 4.4.3). The goal of allowing additional H1 antihistamine therapy after the treatment period is to reduce patient dropout for improved safety evaluation.

In addition to their daily background therapy, for the duration of the study, all patients will be able to use a single approved dose of loratadine (10 mg maximum) or cetirizine (10 mg maximum) within a 24-hour period as rescue medication if symptoms worsen. If a patient needs rescue therapy and is already on background treatment with cetirizine or loratadine, the patient may receive 10 mg more of the same drug only if the total daily dose remains below 4 times the approved dose. Otherwise, the alternate rescue medication may be used. Patients should record the use of this medication in their eDiary. Patients receiving PPIs or H2 receptor antagonists (H2RAs) should be stabilized on a regimen beginning at least 2 weeks prior to randomization and continuing throughout the study (see Section 4.4.2.1).

Figure 1 Study Schema





BID=twice daily; PO = orally; QD = daily.

a Last blinded dose=p.m. before Day 57 visit

# 3.1.1 <u>Internal Monitoring Committee</u>

For Cohort 2, periodic safety reviews and any interim analysis will be performed by the Sponsor's internal monitoring committee (IMC) as outlined in the IMC charter. This committee will be unblinded to treatment assignments and will include Sponsor representatives from the following functions: Clinical Science, Drug Safety, Biostatistics, and Statistical Programming and Analysis. The IMC members will not have direct contact with investigational staff or site monitors. The IMC may decide to unblind the study team to enable decision-making and potential interactions with regulatory bodies. The IMC may invite representatives from other functional areas on an ad-hoc basis when additional expertise is required (e.g., Clinical Pharmacology, Research, etc.) or additional Sponsor scientists to participate in data analyses and review.

At any time during the study, the Sponsor may choose to inactivate and suspend enrollment and further dosing for a given treatment arm (in Cohort 2) or reduce the dose due to safety concerns and as guided by the IMC. In Cohort 2, subsequently enrolled patients will be randomly allocated to the remaining active arms.

# 3.1.2 Open-Label Extension Study GS40868

After completing the 8-week treatment period (at Day 57), eligible patients from Cohorts 1 and 2 will have the option to enter the OLE Study GS40868 and receive open-label fenebrutinib treatment. Patients who do not enter the OLE after completing the treatment period will undergo assessments at 4 weeks after the last dose of study drug (safety follow-up).

Patients who completed the treatment period and 4-week safety follow-up period may also enroll in the OLE study if eligible.

#### 3.2 END OF STUDY AND LENGTH OF STUDY

The end of this study is defined as the date when all patients have completed the study completion visit or early termination visit or have otherwise been discontinued from the study. The total duration of this study for each subject is approximately 14 weeks (for both cohorts), including screening, treatment, and safety follow-up periods.

The total length of the study, from screening of the first patient to the end of the study, is expected to be approximately 19 months.





# 3.3.2 Rationale for Patient Population

Patients enrolled in both cohorts of the study will have a CSU diagnosis for ≥ 6 months and will be refractory to treatment with a combination of H1 antihistamines consistent with standard of care (i.e., up to 4 times the approved dose per local treatment guidelines) as demonstrated by the presence of itch and hives for > 6 consecutive weeks on this treatment at any time prior to enrollment. In addition, patients will have a UAS7

score of  $\geq$  16 during the 7 days prior to randomization despite current use of combination therapy.

While H1 antihistamines are the mainstay of therapy for CSU, some patients do not respond or respond only partially to these therapies, and these patients tend to experience more severe disease. This patient population was selected for this study because of the unmet medical need for more effective oral treatments.

## 3.3.3 Rationale for Control Group

A placebo-treated control group is required for this study in order to achieve its efficacy and safety objectives given the inherent variability in symptoms and the different rates of improvement in the placebo arms of prior studies. Patients in the placebo arm will continue to receive stable standard-of-care anti-H1 therapy throughout the study. In addition, the study will allow for rescue medications for persistent symptoms.

# 3.3.5 Rationale for Pharmacokinetic Sample Collection Schedule

The sampling schedule is designed to assess multiple pre-dose (prior to study drug administration in clinic) plasma fenebrutinib concentrations, which will enable the estimation of systemic fenebrutinib exposures and subsequent exposure-response analyses, both of which may be reported separately. Results will be used to inform dosing regimens for future studies of fenebrutinib.

## 3.3.6 Rationale for Efficacy Endpoints

The change in the UAS7 (see Table 2 for daily assessment of Urticaria Activity Score [UAS]) has been chosen as the primary efficacy endpoint as it has been used in pivotal trials in CSU to measure reduction in CSU disease severity. The UAS7 is a summation of the average daily (a.m./p.m.) scores on the UAS (range: 0-6), which is a composite diary score with numeric severity intensity ratings on a scale of 0-3 (0=none to 3=intense/severe) for two domains: the intensity of the itch and the number of wheals/hives (see Table 2). The UAS will be recorded by the patient twice daily (morning and evening) in the patient Urticaria Patient Daily eDiary. UAS7 scores range from 0-42 and the minimally important difference (MID) is considered to be a reduction from baseline of  $\geq 9.5$  to 10.5 points (Mathias et al. 2012). The baseline UAS7 is the sum of the daily scores on the UAS over the 7 days prior to randomization (Day 1 visit for both cohorts), and the UAS7 at Day 57 is the sum of daily scores on the UAS over the 7 days prior to the Day 57 visit (for both cohorts). The same principles of calculating baseline and Day 57 weekly scores will be applied to the other weekly outcomes unless otherwise stated.

The kinetics of response to fenebrutinib will also be carefully evaluated throughout the course of the study at regular intervals (at least every 1–2 weeks for a period of 8 weeks). In addition, disease recurrence or duration of treatment benefit after study drug is withdrawn during the safety follow-up period will be measured during this study. This will provide initial guidance for the duration of therapy in future studies.

Table 2 Twice Daily Patient Assessment of CSU Disease Activity (UAS Scale)

| Score | Wheals (Hives) | Pruritus (Itch) |
|-------|-------------------------------|-----------------|
| 0 | None | None |
| 1 | Mild (1-6 hives/12 hour) | Mild |
| 2 | Moderate (7–12 hives/12 hour) | Moderate |
| 3 | Intense (>12 hives/12 hour) | Severe |

CSU = chronic spontaneous urticaria; UAS = Urticaria Activity Score.

## 4. MATERIALS AND METHODS

#### 4.1 PATIENTS

Approximately 45 patients in Cohort 1 and approximately 120 patients in Cohort 2, aged 18 to 75 years old who have been diagnosed with refractory CSU and who remain symptomatic despite standard-of-care H1 antihistamine therapy (i.e., up to 4 times the approved dose per local treatment guidelines), will be enrolled in this study.

# 4.1.1 <u>Inclusion Criteria</u>

Patients in Cohort 1 and 2 must meet the following criteria for study entry:

- Willing to give written informed consent, adhere to the visit schedules, comply with the study drug regimen, and meet other study requirements
- Aged 18–75 years, inclusive
- Diagnosis of CSU refractory to H1 antihistamines at the time of randomization, as defined by all of the following:
  - The presence of itch and hives for > 6 consecutive weeks at any time prior to enrollment despite current use of H1 antihistamines, consistent with standard of care (i.e., up to 4 times the approved dose per local treatment guidelines) during this time period
  - UAS7 score ≥ 16 during the 7 days prior to randomization (Day 1)
  - Patients must have been on daily stable doses of H1 antihistamines, consistent with standard-of-care therapy (i.e., up to 4 times the approved dose per local treatment guidelines) for CSU starting at least 3 consecutive days immediately prior to the screening visit through Day 1 and must document current use on all visits.
  - CSU diagnosis for ≥6 months

- Willing and able to complete an Urticaria Patient Daily eDiary for the duration of the study
- Completion of 7 days of the Urticaria Patient Daily eDiary entries in the 7 days prior to randomization (7 of 7 days must be completed [i.e., must complete an entry every day] with up to 2 non-consecutive entries missed)
- No evidence of active or latent or inadequately treated infection with tuberculosis (TB) as defined by the following:
  - A negative QuantiFERON-TB-Gold® (QFT) performed (for German sites only: QFT is the preferred test) at the screening visit or within the 3 months prior to screening

If QFT is unavailable, a negative Mantoux purified protein derivative (PPD) skin test as defined by the Centers for Disease Control and Prevention guidelines, may be performed at the screening visit or within the 3 months prior to screening -AND-

Any additional procedures (e.g., chest X-Ray) only if required per local guidelines/standard of care to rule out latent or active TB

NOTE: A documented negative screening for TB via the PPD test or a negative QFT within 3 months prior to screening and if required per local standard of care, a chest X-ray, is sufficient and no further screening with QFT is required.

Patients with a history of Bacille Calmette-Guérin (BCG) vaccination should be screened using the QFT test, only.

- An indeterminate QFT test should be repeated.
- A positive QFT test or two successive indeterminate QFT results should be considered a positive diagnostic TB test.
- An indeterminate QFT test followed by a negative QFT test should be considered a negative diagnostic TB test.
- Only for patients currently receiving PPIs or H2RAs: Treatment must be at a stable dose during the 2-week screening period prior to randomization and with a plan to remain at a stable dose for the duration of the study.
- For women of childbearing potential: Agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 4 weeks after the last dose of study drug (see Section 5.4.3.1). Women must refrain from donating eggs during this same period.
  - A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).

- Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, established proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. Women using estrogen-containing hormonal contraceptives as a method of contraception <u>must</u> also use a barrier, such as a male condom, in conjunction with the hormonal contraceptives.
- The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient.
   Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
- For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm, as defined below (also see Section 5.4.3.2):
  - With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 4 weeks after the last dose of study treatment to avoid exposing the embryo. Men must refrain from donating sperm during this same period.
  - The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

## 4.1.2 <u>Exclusion Criteria</u>

Patients in Cohort 1 and 2 who meet any of the following criteria will be excluded from study entry:

- Treatment with omalizumab or other monoclonal antibody therapies used to treat CSU within 4 months prior to screening or primary nonresponse to omalizumab
- Use of a non-biologic investigational drug or participation in an investigational study with a non-biologic drug within 30 days prior to study drug administration on Day 1 (or within 5 half-lives of the investigational product, whichever is greater)
- Use of a biologic investigational therapy or participation in an investigational study involving biologic therapy within 90 days or 5 half-lives, whichever is greater, prior to study drug administration on Day 1
- Previous treatment with fenebrutinib or other BTK inhibitors
- Patients whose urticaria is solely due to physical urticaria
- Other diseases with symptoms of urticaria or angioedema, including urticarial vasculitis, urticaria pigmentosa, erythema multiforme, mastocytosis, hereditary or acquired angioedema, lymphoma, or leukemia
- Atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, or other skin disease associated with itch such as psoriasis

- Routine (daily or every other day during 5 or more consecutive days) doses of the following medications within 30 days prior to screening: systemic or cutaneous (topical) corticosteroids (prescription or over the counter), hydroxychloroquine, methotrexate, cyclosporine, or cyclophosphamide
- Prior utilization of IV steroids for treatment of laryngeal angioedema
- IVIG or plasmapheresis within 30 days prior to screening
- History of anaphylactic shock without clearly identifiable avoidable antigen (e.g., due to food allergy)
- Hypersensitivity to fenebrutinib or any component of the formulation
- Major surgery within 8 weeks prior to screening or surgery planned prior to end of study (12 weeks after randomization)
- Require any prohibited concomitant medications (see Section 4.4.3)
- History of live attenuated vaccine within 6 weeks prior to randomization or requirement to receive these vaccinations at any time during study drug treatment
  - Seasonal influenza and H1N1 vaccination is permitted if the inactivated vaccine formulation is administered.
- Evidence of clinically significant cardiac, neurologic, psychiatric, pulmonary, renal, hepatic, endocrine (including uncontrolled diabetes mellitus), metabolic, or GI disease that, in the investigator's opinion, would compromise the safety of the patient, interfere with the interpretation of the study results or otherwise preclude patient participation
  - Any items that are cause for uncertainty must be reviewed with the Medical Monitor.
- Uncontrolled disease states, such as asthma, psoriasis, or inflammatory bowel disease, where flares are commonly treated with oral or parenteral corticosteroids
- History of vasculitis
- Current liver disease
- Any known active infection (with the exception of fungal nail infections or oral herpes)
- History of recurrent bacterial, viral, mycobacterial or fungal infections (defined as >2 similar episodes requiring anti-microbial treatment within the previous 12 months), with the exception of recurrent oral or genital herpes (herpes simplex virus 1/herpes simplex virus 2) or uncomplicated urinary tract infections in females.
- Any history of opportunistic infections that, in the investigator or Sponsor's judgment,
   would raise safety concerns regarding the patient's participation in the study
- Any major episode of infection requiring hospitalization or treatment with IV
  antimicrobials within 8 weeks prior to and during screening or treatment with oral
  antimicrobials within 2 weeks prior to and during screening
  - Antimicrobials include antifungal, antibacterial, and antiviral agents.
- History of or currently active primary or secondary immunodeficiency, including known history of HIV infection

- Evidence of chronic and/or active hepatitis B or C
  - Positive hepatitis B surface antigen (HBsAg) or hepatitis C serology (regardless of treatment status)
  - Positive hepatitis B core antibody (HBcAb)
- History of cancer, including hematologic malignancy and solid tumors, within
   10 years before screening
  - Basal or squamous cell carcinoma of the skin that has been excised and is considered cured and in situ carcinoma of the cervix treated with apparent success by curative therapy > 1 year prior to screening are not exclusionary.
- Women who are pregnant, nursing (breastfeeding), or intending to become pregnant during the study or within 4 weeks after completion of the study
- For women of childbearing potential (including those who have had a tubal ligation): positive serum pregnancy test result at screening or on Day 1.
  - A serum pregnancy test is needed on Day 1 <u>only</u> if the urine pregnancy test is positive (see Section 4.1.1 for definition of "childbearing potential").
- History of alcohol, drug (e.g., tetrahydrocannabinol [THC], marijuana), or chemical abuse within the 12 months prior to screening as determined by the investigator
- Need for systemic anti-coagulation with warfarin, other oral or injectable anti-coagulants, or anti-platelet agents other than NSAIDs, aspirin, and other salicylates
- History of non-gallstone-related pancreatitis or chronic pancreatitis
- History of hospitalizations or transfusion for a GI bleed
- History of cerebrovascular accident (CVA) within 10 years or any history of hemorrhagic CVA
- History of spontaneous intracranial hemorrhage or history of traumatic intracranial hemorrhage within 10 years
- Known bleeding diathesis
- Screening 12-lead ECG that demonstrates clinically relevant abnormalities that may affect patient safety or interpretation of study results, including
  - QT interval corrected using Fridericia's formula (QTcF) > 440 ms demonstrated by at least two ECGs > 30 minutes apart
- History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias such as long QT syndrome and other genetic risk factors (e.g., Brugada syndrome), structural heart disease (e.g., severe left ventricular systolic dysfunction, severe left ventricular hypertrophy), coronary heart disease (symptomatic or with ischemia demonstrated by diagnostic testing, prior coronary artery bypass grafting, or coronary lesions > 70% diameter stenosis that have not been or cannot be re-vascularized), clinically significant electrolyte abnormalities (e.g., hypokalemia, hypomagnesemia, hypocalcemia), or family history of sudden unexplained death or cardiac ion channel mutations (e.g., congenital long QT syndrome)

- Current treatment with medications that are well known to prolong the QT interval (see https://crediblemeds.org/index.php/login/dlcheck) at doses that have a clinically meaningful effect on QT, as determined by the investigator; the investigator may contact the Sponsor for confirmation if needed
- Current treatment with astemizole, terfenadine, and/or ebastine
- Any condition possibly affecting oral drug absorption (e.g., gastrectomy, clinically significant diabetic gastroenteropathy, or certain types of bariatric surgery such as gastric bypass)
  - Procedures such as gastric banding, that simply divide the stomach into separate chambers, are not exclusionary.
- Any uncontrolled clinically significant laboratory abnormality that would affect safety, interpretation of study data, or the patient's participation in the study
- For German sites only: Subjects who live in detention on court order or on regulatory action as per local and national law (see §40 subSection 1 sentence 3 no. 4 Arzneimittelgesetz; Medicinal Products Act).

The following exclusion criteria are based on screening laboratory tests. Laboratory tests may be repeated once during the screening period unless otherwise indicated (see Section 4.5.2.1):

- Creatinine > 1.5 times the upper limit of normal (ULN; may be repeated if 1.5–2×ULN)
- Creatinine clearance < 70 mL/min (may be repeated if 60–69 mL/min) as estimated by the Cockcroft-Gault Equation
- ALT or AST > 1.5 times ULN (may be repeated if 1.5–3×ULN)
- Total bilirubin > ULN (may be repeated if 1–3×ULN)
- Hemoglobin < 11 g/dL (may be repeated if 10–10.9 g/dL)</li>
- ANC  $< 1.5 \times 10^9 / L$  (may be repeated if  $1.2 1.5 \times 10^9 / L$ )
- Platelet count  $< 100 \times 10^9$ /L (may be repeated if  $80-100 \times 10^9$ /L)
- IgG < 500 mg/dL (should not be repeated)
- Abnormalities in hepatic synthetic function tests (e.g., PT, INR, PTT, albumin) judged by the investigator to be clinically significant

## 4.2 METHOD OF TREATMENT ASSIGNMENT AND BLINDING

#### 4.2.1 Randomization and Blinding

This study is randomized, double-blinded, and placebo-controlled to minimize potential bias in treatment assignment, patient monitoring, and efficacy assessments. Random allocation will be conducted via an interactive voice or web-based response system (IxRS) and the Sponsor will provide the specifications of the randomization algorithm to the IxRS vendor. Patients in Cohort 1 will be randomly allocated to 200 mg PO BID fenebrutinib or placebo at an approximately 2:1 ratio using a stratified permuted blocks randomization scheme with stratification by country. Patients in Cohort 2 will be

randomly allocated to each of the four treatment arms at an approximately 1:1:1:1 ratio, using a stratified permuted blocks randomization scheme with stratification by country.

Patients and study site personnel will be blinded to the individual treatment assignments throughout the study. Only standard and safety laboratory data results from the local laboratory (such as CBC, chemistries, and pregnancy testing) will be available to sites. Results of other assessments performed after randomization that might unblind investigators to the treatment patients received will not be provided to sites or to the Sponsor's staff directly involved in study conduct.

Although PK samples must be collected from patients assigned to the comparator arm to maintain the blinding of treatment assignment, PK assay results for these patients are generally not needed for the safe conduct or proper interpretation of this trial. Sponsor personnel or a designee responsible for performing PK assays will be unblinded to patients' treatment assignments to identify appropriate PK samples to be analyzed. Samples from patients assigned to the placebo arm will not be analyzed except by request (e.g., to evaluate a possible error in dosing).

Patient and study site personnel will be blinded to treatment assignments throughout the study. During trial conduct, the Sponsor will monitor blinded clinical and safety data on safety and study conduct on an ongoing basis. For Cohort 1, if required for safety evaluations, Sponsor team personnel, but not the sites, not directly involved in the conduct of the study will have access to unblinded data. These Sponsor team personnel may include individuals with clinical and medical experience, biostatisticians, and individuals responsible for analyzing and interpreting the pharmacodynamics and pharmacokinetics of the study drug. For information on Cohort 2, see Section 3.1.1.

#### 4.2.2 <u>Unblinding</u>

If unblinding is necessary for patient management (e.g., in the case of a serious adverse event for which patient management might be affected by knowledge of treatment assignment), the investigator will be able to break the treatment code by contacting the IxRS. Treatment codes should not be broken except in emergency situations. If the investigator wishes to know the identity of the study drug for any other reason, he or she should contact the Medical Monitor directly. The investigator should document and provide an explanation for any premature unblinding (e.g., accidental unblinding, unblinding due to a serious adverse event).

For regulatory reporting purposes, and if required by local health authorities, the Sponsor will break the treatment code for all serious, unexpected, suspected adverse reactions (see Section 5.7) that are considered by the investigator or Sponsor to be related to study drug.

#### 4.3 STUDY TREATMENT

The investigational medicinal product (IMP) for this study is fenebrutinib.

## 4.3.1 Formulation, Packaging, and Handling

#### 4.3.1.1 Fenebrutinib and Placebo

Fenebrutinib will be provided by the Sponsor as 50-mg dose strength tablets with corresponding matching placebo tablets, which will be indistinguishable in appearance. Study drug (fenebrutinib or placebo) will be dispensed at the Day 1 and 29 visits for both cohorts.

Tablets will be supplied in bottles (Cohort 1) and blister wallets (Cohort 2) for the treatment arm to which the patient is randomly allocated. Each bottle and blister wallet will be labeled per local regulatory requirements. Fenebrutinib and placebo tablets should be stored between 2°C and 8°C. Please refer to the pharmacy manual for detailed instructions on study drug storage and preparation.

For information on the formulation and handling of fenebrutinib, see the Fenebrutinib Investigator's Brochure.

# 4.3.1.2 Background Therapy: Standard-of-Care H1 Antihistamines for CSU

For information on the formulation, packaging, and administration of standard-of-care H1 antihistamines for CSU, see local prescribing information.

# 4.3.2 <u>Dosage, Administration, and Compliance of Fenebrutinib and</u> Placebo

### 4.3.2.1 Fenebrutinib and Placebo Dose and Administration

For Cohort 1, the fenebrutinib dose level is 200 mg (4 tablets) BID (total of 8 tablets each day) with matching placebo (see Section 3.1). For Cohort 2, the fenebrutinib dose levels are 50 mg QD, 150 mg QD, and 200 mg BID, with matching placebos (see Table 3).

Patients in both cohorts will take fenebrutinib/placebo on Day 1 and ending on the Day 56 visit. Although the Day 57 visit is the last day of the study treatment period, no study drug for Study GS39684 will be given on the Day 57 visit. If eligible, patients may enroll into the OLE Study GS40868 to receive their first open-label dose of fenebrutinib on Day 1 of the OLE or they will proceed and return for the safety follow-up visit 4 weeks after the last dose of study drug. For patients enrolling into the OLE, Day 1 of Study GS40868 may be the same day as the Day 57 visit in Study GS39684.

For mandatory morning clinic visits (see Appendix 1 and Section 4.4.5), patients should be instructed that the morning dose of study drug will be taken in the clinic. On other clinic visit days, if the visit occurs in the morning, the patient should be instructed that the morning dose of study drug will be taken in the clinic.

Table 3 Fenebrutinib Dosing Regimen by Treatment Arm (Cohort 2)

| | Number of Tablets | |
|---|---|---|
| Fenebrutinib Dose Arm | Fenebrutinib<br>(a.m./p.m.) | Placebo<br>(a.m./p.m.) |
| 50 mg QD | 1/0 | 3/4 |
| 150 mg QD | 3/0 | 1/4 |
| 200 mg BID | 4/4 | 0/0 |
| Placebo | 0/0 | 4/4 |

BID=twice daily; QD=once daily.

Fenebrutinib or placebo may be taken orally with or without food, except on certain days (see Appendix 1), when the morning dose of oral study drug will be administered at the morning (mandatory) clinic visit while fasting. The dates and times of the most recent prior meal, last dose of oral study drug (prior to clinic visit), and timing of oral study drug administration in clinic should be recorded at each clinic visit. Patients should be instructed that a missed dose should not be taken with the next scheduled dose.

In addition, any antacids (e.g., Pepto-Bismol<sup>®</sup>, Rolaids<sup>®</sup>) should be recorded as concomitant medications, including date and time of last administration. Administration of study drug should be staggered with antacid use (i.e., study drug should be taken 2 hours before or 2 hours after the antacid).

At the Day 1 and 29 visits, sufficient study medication tablets will be dispensed to complete dosing until the end of the study. When study medication is administered at the site, it will be administered under supervision of study personnel, and the amount of study medication dispensed must be recorded.

#### 4.3.2.2 Fenebrutinib and Placebo Compliance

The following measures will be taken to assess patient compliance with study drug. For Cohort 1, patients will be directed to bring the study drug bottle to each visit after randomization. In addition, sites will be responsible for prepopulating the dates on the dosing label (affixed to the bottle) for when patients are scheduled to take study drug. The patients will record the times (a.m. or p.m.) that they take each dose in their eDiary. The number of tablets issued minus the number of tablets returned will be used to calculate the number of tablets taken and compliance.

For Cohort 2, sites will be responsible for prepopulating the dates on the blister wallets for when patients are scheduled to take study drug. The patients will record the times (a.m. or p.m.) that they take each dose in their eDiary. Patients will be instructed to return all blister wallets (used and unused) at each study visit for assessment of compliance and for medication disposal.

Compliance will be documented on the source record. Any overdose or incorrect administration of study drug should be noted on the Study Drug Administration electronic

Case Report Form (eCRF). Adverse events associated with an overdose or incorrect administration of study drug should be recorded on the Adverse Event eCRF. If compliance is  $\leq$  80%, the investigator or designee is to counsel the patient and ensure steps are taken to improve compliance.

# 4.3.2.3 Background Therapy: Standard-of-Care H1 Antihistamines for CSU

The following H1 antihistamine medications are allowed:

- Cetirizine 10–40 mg QD
- Levocetirizine 5-20 mg QD
- Fexofenadine 180–720 mg QD
- Loratadine 10-40 mg QD
- Desloratadine 5-20 mg QD
- Rupatadine 10–40 mg QD
- Bilastine 20–80 mg QD

All patients will be allowed to take study-defined, second-generation, H1 antihistamine medications consistent with standard-of-care (i.e., up to 4 times the approved dose per local treatment guidelines) during the screening, treatment, and follow-up periods. Patients should remain on a stable H1 antihistamine regimen throughout the study period. Loratadine (10 mg) or cetirizine (10 mg) will be provided and used on an as-needed basis (maximum 1 per day) during screening, treatment, and follow-up periods). Therapies used for the treatment of CSU prior to enrollment will be collected as part of the patient's medical history.

Patients taking either LTRAs or H2 blockers for diseases other than CSU (e.g., asthma or gastroesophageal reflux disease, respectively) at screening will be permitted to continue their use at a stable dose during the study. These diseases must be recorded as part of the medical history collected during the screening period. Inhaled asthma controllers, including inhaled corticosteroids, are permitted during the study.

## 4.3.3 Investigational Medicinal Product Accountability

All IMPs required for completion of this study (fenebrutinib and placebo) will be provided by the Sponsor where required by local health authority regulations. The study site will acknowledge receipt of IMPs using the IxRS to confirm the shipment condition and content. Any damaged shipments will be replaced.

IMPs either will be disposed of at the study site according to the study site's institutional standard operating procedure or will be returned to the Sponsor with the appropriate documentation. The site's method of IMP destruction must be agreed to by the Sponsor. The site must obtain written authorization from the Sponsor before any IMP is destroyed, and IMP destruction must be documented on the appropriate form.

Accurate records of all IMPs received at, dispensed from, returned to, and disposed of by the study site should be recorded on the Drug Inventory Log.

## 4.3.4 <u>Post-Trial Access to Fenebrutinib</u>

Patients may be eligible to receive fenebrutinib as part of open-label extension study (GS40868) offered by the Sponsor (Genentech, a member of the Roche Group), as described in Section 3.1.2. The Roche Global Policy on Continued Access to Investigational Medicinal Product is available at the following website:

http://www.roche.com/policy continued access to investigational medicines.pdf

#### 4.4 CONCOMITANT THERAPY AND ADDITIONAL RESTRICTIONS

Concomitant therapy includes any medication (e.g., prescription drugs, over-the-counter drugs, vaccines, herbal or homeopathic remedies, nutritional supplements) used by a patient from 14 days prior to initiation of study drug to the study completion/ discontinuation visit. All such medications (*including standard-of-care H1 antihistamines for CSU*) should be reported to the investigator and recorded on the Concomitant Medications eCRF.

## 4.4.1 <u>Permitted Therapy</u>

Patients who use oral contraceptives, hormone-replacement therapy, or other maintenance therapy should continue their use. All concomitant medications should be reported to the investigator and recorded on the appropriate eCRF. Patients will be encouraged to use the minimal dose required to control their symptoms.

For the purposes of this study, dietary supplements are defined as vitamins, minerals, purified food substances, and herbals with pharmaceutical properties.

Vitamins, minerals, and purified food substances are allowed in amounts not known to be associated with adverse effects (e.g., hypervitaminosis). Herbals with pharmaceutical properties are allowed only if there is acceptable evidence of no CYP3A inhibition or induction (refer to Section 4.4.3 for a list of prohibited concomitant medications, including herbal products). Otherwise, herbals with pharmaceutical properties must be discontinued for at least 4 weeks prior to the first dose of study medication, unless there are sufficient data available regarding the duration of an herbal medication's PK and PD effects to allow a shorter washout to be specified (e.g., 5 half-lives). Please direct any questions to the Medical Monitor.

## 4.4.2 <u>Cautionary Therapy</u>

## 4.4.2.1 Acid-Reducing Agents

Patients who use antacids (e.g., Pepto-Bismol<sup>®</sup>, Rolaids<sup>®</sup>) for symptomatic relief of heartburn should take fenebrutinib or matching placebo at least 2 hours before or 2 hours after antacid administration because gastric acid improves fenebrutinib absorption.

Patients may be treated with PPIs or H2RAs at up to the maximum recommended dose according to local labeling. The dose should remain stable for at least the 2 weeks before randomization and throughout the study.

At visits with scheduled PK assessments (see Appendix 1), any use of PPIs, H2RAs, and/or other antacids (e.g., Pepto-Bismol<sup>®</sup>, Rolaids<sup>®</sup>) should be recorded as concomitant medications, including the date and time of last administration.

#### 4.4.2.2 Statins

Several lipid-lowering agents (statins) are metabolized by CYP3A (simvastatin, lovastatin) and/or transported by BCRP (rosuvastatin, atorvastatin), and thus may be affected by drug-drug interaction with fenebrutinib, therefore, dose adjustments of these medications should be considered (Kellick et al. 2014).

- Simvastatin: recommended maximum dose of 10 mg/day
- Lovastatin: recommended maximum dose of 20 mg/day
- Rosuvastatin: recommended maximum dose of 10 mg/day
- Atorvastatin: recommended maximum dose of 20 mg/day

The use of statins has been associated with myopathy, which can manifest as weakness, tenderness or muscle pain with elevations of creatine kinase (CK) above ten times the ULN. In severe cases, myopathy can cause rhabdomyolysis with or without acute kidney injury secondary to myoglobinuria, and rare fatalities due to rhabdomyolysis have occurred. The risk of myopathy is increased by elevated plasma levels of statins. Predisposing factors for myopathy include advanced age ( $\geq$ 65 years), female gender, uncontrolled hypothyroidism, renal impairment, or the use of concomitant medications that increase the plasma levels of the statin.

## 4.4.2.3 CYP3A and BCRP-Mediated Drug Interactions

Preliminary data from a clinical drug-drug interaction study (Study GP39616) suggest that fenebrutinib can be classified as a mild inhibitor of CYP3A at clinically relevant doses. It is possible that fenebrutinib inhibition of CYP3A may alter the metabolism of CYP3A substrates and result in increased plasma concentrations of CYP3A substrates. Therefore, medications in the following categories (listed in detail in Appendix 5) should be used with caution in consultation with the Medical Monitor (or delegate) as necessary unless otherwise specified in Appendix 5:

- Sensitive CYP3A substrates
- CYP3A substrates with a narrow therapeutic window

The use of hormone-replacement therapy or hormonal contraceptives containing the CYP3A substrate ethinylestradiol (with the concomitant use of a barrier method) is permitted; however, these agents should be used with caution, and patients should be counseled regarding the potential risks and benefit of these medications per the local prescribing information. *Ethinyl estradiol is metabolized by CYP3A so plasma* 

concentrations of ethinyl estradiol are expected to increase in the presence of fenebrutinib (Zhang et al. 2007, Wang et al. 2004). Ethinyl estradiol is not a sensitive substrate of CYP3A (Drug Development and Drug Interactions: Table of Substrates, Inhibitors and Inducers, www.fda.gov). Therefore, the magnitude of increase in ethinyl estradiol plasma concentrations is expected to be less than the increase observed in midazolam concentrations (i.e., less than 2-fold) in Study GP39616, a drug-drug interaction study evaluating the effect of fenebrutinib on the PK of the sensitive CYP3A substrate midazolam. Minor increases in ethinyl estradiol concentrations are not generally associated with adverse events (e.g., Ortho Tri-Cyclen® USPI). Ethinyl estradiol efficacy is expected to be maintained, and ethinyl estradiol continues to be considered a reliable and effective form of contraception in combination with fenebrutinib.

Preliminary data from Study GP39616 also suggest that fenebrutinib can be classified as a moderately sensitive substrate of CYP3A at clinically relevant doses. There is a moderate potential for a drug-drug interaction with any medication that strongly inhibits or induces this enzyme. Therefore, medications in the following categories (listed in detail in Appendix 5) should be avoided for 7 days or 5 half-lives, whichever is longer, prior to the first dose of study drug and until the last dose of study drug. If use of one of these medications is necessary, the risks and benefits should be discussed with the Medical Monitor (or delegate) prior to concomitant administration with study drug:

- Strong CYP3A inhibitors
- Moderate or strong CYP3A inducers

Lastly, preliminary data from Study GP39616 suggest that fenebrutinib is a moderate inhibitor of the breast cancer resistance protein (BCRP) (also known as ABCG2) transporter protein at clinically relevant doses. There is a potential for increased plasma concentrations of drugs that are known to be substrates of the BCRP transporter. Plasma concentrations of the medications in the following category (listed in detail in Appendix 5) may increase; therefore, they should be used with caution in consultation with the Medical Monitor (or delegate) as necessary unless otherwise specified in Section 4.4.1.

The medications listed above and in Section 4.4.1 are not necessarily comprehensive. Thus, the investigator should consult the prescribing information for any concomitant medication as well as the Internet references provided below when determining whether a certain medication is metabolized by or strongly inhibits or induces CYP3A. The investigator should contact the Medical Monitor if questions arise regarding medications not listed above.

https://www.fda.gov/Drugs/DevelopmentApprovalProcess/DevelopmentResources/DrugInteractionsLabeling/ucm093664.htm (Tables 3-1, 3-2, 3-3, and 5-1)

http://medicine.iupui.edu/clinpharm/ddis/table.aspx

## 4.4.3 Prohibited Therapy

Prior to the screening visit (Day –14 for both cohorts) as specified below, and during the study (not including the safety follow-up period if patient failed additional H1 antihistamine for worsened symptoms; see Section 3.1) the following medications and treatments will be restricted. Patients who receive these medications <u>as therapy for CSU</u> will be discontinued from the study treatment but will be followed for safety evaluation:

- Systemic or topical corticosteroids (prescription or over the counter), hydroxychloroquine, methotrexate, cyclosporine, or cyclophosphamide within 30 days prior to screening if used routinely (daily or every other day during 5 or more consecutive days) – The use of corticosteroids may be used for exacerbations
- Doxepin within 30 days prior to screening
- Omalizumab or other monoclonal antibody therapies used to treat CSU within 4 months prior to screening
- IVIG within 30 days prior to screening
- Plasmapheresis within 30 days prior to screening
- LTRAs within 1 day prior to screening
- Astemizole, terfenadine, and ebastine within 1 day prior to screening

#### 4.4.3.1 Live or Attenuated Vaccinations

Immunization with a live or attenuated vaccine is prohibited within 6 weeks prior to study drug administration on Day 1 and for the duration of study participation, including the 4-week safety follow-up period after the administration of the last dose. See Section 5 for further details and precautions around vaccinations.

#### 4.4.4 Prohibited Food

Use of the following foods is prohibited during the study and for at least 7 days prior to initiation of study treatment: furanocoumarin derivatives as found in grapefruit, Seville orange, pomegranate, or star fruit juice or products. Please refer to Appendix 5 for additional information.

# 4.4.5 Additional Restrictions

Patients in both cohorts should be fasting overnight for >8 hours prior to the PK draw and/or fasting lipid panel on Days 1, 8, 29, 57, and 85 (see Appendix 1).

#### 4.5 STUDY ASSESSMENTS

Please see Appendix 1 for the schedule of activities to be performed during the study.

## 4.5.1 Informed Consent Forms and Screening Log

Written informed consent for participation in the study must be obtained before performing any study-related procedures. Informed Consent Forms for enrolled patients and for patients who are not subsequently enrolled will be maintained at the study site.

All screening evaluations must be completed and reviewed to confirm that patients meet all eligibility criteria before enrollment. The investigator will maintain a screening log to record details of all patients screened and to confirm eligibility or record reasons for screening failure, as applicable.

## 4.5.2 Eligibility at Screening

At screening, patients who fail to meet any laboratory inclusion/exclusion criteria or other eligibility criteria may be retested or re-screened as per the instructions in Section 4.5.2.1 and Section 4.5.2.2, respectively.

# 4.5.2.1 Retesting: Laboratory Inclusion/Exclusion

If a patient does not meet certain laboratory inclusion/exclusion criteria at screening, the investigator may repeat the tests once within the screening period (see Section 4.1.2 for laboratory tests and levels that can be retested). If the patient meets the laboratory eligibility criteria on the second assessment, he or she will be permitted to enter the study. It will not be considered a retesting if blood samples have to be redrawn because of sample handling problems, breakage, sample integrity, or laboratory error.

#### 4.5.2.2 Re-screening

Re-screening refers to repeating the entire screening process. Re-screening is required if a patient has not met eligibility criteria within the original screening visit. (Note: patients who have failed two laboratory testing attempts as described in Section 4.1.2 cannot be re-screened). Patients are allowed to be re-screened only once *per cohort*. Each patient must be re-consented before re-screening occurs. It will not be considered a re-screening if blood samples have to be redrawn because of sample handling problems, breakage, sample integrity, or laboratory error.

#### 4.5.3 <u>Medical History and Demographic Data</u>

Comprehensive medical and surgical history, including a comprehensive review of the patient's CSU medical history, will be collected at the Day –14 visit for both cohorts. This review will include onset of symptoms, date of diagnosis, and therapies received for CSU. In addition, history of omalizumab (Xolair®) use and reason for discontinuation will be collected.

Concomitant medical usage will be collected at all visits, including unscheduled visits. Demographic data will include age, sex, and self-reported race/ethnicity.

## 4.5.4 Physical Examinations

A complete physical examination should be performed at the Day –14 visit for both cohorts and should include an evaluation of the head, eyes, ears, nose, and throat, and the cardiovascular, dermatological, musculoskeletal, respiratory, GI, genitourinary, and neurological systems. Any abnormality identified at baseline should be recorded on the General Medical History and Baseline Conditions eCRF.

Subsequent examinations may be limited to detect changes in symptoms of CSU as well as directed by patient complaints regarding adverse events. Changes from baseline abnormalities should be recorded in patient notes. New or worsened clinically significant abnormalities should be recorded as adverse events on the Adverse Event eCRF.

# 4.5.5 <u>Vital Signs</u>

Vital signs will include measurements of heart rate, systolic and diastolic blood pressure while the patient is in a seated position, and temperature. Vital signs will be assessed as outlined in the Schedule of Activities in Appendix 1 and during other unscheduled study visits when clinically indicated. The patients' height and weight will be measured once during the screening visit for both cohorts.

#### 4.5.6 FricTest

For subjects who have a history of dermographism, a FricTest® will be performed at screening (Day –14), baseline (Day 1), and Days 57 and 85 for both cohorts. The FricTest® is a flat, plastic comb with four round-ended plastic pins, 3 mm in diameter and of different lengths. The FricTest® defines provocation thresholds and severity of dermographism (i.e., 4 pins inducing wheals defines severe dermographism).

# 4.5.7 <u>Laboratory,</u> and Other Biological Samples

Samples for the following laboratory tests will be sent to one or several central laboratories for analysis as per the Schedule of Activities in Appendix 1. Laboratory tests prior to randomization and dosing may be performed locally on Day 0, if central laboratory tests are not available due to sampling handling problems, breakage, or lab error.

- Hematology: hemoglobin, hematocrit, platelet count, RBC count, WBC count, percent and absolute differential counts (neutrophils, bands, lymphocytes, monocytes, eosinophils, basophils, other cells)
- Serum chemistry: sodium, potassium, chloride, bicarbonate, glucose, BUN, creatinine, calcium, phosphorus, magnesium, total and direct bilirubin, total protein, albumin, ALT, AST, LDH, alkaline phosphatase, creatine phosphokinase, CRP, lipase, and uric acid
- Urinalysis including dipstick (pH, specific gravity, glucose, protein, ketones, blood) and microscopic examination (sediment, RBCs, WBCs, casts, crystals, epithelial cells, bacteria)
- Coagulation: INR, activated PTT, PT, fibrinogen
- Fasting lipid panel
- Viral serology
- Hepatitis B: HBsAg, total HBcAb, and hepatitis B surface antibody
- Hepatitis C antibody

- The following samples will be sent to the Sponsor or a designee for analysis:
- Plasma samples for PK analysis
- See the Schedule of Activities provided in Appendix 1 for specific timepoints.
- Samples for the following laboratory tests will be sent to the study site's local laboratory for analysis:
- Pregnancy test

All women of childbearing potential (including those who have had a tubal ligation) will have a serum pregnancy test at screening. Urine pregnancy tests will be performed at specified subsequent visits. If a urine pregnancy test result is positive, it must be confirmed by a serum pregnancy test. Should a positive result be recorded at any time, the procedures detailed in Section 5.4.3 should be followed. If a local urine pregnancy test shows a positive result, then study drug will not be administered that day. Other study procedures should also be postponed and the result must be confirmed by a serum pregnancy test prior to proceeding.

 QFT or PPD (if QFT not available) and additional procedures (e.g., chest X-ray) to rule out latent or active TB per local guidelines

See the Schedule of Activities provided in Appendix 1 for specific timepoints.



For sampling procedures, storage conditions, and shipment instructions, see the laboratory manual.

Biological samples will be destroyed when the final clinical study report (CSR) has been completed, with the following exceptions:

- Plasma samples collected for PK analysis will be destroyed no later than 5 years after the final CSR has been completed.
- Blood, urine, and serum samples collected will be destroyed no later than 15 years after the final CSR has been completed.

When a patient withdraws from the study, samples collected prior to the date of withdrawal may still be analyzed, unless the patient specifically requests that the samples be destroyed or local laws require destruction of the samples. *However, if samples have been tested prior to withdrawal, results from those tests will remain as part of the overall research data.* 

Data arising from sample analysis will be subject to the confidentiality standards described in Section 8.4.

# 4.5.8 <u>Electrocardiograms</u>

A single ECG recording, without artifacts, must be obtained at specified timepoints, as indicated in Appendix 1. The ECG intervals (e.g., PR, QRS, QT, QTcF, and RR) and heart rate from this ECG will be entered into the eCRF. Any morphologic waveform changes or other ECG abnormalities must be documented on the eCRF.

All ECG recordings must be performed using a standard high-quality, high-fidelity digital electrocardiograph machine equipped with computer-based interval measurements. Lead placement should be as consistent as possible. ECGs for each patient should be obtained from the same machine whenever possible. ECG recordings must be performed after the patient has been resting in a supine position for at least 10 minutes prior to beginning the ECG recording. All ECGs can be performed without specific restrictions (e.g., can be performed at any time of day, before or after dosing, fasting or fed) but are to be obtained prior to other procedures scheduled at that same time (e.g., vital sign measurements, blood draws). Body position should be consistently maintained for each ECG evaluation to prevent changes in heart rate. Circumstances that may induce changes in heart rate, including environmental distractions (e.g., television, radio, conversation) should be avoided during the pre-ECG resting period and during ECG recording.

For safety monitoring purposes, the investigator must review, sign, and date all ECG tracings. Paper copies of ECG tracings will be kept as part of the patient's permanent study file at the site. If considered appropriate by the Sponsor, ECGs may be analyzed retrospectively at a central laboratory.

If at a particular post-dose timepoint the mean QTcF is > 500 ms or > 60 ms longer than the baseline value, another ECG must be recorded, ideally within the next 5 minutes, and ECG monitoring should continue until QTcF has stabilized on two successive ECGs.

The Medical Monitor should be notified as soon as possible within 24 hours. Standard-of-care treatment may be instituted per the discretion of the investigator. If a PK sample is not scheduled for that timepoint, an unscheduled PK sample should be obtained. A decision on study drug discontinuation should be made, as described in Section 4.6.2. The investigator should also evaluate the patient for potential concurrent risk factors (e.g., electrolyte abnormalities, co-medications known to prolong the QT interval, severe bradycardia).

## 4.5.9 <u>Patient-Reported Outcomes</u>



Patients will use an electronic device to capture the Urticaria Patient Daily eDiary (see Appendix 3). The electronic device and/or instructions for completing the questionnaires electronically will be provided by the investigator staff. The data will be transmitted to a centralized database maintained by the electronic device vendor. The data will be available for access by appropriate study personnel.



#### 4.5.9.1 Urticaria Patient Daily eDiary

The Urticaria Patient Daily eDiary includes the UAS, which will be used to calculate the UAS7. The eDiary comprises questions regarding largest hive size, sleep interference score, activity interference question, rescue medication use, angioedema episodes, number of calls to doctor or nurse practitioner, and study medication compliance.

The eDiary is to be completed twice per day (a.m./p.m.) by the patient for the duration of the study. The eDiary will be given to the patient at the Day –14 visit for both cohorts.

## 4.5.9.2 Urticaria Activity Score

During the week prior to Day 1 (i.e., Week –1), UAS7 will be recorded twice daily for the purposes of enrollment eligibility for both cohorts. Subsequently, the UAS will be recorded twice daily using the Urticaria Patient Daily eDiary.

The UAS is a composite, eDiary-recorded score with numeric severity intensity ratings (0=none to 3=intense/severe) for a) the number of wheals (hives) and b) the intensity of the pruritus (itch) over the past 12 hours (twice daily; see Section 3.3.6). The daily UAS is calculated as the average of the morning and evening scores. The UAS7 will be calculated and is the weekly sum of the daily UAS, which is the composite score of the intensity of pruritus and the number of wheals. The maximum UAS7 value is 42; the intensity of the itch/pruritus and the number of wheals/hives are graded in Table 2.





# 4.6 PATIENT, TREATMENT, STUDY, AND SITE DISCONTINUATION

#### 4.6.1 <u>Patient Discontinuation</u>

Patients have the right to voluntarily withdraw from the study at any time for any reason. In addition, the investigator must withdraw a patient from the study for the following, but not limited to, reasons:

- Patient withdrawal of consent at any time
- Any medical condition that the investigator or Sponsor determines may jeopardize the patient's safety if he or she continues in the study
- Investigator or Sponsor determines it is in the best interest of the patient
- The investigator may withdraw a patient from the study at any time due to patient non-compliance (e.g., drug compliance ≤ 80%, missed visits, missing Urticaria Patient Daily eDiary entries)

For patients who withdraw from the study, every effort should be made to complete an early termination visit including the assessments on the Schedule of Activities (see Appendix 1). The primary reason for withdrawal from the study should be documented

on the appropriate eCRF. However, patients will not be followed for any reason after consent has been withdrawn. Patients who withdraw from the study will not be replaced.

If the patient discontinues the study prior to Day 85 visit, the patient will be asked to return to the clinic for a safety follow–up visit 4 weeks after the last dose of study drug. Patients who refuse to complete the safety follow–up period should undergo an early termination visit. Patients who discontinue during the safety follow-up period prior to completion of the 4-week safety follow-up will be asked to complete an early termination visit (see Appendix 1).

If a patient withdraws for reasons related to a serious adverse event, every attempt should be made to follow the patient until resolution of the event.

#### 4.6.2 Study Treatment Discontinuation

Patients must discontinue study treatment if they experience any of the following:

- Pregnancy
- Malignancy
- Any serious infection or infection requiring treatment with an IV antimicrobial agent
- Any prohibited medication as defined in Section 4.4.3

Patients who discontinue study treatment prematurely (prior to Day 85 visit), including but not limited to the reasons listed above, will be asked to return to the clinic for a safety follow-up visit 4 weeks after the last dose of study drug. Patients who refuse to complete the safety follow up period should return to the clinic for an early termination visit.

The primary reason for study treatment discontinuation should be documented on the appropriate eCRF. Patients who discontinue study treatment prematurely will not be replaced.

#### 4.6.3 <u>Study and Site Discontinuation</u>

The Sponsor has the right to terminate this study at any time. Reasons for terminating the study include, but are not limited to, the following:

- The Sponsor must terminate the study if the Sponsor believes that the incidence or severity of adverse events in this or other studies indicates a potential health hazard to patients.
- The Sponsor may terminate the study if patient enrollment or completion of the study unsatisfactory.

The Sponsor will notify the investigator if the Sponsor decides to discontinue the study.

The Sponsor has the right to close a site at any time. Reasons for closing a site may include, but are not limited to, the following:

- The Sponsor must close a site if corrective actions to improve site performance in the following areas do not yield significant improvement:
  - Excessively slow recruitment
  - Poor protocol adherence
  - Inaccurate or incomplete data recording
  - Non-compliance with the International Council on Harmonisation (ICH) guideline for Good Clinical Practice
- No study activity (i.e., all patients have completed the study and all obligations have been fulfilled).

## 5. <u>ASSESSMENT OF SAFETY</u>

#### 5.1 SAFETY PLAN

The safety plan for patients in this study is based on nonclinical and clinical experience with fenebrutinib in completed and ongoing studies, as well as published literature, on other BTK inhibitors and BTK biology. The important potential safety risks for fenebrutinib are outlined below. Please refer to the Fenebrutinib Investigator's Brochure for a complete summary of safety information.

Several measures will be taken to ensure the safety of patients participating in this study. Eligibility criteria have been designed to exclude patients at higher risk for potential toxicities. Patients will undergo safety monitoring during the study, including monitoring of vital signs, physical examination, ECGs, and routine laboratory safety assessments (hematology, chemistry, and urinalysis) and assessment of the nature, frequency, and severity of adverse events. In addition, guidelines for managing potential adverse events, including criteria for treatment interruption or discontinuation, and enhanced safety reporting are provided below.

In addition, an unblinded IMC will monitor patient safety throughout the study for Cohort 2 (see Section 3.1.1).

# 5.1.1 Safety Plan for Potential Risks Associated with Fenebrutinib 5.1.1.1 Infections

Fenebrutinib is a reversible inhibitor of BTK, and the degree to which fenebrutinib antagonism of BTK signaling may suppress immune activity is unknown. On the basis of patients with XLA, a primary immunodeficiency *caused by mutations in the BTK gene*, it is anticipated that inhibitors of BTK may raise the risk for certain bacterial infections (Lederman and Winkelstein 1985; Broides et al. 2006), enteroviral infections (Misbah et al. 1992; Ziegner et al. 2002), intestinal infections with giardia and *Campylobacter* species (Winkelstein et al. 2006; van den Bruele et al. 2010), or other opportunistic infections, which are cleared primarily by B-cell adaptive immune

Fenebrutinib (GDC-0853)—Genentech, Inc. 63/Protocol GS39684, Version 4

responses. This risk is likely independent of sex for patients exogenously administered fenebrutinib.

Effects on lymphocytes and immunoglobulins in rats and dogs were reversible and considered to be related to pharmacological activity involving BTK inhibition. See Section 1.2.2 for related primary nonclinical toxicity findings and the Fenebrutinib Investigator's Brochure for further details.

To date, no immune-challenge experiments (e.g., T-dependent antigen response test) have been conducted in animals. It is not known whether these effects on B cells and IgG concentrations in animals will translate to humans or whether such changes would have functional or deleterious impact on immune function.

Infections, including pneumonia and fatal influenza, have occurred in patients with B-cell malignancies treated with fenebrutinib. In studies with healthy subjects with single doses and with dosing for 14 days, self-limited Grade 1 events of nasopharyngitis were reported but did not lead to any change in study drug dosing. One healthy subject had asymptomatic bacteriuria, which resolved while study drug dosing continued. *In blinded and open-label studies in autoimmune indications, serious, severe, and opportunistic infections have been reported, including one case of pulmonary tuberculosis as well as cases of pneumonia, bronchitis, cellulitis, enterobacter infection, herpes zoster, acute pyelonephritis, necrotizing soft tissue infection, colitis, periorbital cellulitis, and sinusitis. As a safety precaution, the study protocol contains exclusion criteria for infections and potential infection risk and guidelines for study drug management in the event of infection. Study subjects and patients should be monitored for fever and potential infectious complications, including opportunistic infections, and evaluated promptly.* 

Patients will be excluded from the study if they have a history of hospitalization due to an infection in the 8 weeks before screening, evidence of active or latent or inadequately treated infection with *Mycobacterium* TB, known active infection (current) or history of recurrent infection, or any known immunodeficiency including IgG < 500 mg/dL.

patients in the study should be monitored for fever and potential infectious complications, including opportunistic infections and TB, and should be evaluated promptly. Physicians or a health care provider should give patients advice to prevent potential transmission of and exposure to endemic infections according to local or Centers for Disease Control and Prevention guidelines. Patients should be advised to seek immediate medical attention if they develop signs and symptoms suggestive of an infection. All infections occurring during the study, including but not limited to respiratory infections, cutaneous infections, urinary tract infections, systemic viral infections, and episodes of suspicious or febrile diarrhea, should be evaluated using serology or polymerase chain reaction, if available, and cultured, if feasible, and any identified organisms noted in the eCRF. Any serious infection, infection requiring IV antimicrobials, or any opportunistic infection is

considered an adverse event of special interest and should be reported to the Sponsor as outlined in Section 5.4.2.

Guidelines for management of study treatment in the event that infections are observed in patients are provided in Section 5.1.2.

Please refer to the Fenebrutinib Investigator's Brochure for further details.

#### 5.1.1.2 Vaccinations

The effect of fenebrutinib upon the efficacy of vaccinations is unknown. It is recommended that appropriate vaccinations per local guidelines be up to date before study participation. Patients will be excluded from study participation and will not be dosed with fenebrutinib if they have been vaccinated with live, attenuated vaccines (e.g., the intranasal live attenuated influenza vaccines, BCG, varicella) within 6 weeks before planned dosing. In addition, immunization with a live or attenuated vaccine is prohibited for the duration of study participation, including the 4-week safety follow-up period after the administration of the last dose.

In addition, current routine household contact with children or others who have been vaccinated with live vaccine components may pose a risk to the patient during study treatment with fenebrutinib. Some of these vaccines include varicella ("chickenpox") vaccine, oral polio vaccine, and the inhaled flu vaccine. Following vaccination with live component vaccines, the virus may be shed in bodily fluids, including stool, and there is a potential risk that the virus may be transmitted to the patient.

General guidelines for immunosuppressed patients suggest that exposure to vaccinated individuals should be avoided following vaccination with these vaccines for the stated time periods:

- Varicella or attenuated typhoid fever vaccination for 4 weeks following vaccination
- Oral polio vaccination for 6 weeks following vaccination
- Attenuated rotavirus vaccine for 10 days following vaccination
- FluMist® (inhaled flu vaccine) for 1 week following vaccination

Please refer to the Fenebrutinib Investigator's Brochure for further details.

#### **5.1.1.3** Bleeding

No decrease in platelets, changes in coagulation parameters, or bleeding events were observed in nonclinical studies with fenebrutinib. Bleeding events, including non-serious NCI CTCAE v4.0 Grade 1 bruising and serious Grade ≥3 GI bleeding, have been reported in patients with hematological malignancies treated with fenebrutinib in Study GO29089. The GI bleeding events have not been dose related, and the events occurred in patients who were taking concomitant NSAIDs and who had a history of gastroesophageal or peptic ulcer disease. The impact of BTK inhibition as a potential risk factor for bleeding is unknown. BTK is expressed in platelets and is involved in

platelet function via GPVI/collagen receptor signaling and GP1b receptor signaling. Platelets from patients with XLA, a genetic deficiency of BTK, demonstrate decreased activation in response to submaximal collagen stimulation but normal response to thrombin; clinically, there is no reported bleeding propensity of patients with XLA.

Bruising or bleeding events related to fenebrutinib have not been reported in healthy subjects. Grade  $\geq 2$  bleeding events have been reported in blinded and open-label studies of fenebrutinib in autoimmune indications, including hematuria, purpura, hematoma, and uterine and vaginal bleeding.

It is unknown whether fenebrutinib will increase the risk of bleeding in patients, especially in those receiving anti-platelet or anticoagulant therapies. As a precautionary safety measure, patients will be excluded from study participation if they have a need for systemic anticoagulation with warfarin or other oral or injectable anticoagulants or anti-platelet agents (other than NSAIDs, aspirin, and other salicylates), any history of hospitalizations or transfusion for a GI bleed, any history of a hemorrhagic CVA, any history of spontaneous intracranial hemorrhage, traumatic intracranial hemorrhage within 10 years prior to the study, or a known bleeding diathesis. Patients should be advised to seek immediate medical attention if they develop signs and symptoms suggestive of clinically significant bleeding.

Bleeding events of moderate or greater severity are considered adverse events of special interest and should be reported to the Sponsor in an expedited manner as outlined in Section 5.4.2.

Guidelines for management of study treatment in the event that bleeding is observed in patients are provided in Section 5.1.2. Please refer to the Fenebrutinib Investigator's Brochure for further details.

### 5.1.1.4 Cytopenias

Cytopenias have been observed in patients with hematological malignancies who received fenebrutinib as well as in the ongoing, blinded Phase II studies and OLEs in autoimmune diseases. Cytopenias have included neutropenia, anemia, and thrombocytopenia; events have been monitorable and clinically manageable (see the Fenebrutinib Investigator's Brochure for further details).

Patients should be monitored regularly with hematology laboratory evaluations as outlined in the schedule of activities (see Appendix 1) and should receive appropriate supportive care as clinically indicated. Patients should be advised to seek immediate medical attention if they develop signs and symptoms suggestive of cytopenias (e.g., persistent fever, bruising, bleeding, pallor). Cytopenias should be managed according to local clinical guidelines.

Guidelines for managing study treatment in the event that cytopenia is observed are provided in Section 5.1.2. Please refer to the Fenebrutinib Investigator's Brochure for further details.

#### 5.1.1.5 Gastrointestinal Effects

Body weight gain and food consumption changes have been observed in animals, including nonsignificant increases in male Wistar-Han rats administered  $\geq 2$  mg/kg/day (4.3  $\mu\text{M} \bullet \text{hr})$  for 6 months, and significant reductions in rats administered 100 mg/kg/day (1438  $\mu\text{M} \bullet \text{hr})$  and dogs administered 25 mg/kg (180  $\mu\text{M} \bullet \text{hr})$  for 4 weeks. These effects on body weight gain and food consumption were reversible following discontinuation of fenebrutinib dosing.

NCI CTCAE v4.0 Grade 1 diarrhea, nausea, and abdominal pain have been reported in patients with B-cell malignancies; however, the events have resolved and have not led to study drug discontinuation. Healthy subjects in the MAD Study GA29347 reported events of mild self-limited nausea. *Across studies with immune indications receiving blinded or open-label treatment, approximately 5% of enrolled patients have reported nausea, vomiting, diarrhea, or other gastrointestinal symptoms.* 

Throughout the study, patients will be monitored for GI side effects.

Guidelines for management of study treatment in the event of GI side effects in patients are provided in Section 5.1.1.5. Please refer to the Fenebrutinib Investigator's Brochure for further details.

#### 5.1.1.6 Hepatotoxicity

Evidence of hepatobiliary injury was observed in animals administered relatively high doses of fenebrutinib in repeat-dose toxicity studies. Dose-dependent increases in ALT, AST, and/or bilirubin have been observed in rats administered  $\geq 6$  mg/kg/day ( $\geq 17~\mu\text{M} \cdot \text{hr}$ ) and dogs administered  $\geq 10$  mg/kg/day ( $\geq 36~\mu\text{M} \cdot \text{hr}$ ), with corresponding microscopic changes in the liver of dogs administered 25 mg/kg/day (180  $\mu\text{M} \cdot \text{hr}$ ). The hepatotoxicity findings in dogs were associated with moribundity in two high-dose animals. The NOAEL for these findings was considered to be 10 mg/kg (36  $\mu\text{M} \cdot \text{hr}$ ) in dogs, the most sensitive species, given the absence of fenebrutinib–related hepatotoxicity at this dose when administered for 9 months.

The hepatotoxicity findings were fully reversible and considered monitorable by changes in plasma transaminases and bilirubin that occurred at doses lower than those producing histopathology findings (see the Fenebrutinib Investigator's Brochure for further details).

In clinical studies in autoimmune indications, including in patients with CSU, cases of Grade 3 (or severe) transaminase elevations, including cases that were considered serious by the investigator have been reported. These transaminase elevations have occurred in both the randomized clinical studies, which remain blinded to the Sponsor

in terms of treatment assignment, and the open-label extension. The transaminase levels returned to normal after discontinuation of the study treatment. There have been no observed AEs of liver enzyme elevation in clinical studies to date in healthy subjects or patients with hematological malignancies. To date, no cases of transaminase elevations have led to clinical jaundice or bilirubin >2 × ULN (Hy's Law). All transaminase elevations have been reversible when dosing of blinded study medication/placebo was withheld.

As a safety risk-mitigation measure, to be eligible for the study, AST and/or ALT levels should be no more than 1.5×ULN, and total bilirubin levels should be normal at screening. Safety monitoring for potential hepatotoxicity includes baseline and routine evaluations of AST/ALT and total bilirubin levels throughout the study as outlined in the schedule of activities (see Appendix 1).

Laboratory results of either an AST or ALT  $> 5 \times$  ULN or an AST or ALT  $> 3 \times$  ULN in combination with a total bilirubin  $> 2 \times$  ULN, of which at least 35% is direct bilirubin or there is clinical jaundice, are considered adverse events of special interest and should be reported to the Sponsor in an expedited manner as outlined in Section 5.4.2.

Guidelines for the management of study treatment in the event of hepatotoxicity in patients are provided in Section 5.1.2. Please refer to the Fenebrutinib Investigator's Brochure for further details.

#### 5.1.1.7 Cardiovascular Effects

Fenebrutinib is considered to have a low potential to cause QT interval prolongation or to directly affect other cardiovascular parameters, at therapeutic exposures. A minimal increase in QTc (7 ms or 3%) interval was noted at 45 mg/kg in the single-dose cardiovascular safety pharmacology study in telemetry-instrumented dogs.

There

have been no fenebrutinib-related changes in ECG parameters in the 4-week or 9-month dog toxicity studies.

Analysis of ECG data from the SAD and MAD studies in healthy subjects did not demonstrate any significant increase in either QRS interval or QTcF intervals. However, cardiac safety will be evaluated in all patients at baseline and throughout this study, with routine monitoring of vital signs (including heart rate and blood pressure), routine safety ECGs, and collection of adverse events (see Section 5.1.1.7 and Section 5.2.1).

Management of patients with sustained QTcF prolongation (QTcF that is >500 ms or >60 ms longer than the baseline value) should include recording another ECG, ideally within the next 5 minutes, and ECG monitoring should continue until QTcF has stabilized on two successive ECGs. The Medical Monitor should be notified as soon as possible within 24 hours. Standard-of-care treatment may be instituted per the discretion of the

investigator. If a PK sample is not scheduled for that timepoint, an unscheduled PK sample should be obtained. A decision on study drug discontinuation should be made, as described in Section 4.6.2. The investigator should also evaluate the patient for potential concurrent risk factors (e.g., electrolyte abnormalities, co-medications known to prolong the QT interval, severe bradycardia).

Guidelines for management of study treatment in the event in the event of cardiovascular effects in patients are provided in Section 5.1.2. Please refer to the Fenebrutinib Investigator's Brochure for further details.

#### 5.1.1.8 Vascular Inflammation

Vascular inflammation (vasculitis) was observed in dogs administered fenebrutinib at  $\geq$  10 mg/kg/day ( $\geq$  56  $\mu$ M • hr) in the 4-week toxicity study, and these changes were not completely reversed by the end of the 4-week recovery period. There was no consistent correlation with any clinical biomarkers. However, in the 9-month toxicity study in dogs, no fenebrutinib–related vascular inflammation was observed up to the highest dose of 10 mg/kg/day (36  $\mu$ M • hr), which is considered to be the NOAEL (AUC) for the canine vascular inflammation findings.

The translatability of

these findings to humans is unknown; however, Beagle dogs are susceptible to spontaneous development of polyarteritis syndrome (Snyder et al. 1995) and may be more sensitive to any drug-induced effects. Further, there are several examples of approved therapies for which there is no correlation between the finding of vasculitis in dogs or rats at clinically relevant exposures and adverse outcomes in patients (FDA 2011). Guidelines for management of study treatment in the event of vasculitis in patients are provided in Section 5.1.2. Please refer to the Fenebrutinib Investigator's Brochure for further details.

#### 5.1.1.9 Malignancy

The impact of BTK inhibition on the development of malignancies is not known; however, malignancies have been identified as a potential concern for immunomodulatory agents. Malignancies have been reported in patients with XLA, including lymphoreticular malignancies, gastric and colorectal adenocarcinoma, and squamous cell carcinoma of the lung.

Patients with a history of cancer, including hematologic malignancy and solid tumors, within 10 years before screening will be excluded from the study. Basal or squamous cell carcinoma of the skin that has been excised and is considered cured and in situ carcinoma of the cervix treated with apparent success by curative therapy more than 1 year prior to screening are not exclusionary.

All malignancies are adverse events of special interest and should be reported to the Sponsor in an expedited manner as outlined in Section 5.2.3.

Guidelines for management of study treatment in the event of malignancies in patients are provided in Section 5.1.2. Please refer to the Fenebrutinib Investigator's Brochure for further details.

# 5.1.2 <u>Management of Patients Who Experience Specific Adverse Events</u>

# **5.1.2.1 Management of Specific Adverse Events**

Guidelines for management of specific adverse events are outlined in Table 5.

Table 5 Guidelines for Management of Patients Who Experience Specific Adverse Events

| Event | Action to be Taken <sup>a</sup> |
|---|---|
| Infection <sup>b</sup> | |
| Serious infection, opportunistic infection, or any infection requiring treatment with an IV antimicrobial agent | Discontinue study treatment and report event as an adverse event of special interest. |
| Self-limited infections that require treatment | Withhold study treatment during antimicrobial therapy. Study treatment may resume after consultation with the Medical Monitor. |
| Bleeding | Bleeding events of moderate or greater severity are considered adverse events of special interest and should be reported to the Sponsor in an expedited manner. |
| | For serious bleeding events or bleeding events requiring transfusion, radiologic endoscopic, or elective operative intervention, withhold study treatment and consult with the Medical Monitor. |
| Gastrointestinal effects | |
| Nausea, vomiting, and/or diarrhea | Manage according to site institutional guidelines. |
| | Consider administration of study treatment with food as a possible mitigation strategy. |
| Malignancy | |
| Any malignancy | Discontinue study treatment, with the exception of non-serious local and resectable basal or squamous cell carcinoma of the skin. Report event as an adverse event of special interest to the Sponsor in an expedited manner. |
| Hepatotoxicity | |
| AST or ALT 3.0-5.0 × ULN | Withhold study treatment and consult with the Medical Monitor. |
| AST or ALT > 3 × ULN in combination with a total bilirubin > 2 × ULN, of which at least 35% is direct bilirubin, or clinical jaundice | Discontinue study treatment. Report event(s) as adverse event of special interest (Hy's law) to the Sponsor in an expedited manner. |

Table 5 Guidelines for Management of Patients Who Experience Specific Adverse Events (cont.)

| Event | Action to be Taken <sup>a</sup> |
|---|---|
| AST or ALT > 5 × ULN | Discontinue study treatment. Any elevation of an AST or ALT $> 5 \times$ ULN should be reported as an adverse event of special interest to the Sponsor in an expedited manner. |
| Cardiovascular effects | |
| Sustained (at least two ECG measurements > 30 minutes apart) QTcF that is > 500 ms or > 60 ms longer than the baseline value | Unless there is a clear alternative cause other than study drug, discontinue study treatment. c |
| Sustained absolute QTcF that is > 515 ms | Unless there is a clear alternative cause other than study drug, discontinue study treatment. ° |
| An episode of torsades de pointes or a new ECG finding of clinical concern | Unless there is a clear alternative cause other than study drug, discontinue study treatment. ° |
| Vascular inflammation | |
| Vasculitis | Discontinue study treatment and consult with the Medical Monitor. |

IV = intravenous; QTcF = QT interval corrected using Fridericia's formula; ULN = upper limit of normal. Note: "Study treatment" includes study drug (fenebrutinib or placebo).

- <sup>a</sup> Any patient who discontinues study treatment should enter safety follow-up, if possible.
- <sup>b</sup> Appropriate laboratory investigations, including but not limited to cultures, should be performed to establish the etiology of any serious infection.
- <sup>c</sup> In rare circumstances, it may be acceptable to resume study drug, provided that any ECG abnormalities have resolved and that the patient is appropriately monitored. Clinical judgment should be applied.

#### 5.1.2.2 Management of Increases in QT Interval

Study drug should be discontinued in patients who develop any of the following:

- Sustained (at least two ECG measurements > 30 minutes apart) QTcF that is
   > 500 ms or > 60 ms longer than the baseline value
- Sustained absolute QTcF that is > 515 ms
- An episode of torsades de pointes or a new ECG finding of clinical concern

Of note, if there is a new intraventricular conduction block, the increase in QRS complex duration should be subtracted from the QTcF change, because this represents an increase in QTcF unrelated to alterations in repolarization. Also of note, it is not uncommon to record arrhythmias, such as non-sustained ventricular tachycardia, supraventricular tachycardia, pauses, or atrial fibrillation, in healthy volunteers receiving placebo during periods of extended ECG monitoring. Therefore, it is critical that expert cardiology advice be sought to confirm any ECG changes and to ascertain the likelihood of a drug-induced arrhythmia versus the background occurrence of this arrhythmia. In such a situation, saving all available ECG data is highly suggested.
Management of patients with sustained QTcF prolongation should include close monitoring, with ECGs repeated at least hourly until two successive ECGs show resolution of the findings, correction of any electrolyte abnormalities, and possible discontinuation of other concomitant medications that are known to prolong the QT interval. Consultation with a cardiologist or electrophysiologist is recommended to help in the management of such patients.

#### 5.2 SAFETY PARAMETERS AND DEFINITIONS

Safety assessments will consist of monitoring and recording adverse events, including serious adverse events and adverse events of special interest, performing protocol-specified safety laboratory assessments, measuring protocol-specified vital signs, and conducting other protocol-specified tests that are deemed critical to the safety evaluation of the study.

Certain types of events require immediate reporting to the Sponsor, as outlined in Section 5.4.

#### 5.2.1 Adverse Events

According to the ICH guideline for Good Clinical Practice, an adverse event is any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product, regardless of causal attribution. An adverse event can therefore be any of the following:

- Any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product
- Any new disease or exacerbation of an existing disease (a worsening in the character, frequency, or severity of a known condition), except as described in Section 5.3.5.10
- Recurrence of an intermittent medical condition (e.g., headache) not present at haseline
- Any deterioration in a laboratory value or other clinical test (e.g., ECG, X-ray) that is associated with symptoms or leads to a change in study treatment or concomitant treatment or discontinuation from study drug
- Adverse events that are related to a protocol-mandated intervention, including those that occur prior to assignment of study treatment (e.g., screening invasive procedures such as biopsies)

# 5.2.2 <u>Serious Adverse Events (Immediately Reportable to the Sponsor)</u>

A serious adverse event is any adverse event that meets any of the following criteria:

• Is fatal (i.e., the adverse event actually causes or leads to death)

- Is life threatening (i.e., the adverse event, in the view of the investigator, places the patient at immediate risk of death)
  - This does not include any adverse event that had it occurred in a more severe form or was allowed to continue might have caused death.
- Requires or prolongs inpatient hospitalization (see Section 5.3.5.11)
- Results in persistent or significant disability/incapacity (i.e., the adverse event results in substantial disruption of the patient's ability to conduct normal life functions)
- Is a congenital anomaly/birth defect in a neonate/infant born to a mother exposed to study drug
- Is a significant medical event in the investigator's judgment (e.g., may jeopardize the
  patient or may require medical/surgical intervention to prevent one of the outcomes
  listed above)

The terms "severe" and "serious" are <u>not</u> synonymous. Severity refers to the intensity of an adverse event (e.g., rated as mild, moderate, or severe; see Section 5.3.3); the event itself may be of relatively minor medical significance (such as severe headache without any further findings).

Severity and seriousness need to be independently assessed for each adverse event recorded on the eCRF.

Serious adverse events are required to be reported by the investigator to the Sponsor immediately (i.e., no more than 24 hours after learning of the event; see Section 5.4.2 for reporting instructions).

# 5.2.3 <u>Adverse Events of Special Interest (Immediately Reportable to the Sponsor)</u>

Adverse events of special interest are required to be reported by the investigator to the Sponsor immediately (i.e., no more than 24 hours after learning of the event; see Section 5.4.2 for reporting instructions). Adverse events of special interest for this study include the following:

- Any serious infection, any infections requiring IV antimicrobials and any opportunistic infections
- Bleeding events of moderate or greater severity
- All malignancies
- Adverse events of special interest for general drug development
  - A laboratory result of AST or ALT > 5 × ULN
  - Cases of potential drug-induced liver injury that include an ALT or AST > 3 × ULN in combination with a total bilirubin > 2 × ULN, of which at least 35% is direct bilirubin or there is clinical jaundice, as defined by Hy's law (see Section 5.1.1.6)

Suspected transmission of an infectious agent by the study drug, as defined below:
 Any organism, virus, or infectious particle (e.g., prion protein transmitting transmissible spongiform encephalopathy), pathogenic or non-pathogenic, is considered an infectious agent. A transmission of an infectious agent may be suspected from clinical symptoms or laboratory findings that indicate an infection in a patient exposed to a medicinal product. This term applies only when a contamination of the study drug is suspected.

# 5.3 METHODS AND TIMING FOR CAPTURING AND ASSESSING SAFETY PARAMETERS

The investigator is responsible for ensuring that all adverse events (see Section 5.2.1 for definition) are recorded on the Adverse Event eCRF and reported to the Sponsor in accordance with instructions provided in this Section and in Section 5.4 – Section 5.6.

For each adverse event recorded on the Adverse Event eCRF, the investigator will make an assessment of seriousness (see Section 5.2.2), severity (see Section 5.3.3), and causality (see Section 5.3.4).

### 5.3.1 Adverse Event Reporting Period

Investigators will seek information on adverse events at each patient contact. All adverse events, whether reported by the patient or noted by study personnel, will be recorded in the patient's medical record and on the Adverse Event eCRF.

**After informed consent** has been obtained **but prior to initiation of study drug**, only serious adverse events caused by a protocol-mandated intervention (e.g., invasive procedures such as biopsy sample collection, discontinuation of medications) should be reported (see Section 5.4.2 for instructions for reporting serious adverse events).

**After initiation of study drug**, all adverse events will be reported until 4 weeks after the last dose of study drug the patients receives. After this period, the investigator should report any serious adverse events that are believed to be related to prior study drug treatment (see Section 5.4.2).

#### 5.3.2 Eliciting Adverse Event Information

A consistent methodology of non-directive questioning should be adopted for eliciting adverse event information at all patient evaluation timepoints. Examples of non-directive questions include the following:

"How have you felt since your last clinic visit?"

"Have you had any new or changed health problems since you were last here?"

#### 5.3.3 Assessment of Severity of Adverse Events

Table 6 provides the adverse event grading scale for severity.

Table 6 Adverse Event Severity Grading Scale

| Severity | Description |
|---|---|
| Mild | Discomfort noticed, but no disruption of normal daily activity |
| Moderate | Discomfort sufficient to reduce or affect normal daily activity |
| Severe | Incapacitating with inability to work or to perform normal daily activity |

Note: Regardless of severity, some events may also meet seriousness criteria. Refer to definition of a serious adverse event (see Section 5.2.2).

### 5.3.4 Assessment of Causality of Adverse Events

Investigators should use their knowledge of the patient, the circumstances surrounding the event, and an evaluation of any potential alternative causes to determine whether an adverse event is considered to be related to the study drug, indicating "yes" or "no" accordingly. The following guidance should be taken into consideration (see also Table 7):

- Temporal relationship of event onset to the initiation of study drug
- Course of the event, with special consideration of the effects of dose reduction, discontinuation of study drug, or reintroduction of study drug (as applicable)
- Known association of the event with the study drug or with similar treatments
- Known association of the event with the disease under study
- Presence of risk factors in the patient or use of concomitant medications known to increase the occurrence of the event
- Presence of non-treatment—related factors that are known to be associated with the occurrence of the event

#### **Table 7 Causal Attribution Guidance**

Is the adverse event suspected to be caused by the study drug on the basis of facts, evidence, science-based rationales, and clinical judgment?

YES There is a plausible temporal relationship between the onset of the adverse event and

- YES There is a plausible temporal relationship between the onset of the adverse event and administration of the study drug, and the adverse event cannot be readily explained by the patient's clinical state, intercurrent illness, or concomitant therapies; and/or the adverse event follows a known pattern of response to the study drug; and/or the adverse event abates or resolves upon discontinuation of the study drug or dose reduction and, if applicable, reappears upon re-challenge.
- NO An adverse event will be considered related, unless it fulfills the criteria specified below. Evidence exists that the adverse event has an etiology other than the study drug (e.g., preexisting medical condition, underlying disease, intercurrent illness, or concomitant medication); and/or the adverse event has no plausible temporal relationship to administration of the study drug (e.g., cancer diagnosed 2 days after first dose of study drug).

For patients receiving combination therapy, causality will be assessed individually for each protocol-mandated therapy.

### 5.3.5 <u>Procedures for Recording Adverse Events</u>

Investigators should use correct medical terminology/concepts when recording adverse events on the Adverse Event eCRF. Avoid colloquialisms and abbreviations.

Only one adverse event term should be recorded in the event field on the Adverse Event eCRF.

### 5.3.5.1 Diagnosis versus Signs and Symptoms

A diagnosis (if known) should be recorded on the Adverse Event eCRF rather than individual signs and symptoms (e.g., record only liver failure or hepatitis rather than jaundice, asterixis, and elevated transaminases). However, if a constellation of signs and/or symptoms cannot be medically characterized as a single diagnosis or syndrome at the time of reporting, each individual event should be recorded on the Adverse Event eCRF. If a diagnosis is subsequently established, all previously reported adverse events based on signs and symptoms should be nullified and replaced by one adverse event report based on the single diagnosis, with a starting date that corresponds to the starting date of the first symptom of the eventual diagnosis.

#### 5.3.5.2 Adverse Events That Are Secondary to Other Events

In general, adverse events that are secondary to other events (e.g., cascade events or clinical sequelae) should be identified by their primary cause, with the exception of severe or serious secondary events. A medically significant secondary adverse event that is separated in time from the initiating event should be recorded as an independent event on the Adverse Event eCRF. For example:

- If vomiting results in mild dehydration with no additional treatment in a healthy adult, only vomiting should be reported on the eCRF.
- If vomiting results in severe dehydration, both events should be reported separately on the eCRF.
- If a severe GI hemorrhage leads to renal failure, both events should be reported separately on the eCRF.
- If dizziness leads to a fall and consequent fracture, all three events should be reported separately on the eCRF.
- If neutropenia is accompanied by an infection, both events should be reported separately on the eCRF.

All adverse events should be recorded separately on the Adverse Event eCRF if it is unclear as to whether the events are associated.

#### 5.3.5.3 Persistent or Recurrent Adverse Events

A persistent adverse event is one that extends continuously, without resolution, between patient evaluation timepoints. Such events should be recorded only once on the Adverse Event eCRF. The initial severity (intensity or grade) of the event will be recorded at the time the event is first reported. If a persistent adverse event becomes

more severe, the most extreme severity should also be recorded on the Adverse Event eCRF. If the event becomes serious, it should be reported to the Sponsor immediately (i.e., no more than 24 hours after learning that the event became serious; see Section 5.4.2 for reporting instructions). The Adverse Event eCRF should be updated by changing the event from "non-serious" to "serious," providing the date that the event became serious and completing all data fields related to serious adverse events.

A recurrent adverse event is one that resolves between patient evaluation timepoints and subsequently recurs. Each recurrence of an adverse event should be recorded as a separate event on the Adverse Event eCRF.

### 5.3.5.4 Abnormal Laboratory Values

Not every laboratory abnormality qualifies as an adverse event. A laboratory test result must be reported as an adverse event if it meets any of the following criteria:

- Is accompanied by clinical symptoms
- Results in a change in study treatment (e.g., dosage modification, treatment interruption, or treatment discontinuation)
- Results in a medical intervention (e.g., potassium supplementation for hypokalemia) or a change in concomitant therapy
- Is clinically significant in the investigator's judgment

It is the investigator's responsibility to review all laboratory findings. Medical and scientific judgment should be exercised in deciding whether an isolated laboratory abnormality should be classified as an adverse event.

If a clinically significant laboratory abnormality is a sign of a disease or syndrome (e.g., alkaline phosphatase and bilirubin  $5 \times ULN$  associated with cholestasis), only the diagnosis (i.e., cholestasis) should be recorded on the Adverse Event eCRF.

If a clinically significant laboratory abnormality is not a sign of a disease or syndrome, the abnormality itself should be recorded on the Adverse Event eCRF, along with a descriptor indicating whether the test result is above or below the normal range (e.g., "elevated potassium," as opposed to "abnormal potassium"). If the laboratory abnormality can be characterized by a precise clinical term per standard definitions, the clinical term should be recorded as the adverse event. For example, an elevated serum potassium level of 7.0 mEq/L should be recorded as "hyperkalemia."

Observations of the same clinically significant laboratory abnormality from visit to visit should only be recorded once on the Adverse Event eCRF (see Section 5.3.5.3 for details on recording persistent adverse events).

### 5.3.5.5 Abnormal Vital Sign Values

Not every vital sign abnormality qualifies as an adverse event. A vital sign result must be reported as an adverse event if it meets any of the following criteria:

- Is accompanied by clinical symptoms
- Results in a change in study treatment (e.g., dosage modification, treatment interruption, or treatment discontinuation)
- Results in a medical intervention or a change in concomitant therapy
- Is clinically significant in the investigator's judgment

It is the investigator's responsibility to review all vital sign findings. Medical and scientific judgment should be exercised in deciding whether an isolated vital sign abnormality should be classified as an adverse event.

If a clinically significant vital sign abnormality is a sign of a disease or syndrome (e.g., high blood pressure), only the diagnosis (i.e., hypertension) should be recorded on the Adverse Event eCRF.

Observations of the same clinically significant vital sign abnormality from visit to visit should only be recorded once on the Adverse Event eCRF (see Section 5.3.5.3 for details on recording persistent adverse events).

#### 5.3.5.6 Abnormal Liver Function Tests

The finding of an elevated ALT or AST ( $> 3 \times$  baseline value) in combination with either an elevated total bilirubin ( $> 2 \times$  ULN) or clinical jaundice in the absence of cholestasis or other causes of hyperbilirubinemia is considered to be an indicator of severe liver injury (as defined by Hy's law). Therefore, investigators must report as an adverse event the occurrence of either of the following:

- Treatment-emergent ALT or AST > 3 × baseline value in combination with total bilirubin > 2 × ULN (of which ≥ 35% is direct bilirubin)
- Treatment-emergent ALT or AST > 3 x baseline value in combination with clinical jaundice

The most appropriate diagnosis or (if a diagnosis cannot be established) the abnormal laboratory values should be recorded on the Adverse Event eCRF (see Section 5.3.5.2) and reported to the Sponsor immediately (i.e., no more than 24 hours after learning of the event), either as a serious adverse event or an adverse event of special interest (see Section 5.4.2).

#### 5.3.5.7 Deaths

All deaths that occur during the protocol-specified adverse event reporting period (see Section 5.3.1), regardless of relationship to study drug, must be recorded on the Adverse Event eCRF and immediately reported to the Sponsor (see Section 5.4.2). This includes death attributed to progression of chronic spontaneous urticaria.

Death should be considered an outcome and not a distinct event. The event or condition that caused or contributed to the fatal outcome should be recorded as the single medical concept on the Adverse Event eCRF. Generally, only one such event should be reported. If the cause of death is unknown and cannot be ascertained at the time of reporting, "unexplained death" should be recorded on the Adverse Event eCRF. If the cause of death later becomes available (e.g., after autopsy), "unexplained death" should be replaced by the established cause of death. The term "sudden death" should not be used unless combined with the presumed cause of death (e.g., "sudden cardiac death").

If the death is attributed to angioedema of CSU, "chronic spontaneous urticaria angioedema" should be recorded on the Adverse Event eCRF.

Deaths that occur after the adverse event reporting period should be reported as described in Section 5.6.

# **5.3.5.8** Preexisting Medical Conditions

A preexisting medical condition is one that is present at the screening visit for this study. Such conditions should be recorded on the General Medical History and Baseline Conditions eCRF.

A preexisting medical condition should be recorded as an adverse event <u>only</u> if the frequency, severity, or character of the condition worsens during the study. When recording such events on the Adverse Event eCRF, it is important to convey the concept that the preexisting condition has changed by including applicable descriptors (e.g., "more frequent headaches").

# 5.3.5.9 Lack of Efficacy or Worsening of Chronic Spontaneous Urticaria

Medical occurrences or symptoms of deterioration that are anticipated as part of CSU should be recorded as an adverse event if judged by the investigator to have unexpectedly worsened in severity or frequency or changed in nature compared to baseline at any time during the study. When recording an unanticipated worsening of CSU on the Adverse Event eCRF, it is important to convey the concept that the condition has changed by including applicable descriptors (e.g., "accelerated CSU").

#### 5.3.5.10 Hospitalization or Prolonged Hospitalization

Any adverse event that results in hospitalization (i.e., inpatient admission to a hospital) or prolonged hospitalization should be documented and reported as a serious adverse event (per the definition of serious adverse event in Section 5.2.2), except as outlined below.

An event that leads to hospitalization under the following circumstances should not be reported as an adverse event or a serious adverse event:

Hospitalization for respite care

- Hospitalization for a preexisting condition, provided that all of the following criteria are met:
  - The hospitalization was planned prior to the study or was scheduled during the study when elective surgery became necessary because of the expected normal progression of the disease
  - The patient has not experienced an adverse event

An event that leads to hospitalization under the following circumstances is not considered to be a serious adverse event, but should be reported as an adverse event instead:

 Hospitalization that was necessary because of patient requirement for outpatient care outside of normal outpatient clinic operating hours. For this scenario, record the underlying medical condition which resulted in hospitalization on the Adverse Event eCRF.

# 5.3.5.11 Adverse Events Associated with an Overdose or Error in Drug Administration

An overdose is the accidental or intentional use of a drug in an amount higher than the dose being studied. An overdose or incorrect administration of study treatment is not itself an adverse event, but it may result in an adverse event. All adverse events associated with an overdose or incorrect administration of study drug should be recorded on the Adverse Event eCRF. If the associated adverse event fulfills seriousness criteria, the event should be reported to the Sponsor immediately (i.e., no more than 24 hours after learning of the event; see Section 5.4.2).

No safety data related to overdosing of GDC-0853 are available.

### 5.3.5.12 Patient-Reported Outcome Data

Adverse event reports will not be derived from PRO data by the Sponsor, and safety analyses will not be performed using PRO data. However, if any PRO responses suggestive of a possible adverse event are identified during site review of the PRO data, the investigator will determine whether the criteria for an adverse event have been met and, if so, will report the event on the Adverse Event eCRF.

# 5.4 IMMEDIATE REPORTING REQUIREMENTS FROM INVESTIGATOR TO SPONSOR

Certain events require immediate reporting to allow the Sponsor to take appropriate measures to address potential new risks in a clinical trial. The investigator must report such events to the Sponsor immediately; under no circumstances should reporting take place more than 24 hours after the investigator learns of the event. The following is a list of events that the investigator must report to the Sponsor within 24 hours after learning of the event, regardless of relationship to study drug:

• Serious adverse events (see Section 5.4.2 for further details)

- Adverse events of special interest (see Section 5.4.2 for further details)
- Pregnancies (see Section 5.4.3 for further details)

The investigator must report new significant follow-up information for these events to the Sponsor immediately (i.e., no more than 24 hours after becoming aware of the information). New significant information includes the following:

- · New signs or symptoms or a change in the diagnosis
- Significant new diagnostic test results
- Change in causality based on new information
- Change in the event's outcome, including recovery
- Additional narrative information on the clinical course of the event

Investigators must also comply with local requirements for reporting serious adverse events to the local health authority and Institutional Review Board or Ethics Committee (IRB/EC).

### 5.4.1 <u>Emergency Medical Contacts</u>

#### **Medical Monitor Contact Information**

Medical Monitor contact information:

Medical Monitor: , M.D.

Telephone Nos.: Mobile:

# 5.4.2 Reporting Requirements for Serious Adverse Events and Adverse Events of Special Interest

# 5.4.2.1 Events That Occur prior to Study Drug Initiation

After informed consent has been obtained but prior to initiation of study drug, only serious adverse events caused by a protocol-mandated intervention should be reported. The Serious Adverse Event/Adverse Event of Special Interest Reporting Form provided to investigators should be completed and submitted to the Sponsor or its designee immediately (i.e., no more than 24 hours after learning of the event), either by faxing or by scanning and emailing the form using the fax number or email address provided to investigators.

# 5.4.2.2 Events That Occur after Study Drug Initiation

After initiation of study drug, serious adverse events and adverse events of special interest will be reported until 4 weeks after the last dose of study drug. Investigators should record all case details that can be gathered immediately (i.e., within 24 hours after learning of the event) on the Adverse Event eCRF and submit the report via the electronic data capture (EDC) system. A report will be generated and sent to Safety Risk Management by the EDC system.

In the event that the EDC system is unavailable, the Serious Adverse Event/Adverse Event of Special Interest Reporting Form provided to investigators should be completed and submitted to the Sponsor or its designee immediately (i.e., no more than 24 hours after learning of the event), either by faxing or by scanning and emailing the form using the fax number or email address provided to investigators. Once the EDC system is available, all information will need to be entered and submitted via the EDC system.

Instructions for reporting serious adverse events that occur > 4 weeks after the last dose of study treatment are provided in Section 5.6.

### 5.4.3 Reporting Requirements for Pregnancies

## 5.4.3.1 Pregnancies in Female Patients

Female patients of childbearing potential will be instructed to immediately inform the investigator if they become pregnant during the study or within 4 weeks after the last dose of study drug. A Clinical Trial Pregnancy Reporting Form should be completed and submitted to the Sponsor or its designee immediately (i.e., no more than 24 hours after learning of the pregnancy), either by faxing or by scanning and emailing the form using the fax number or email address provided to investigators. Pregnancy should not be recorded on the Adverse Event eCRF. The investigator should discontinue study drug and counsel the patient, discussing the risks of the pregnancy and the possible effects on the fetus. Monitoring of the patient should continue until conclusion of the pregnancy. Any serious adverse events associated with the pregnancy (e.g., an event in the fetus, an event in the mother during or after the pregnancy, or a congenital anomaly/birth defect in the child) should be reported on the Adverse Event eCRF. In addition, the investigator will submit a Clinical Trial Pregnancy Reporting Form when updated information on the course and outcome of the pregnancy becomes available.

#### **5.4.3.2** Pregnancies in Female Partners of Male Patients

Male patients will be instructed through the Informed Consent Form to immediately inform the investigator if their partner becomes pregnant during the study or within 4 weeks after the last dose of study drug. A Clinical Trial Pregnancy Reporting Form should be completed and submitted to the Sponsor or its designee immediately (i.e., no more than 24 hours after learning of the pregnancy), either by faxing or by scanning and emailing the form using the fax number or email address provided to investigators. Attempts should be made to collect and report details of the course and outcome of any pregnancy in the partner of a male patient exposed to study drug. When permitted by the site, the pregnant partner would need to sign an Authorization for Use and Disclosure of Pregnancy Health Information to allow for follow-up on her pregnancy. If the authorization has been signed, the investigator should submit a Clinical Trial Pregnancy Reporting Form when updated information on the course and outcome of the pregnancy becomes available. An investigator who is contacted by the male patient or his pregnant partner may provide information on the risks of the pregnancy and the possible effects on the fetus, to support an informed decision in cooperation with the treating physician and/or obstetrician.

Fenebrutinib (GDC-0853)—Genentech, Inc. 82/Protocol GS39684, Version 4

### 5.4.3.3 Congenital Anomalies/Birth Defects and Abortions

Any congenital anomaly/birth defect in a child born to a female patient exposed to study drug or the female partner of a male patient exposed to study drug should be classified as a serious adverse event, recorded on the Adverse Event eCRF, and reported to the Sponsor immediately (i.e., no more than 24 hours after learning of the event; see Section 5.4.2). Any abortion should be reported in the same fashion (as the Sponsor considers abortions to be medically significant).

### 5.5 FOLLOW-UP OF PATIENTS AFTER ADVERSE EVENTS

# 5.5.1 <u>Investigator Follow-Up</u>

The investigator should follow each adverse event until the event has resolved to baseline grade or better, the event is assessed as stable by the investigator, the patient is lost to follow-up, or the patient withdraws consent. Every effort should be made to follow all serious adverse events considered to be related to study drug or trial-related procedures until a final outcome can be reported.

During the study period, resolution of adverse events (with dates) should be documented on the Adverse Event eCRF and in the patient's medical record to facilitate source data verification.

All pregnancies reported during the study should be followed until pregnancy outcome.

### 5.5.2 Sponsor Follow-Up

For serious adverse events, adverse events of special interest, and pregnancies, the Sponsor or a designee may follow up by telephone, fax, email, and/or a monitoring visit to obtain additional case details and outcome information (e.g., from hospital discharge summaries, consultant reports, autopsy reports) in order to perform an independent medical assessment of the reported case.

# 5.6 ADVERSE EVENTS THAT OCCUR AFTER THE ADVERSE EVENT REPORTING PERIOD

The Sponsor should be notified if the investigator becomes aware of any serious adverse event that occurs after the end of the adverse event reporting period (defined as 4 weeks after the last dose of study drug; see Section 5.3.1), if the event is believed to be related to prior study drug treatment. These events should be reported through use of the Adverse Event eCRF. However, if the EDC system is not available, the investigator should report these events directly to the Sponsor or its designee, either by faxing or by scanning and emailing the Serious Adverse Event/Adverse Event of Special Interest Reporting Form using the fax number or email address provided to investigators.

# 5.7 EXPEDITED REPORTING TO HEALTH AUTHORITIES, INVESTIGATORS, INSTITUTIONAL REVIEW BOARDS, AND ETHICS COMMITTEES

The Sponsor will promptly evaluate all serious adverse events and adverse events of special interest against cumulative product experience to identify and expeditiously communicate possible new safety findings to investigators, IRBs, ECs, and applicable health authorities based on applicable legislation.

To determine reporting requirements for single adverse event cases, the Sponsor will assess the expectedness of these events using the following reference document:

Fenebrutinib Investigator's Brochure

The Sponsor will compare the severity of each event and the cumulative event frequency reported for the study with the severity and frequency reported in the applicable reference document.

Reporting requirements will also be based on the investigator's assessment of causality and seriousness, with allowance for upgrading by the Sponsor as needed.

## 6. STATISTICAL CONSIDERATIONS AND ANALYSIS PLAN

The primary and secondary efficacy analyses will be based on a modified intent-to-treat (mITT) approach. All patients who received at least one dose of study drug will be included in the mITT population, with patients grouped according to the treatment assigned at randomization. Safety analyses will be conducted on the safety-evaluable population, defined as all patients who received at least one dose of study drug, with patients grouped according to the actual treatment received.

For each cohort, the final analysis of data from the 8-week, placebo-controlled period will be performed when the following two criteria have been met: 1) All patients in the cohort have either completed the Day 57 visit or discontinued from the placebo-controlled period prematurely and 2) all data from the placebo-controlled period in the cohort are in the database and have been cleaned and verified. Patients and study site personnel will remain blinded to the individual treatment assignment until after the study is completed (i.e., after all patients in both cohorts have either completed the safety follow-up period or discontinued early from the study), the database is locked, and the study analyses are final for both cohorts.

The focus of the trial is estimation and generation of hypotheses to be confirmed in future trials; therefore, Type I error control is not addressed.

#### 6.1 DETERMINATION OF SAMPLE SIZE

# 6.1.1 Cohort 1: Pilot Assessment

The purpose of this cohort is to evaluate the efficacy of fenebrutinib at 200 mg PO BID compared with placebo in improving the UAS7. Point and interval estimates of the

change from baseline of the UAS7 within each treatment group as well as of the difference in change from baseline of the UAS7 between treatment groups will be presented.

The cohort will enroll approximately 45 patients. Patients will be randomized in a 2:1 ratio to receive treatment with either fenebrutinib or placebo. The sample size of approximately 30 patients in the fenebrutinib arm and 15 patients in the placebo arm provides approximately 80% power to detect an 11-point difference in the UAS7 change from baseline at Day 57 between treatment groups under the following assumptions:

- The absolute change from baseline at Day 57 is normally distributed with a standard deviation of 13.
- Two-sided alpha is 0.10.
- Dropout rate at Day 57 is 10%, leading to a 10% loss of information.

## 6.1.2 Cohort 2: Dose-Ranging Assessment

The purpose of this cohort is estimation and hypothesis generation regarding the doseranging effects of fenebrutinib compared with placebo in improving the UAS7. Point and interval estimates of the change from baseline of the UAS7 within each treatment group as well as of the difference in change from baseline of the UAS7 between treatment groups vs placebo will be presented.

The cohort will enroll approximately 120 patients. Patients will be randomly allocated in a 1:1:1:1 ratio to receive treatment with one of three dose levels of fenebrutinib or placebo. The sample size of approximately 30 in each arm provides approximately 90% power to detect an 11-point difference in the UAS7 change from baseline at Day 57 between treatment groups, under the following assumptions:

- The absolute change from baseline at Day 57 is normally distributed with a standard deviation of 13
- Two-sided alpha is 0.10
- Dropout rate at Day 57 is 10%, leading to a 10% loss of information.

The overall sample size may be adjusted depending on the outcome of a planned interim analysis for Cohort 1 (see Section 6.8), which will include an evaluation of these assumptions.

#### 6.2 SUMMARIES OF CONDUCT OF STUDY

The number of patients who enroll, discontinue, or complete the study will be summarized. Reasons for premature study withdrawal will be listed and summarized. Enrollment and major protocol deviations will be listed and evaluated for their potential effects on the interpretation of study results.

#### 6.3 SUMMARIES OF TREATMENT GROUP COMPARABILITY

Baseline demographics, disease characteristics, and exposure to study drug will be summarized by treatment group using descriptive statistics. For categorical endpoints, the descriptive statistics will include counts and proportions. For continuous endpoints, the descriptive statistics will include the number of observations, mean, standard deviation, median, minimum, and maximum.

#### 6.4 EFFICACY ANALYSES

Statistical analysis will be conducted for each cohort separately. Statistical testing will be performed as a two-sided test with a statistical significance level of 0.10. No multiplicity adjustments will be performed to control overall Type I error, and positive tests will be viewed as hypothesis generating rather than confirmatory.

Continuous longitudinal efficacy endpoints will be analyzed using a mixed model for repeated measures (MMRM) and descriptive statistics as appropriate. An unstructured covariance pattern will be specified to model the within-subject errors. Parameters will be estimated with the use of restricted maximum likelihood, and the Kenward-Roger method will be used for calculating the denominator degrees of freedom. The MMRM method assumes that data are missing at random. That is, MMRM assumes that given the statistical model and given the observed values of the endpoint, missing data are independent of the unobserved values (O'Kelly and Ratitch 2014). High correlation between successive observations on a subject allows data from subjects who dropped out to make a contribution to estimation of the effects at the final timepoint.

All MMRM models will include country, treatment group, visit, and visit by treatment group interaction as covariates.

Time-to-event endpoints will be analyzed using a Cox proportional hazards model. Categorical endpoints will be analyzed using an appropriate statistical method, such as Cochran-Mantel-Haenszel test or Fisher's exact test.

Details of all statistical methods will be provided in the Data Analysis Plans (DAP).

## 6.4.1 Primary Efficacy Endpoint

The primary efficacy endpoint is the change from baseline in the UAS7 at Day 57 (Week 8).

The UAS is to be recorded twice daily (i.e., morning and evening) using an eDiary that will be provided to each patient. Scores ranging from 0 (none) to 3 (severe) will be entered for each of the two UAS domains consisting of number of wheals (hives) and intensity of pruritis (itch) resulting in a total possible score of 0 to 6 (see Table 2). The daily UAS is calculated as the average of the morning and evening scores. When either the morning or evening score is missing, the non-missing UAS for that day (morning or evening) will be used as the daily UAS, and when both the morning and evening UAS

are missing, the daily UAS will be deemed missing. The UAS7 is the sum of the daily UAS over the 7 days prior to the timepoint of interest. The baseline UAS7 will be calculated as the sum of daily UAS values over the week (7 days) prior to Day 1.

When one or more daily UAS values is missing, over the week prior to a timepoint of interest, rules for deriving UAS7 will be as follows:

- If a patient has at least 4 completed daily scores on the UAS (both domains) over the 7 days prior to the timepoint of interest, the UAS7 will be defined as the average of the available daily scores, multiplied by 7.
- If a patient has fewer than 4 completed daily scores on the UAS over the 7 days prior to the timepoint of interest, then the UAS7 will be considered missing for that timepoint.

The primary endpoint will be analyzed using a MMRM model as specified in Section 6.4. Additional model covariates will include baseline UAS7 and its interaction with visit. Missing data will be handled by the model under the missing-at-random assumption without need for imputation.

As a sensitivity analysis, an analysis-of-covariance (ANCOVA) model adjusted for country and baseline UAS7 will be fit. Missing Day 57 data will be imputed by last observation carried forward.

### 6.4.2 Secondary Efficacy Endpoints

The secondary efficacy endpoints are as follows:

- Proportion of patients who are well controlled (UAS7 ≤6) at Day 57
- Change from baseline in the UAS7 at Day 29 (Week 4)

These endpoints will be analyzed as specified in Section 6.4.

#### 6.4.3 **Exploratory Efficacy Endpoints**

The exploratory efficacy endpoints include the following:

- Change from baseline in the weekly itch score at Day 29
- Change from baseline in the weekly itch score at Day 57
- Change from baseline in the weekly hives score at Day 57
- Proportion of patients who are well controlled (UAS7 ≤6) at Day 29
- Proportion of patients who achieve complete response (UAS7 = 0) at Day 29
- Proportion of patients who achieve complete response (UAS7 = 0) at Day 57
- Proportion of patients achieving MID in UAS7 at Day 57 (reduction from baseline ≥ 11 points)
- Proportion of patients achieving MID in the weekly itch score at Day 57 (reduction from baseline ≥5 points)

| • | Time to achieving MID in UAS7 (reduction from baseline ≥11 points) |
|---|---|
| Fu | rther details on the analysis of exploratory endpoints will be included in the DAP. |
| 6.5 | SAFETY ANALYSES |
| de: | verse events will be graded according to the adverse event severity grading scale scribed in Section 5.3.3. Summaries of adverse events, serious adverse events, aths, adverse events of special interest, adverse events that lead to discontinuation, CG findings, laboratory test results, and vital sign measurements will be presented. |
| 6.6 | PHARMACOKINETIC ANALYSES |
| Th | e PK endpoints are as follows: |
| • | Plasma concentration data for fenebrutinib will be tabulated and summarized by visits. Descriptive summary statistics will include the arithmetic mean, median, range, SD, and coefficient of variation, as appropriate |
| Ī | |
| pa | e PK analyses will include patients with sufficient data to enable estimation of key rameters (e.g., AUC, t <sub>max</sub> , C <sub>max</sub> , t <sub>1/2</sub> ), with patients grouped according to treatment ceived. |
| | ditional PK analyses will be conducted as appropriate. |
| Λu | anional i ix analyses will be conducted as appropriate. |



#### 6.8 INTERIM ANALYSIS

# 6.8.1 Cohort 1: Planned Interim Analysis

An interim analysis will be performed after approximately 33 patients have completed their 8–week treatment period. The purpose of this analysis is to assess the efficacy of the 200mg fenebrutinib BID daily arm compared with the placebo, to guide internal decision-making around issues such as ungating of Cohort 2, adequacy of sample sizes for safety and/or efficacy analyses in Cohort 2, or to inform further development decisions. Summaries of safety and efficacy data by treatment groups will be prepared and reviewed by Sponsor personnel who do not have direct contact with investigational staff, monitors, and patients. Further details of the interim analysis will be specified in the DAP prior to the conduct of the interim analysis. Access to treatment assignment information will follow the Sponsor's standard procedures.

### 6.8.2 Cohort 2: Optional Interim Analysis

Given the hypothesis-generating nature of this study, the Sponsor may choose to conduct up to two interim efficacy analyses. The decision to conduct an optional interim analysis and the timing of the analysis will be documented in the Sponsor's trial master file prior to the conduct of the interim analysis. The interim analysis will be performed and interpreted by members of the IMC. Access to treatment assignment information will follow the Sponsor's standard procedures.

### 7. DATA COLLECTION AND MANAGEMENT

#### 7.1 DATA QUALITY ASSURANCE

The Sponsor will be responsible for data management of this study, including quality checking of the data. Data entered manually will be collected via EDC through use of eCRFs. Sites will be responsible for data entry into the EDC system. In the event of discrepant data, the Sponsor will request data clarification from the sites, which the sites will resolve electronically in the EDC system.

The Sponsor will produce an EDC Study Specification document that describes the quality checking to be performed on the data. Central laboratory data will be sent directly to the Sponsor, using the Sponsor's standard procedures to handle and process the electronic transfer of these data.

eCRFs and correction documentation will be maintained in the EDC system's audit trail. System backups for data stored by the Sponsor and records retention for the study data will be consistent with the Sponsor's standard procedures.

Fenebrutinib (GDC-0853)—Genentech, Inc. 89/Protocol GS39684. Version 4

PRO data will be collected through the use of an electronic device provided by a vendor. The device is designed for entry of data in a way that is attributable, secure, and accurate, in compliance with U.S. Food and Drug Administration (FDA) regulations for electronic records (21 CFR Part 11). The electronic data are available for view access only via secure access to a web server method. Only identified and trained users may view the data, and their actions become part of the audit trail. The Sponsor will have view access only. System backups for data stored by the Sponsor and records retention for the study data will be consistent with the Sponsor's standard procedures.

#### 7.2 ELECTRONIC CASE REPORT FORMS

eCRFs are to be completed through use of a Sponsor-designated EDC system. Sites will receive training and have access to a manual for appropriate eCRF completion. eCRFs will be submitted electronically to the Sponsor and should be handled in accordance with instructions from the Sponsor.

All eCRFs should be completed by designated, trained site staff. eCRFs should be reviewed and electronically signed and dated by the investigator or a designee.

At the end of the study, the investigator will receive patient data for his or her site in a readable format on a compact disc that must be kept with the study records. Acknowledgement of receipt of the compact disc is required.

#### 7.3 ELECTRONIC PATIENT-REPORTED OUTCOME DATA

Patients will use an electronic device to capture PRO data. The data will be transmitted via wireless or web automatically after entry or uploaded by site staff at the appropriate frequency to a centralized database maintained by the electronic device vendor.

Once the study is complete, the data, audit trail, and trial and system documentation will be archived. The investigator will receive patient data for the site in both human- and machine-readable formats on an archival-quality compact disc that must be kept with the study records as source data. Acknowledgement of receipt of the compact disc is required. In addition, the Sponsor will receive all data in a machine-readable format on a compact disc.

#### 7.4 SOURCE DATA DOCUMENTATION

Study monitors will perform ongoing source data verification to confirm that critical protocol data (i.e., source data) entered into the eCRFs by authorized site personnel are accurate, complete, and verifiable from source documents.

Source documents (paper or electronic) are those in which patient data are recorded and documented for the first time. They include, but are not limited to, hospital records, clinical and office charts, laboratory notes, memoranda, patient-reported outcomes, evaluation checklists, pharmacy dispensing records, recorded data from automated instruments, copies of transcriptions that are certified after verification as being accurate

and complete, microfiche, photographic negatives, microfilm or magnetic media, X-rays, patient files, and records kept at pharmacies, laboratories, and medico-technical departments involved in a clinical trial.

Before study initiation, the types of source documents that are to be generated will be clearly defined in the Trial Monitoring Plan. This includes any protocol data to be entered directly into the eCRFs (i.e., no prior written or electronic record of the data) and considered source data.

Source documents that are required to verify the validity and completeness of data entered into the eCRFs must not be obliterated or destroyed and must be retained per the policy for retention of records described in Section 7.6.

To facilitate source data verification, the investigators and institutions must provide the Sponsor direct access to applicable source documents and reports for trial-related monitoring, Sponsor audits, and IRB/EC review. The study site must also allow inspection by applicable health authorities.

#### 7.5 USE OF COMPUTERIZED SYSTEMS

When clinical observations are entered directly into a study site's computerized medical record system (i.e., in lieu of original hardcopy records), the electronic record can serve as the source document if the system has been validated in accordance with health authority requirements pertaining to computerized systems used in clinical research. An acceptable computerized data collection system allows preservation of the original entry of data. If original data are modified, the system should maintain a viewable audit trail that shows the original data as well as the reason for the change, name of the person making the change, and date of the change.

### 7.6 RETENTION OF RECORDS

Records and documents pertaining to the conduct of this study and the distribution of IMP, including eCRFs, electronic PRO data (if applicable), Informed Consent Forms, laboratory test results, and medication inventory records, must be retained by the Principal Investigator for at least 15 years after completion or discontinuation of the study or for the length of time required by relevant national or local health authorities, whichever is longer. After that period of time, the documents may be destroyed, subject to local regulations.

No records may be disposed of without the written approval of the Sponsor. Written notification should be provided to the Sponsor prior to transferring any records to another party or moving them to another location.

Roche will retain study data for 25 years after the final Clinical Study Report has been completed or for the length of time required by relevant national or local health authorities, whichever is longer.

# 8. <u>ETHICAL CONSIDERATIONS</u>

#### 8.1 COMPLIANCE WITH LAWS AND REGULATIONS

This study will be conducted in full conformance with the ICH E6 guideline for Good Clinical Practice and the principles of the Declaration of Helsinki, or the laws and regulations of the country in which the research is conducted, whichever affords the greater protection to the individual. The study will comply with the requirements of the ICH E2A guideline (Clinical Safety Data Management: Definitions and Standards for Expedited Reporting). Studies conducted in the United States or under a U.S. Investigational New Drug (IND) application will comply with U.S. FDA regulations and applicable local, state, and federal laws. Studies conducted in the European Union or European Economic Area will comply with the E.U. Clinical Trial Directive (2001/20/EC).

#### 8.2 INFORMED CONSENT

The Sponsor's sample Informed Consent Form (and ancillary sample Informed Consent Forms, if applicable) will be provided to each site. If applicable, it will be provided in a certified translation of the local language. The Sponsor or its designee must review and approve any proposed deviations from the Sponsor's sample Informed Consent Forms or any alternate consent forms proposed by the site (collectively, the "Consent Forms") before IRB/EC submission. The final IRB/EC—approved Consent Forms must be provided to the Sponsor for health authority submission purposes according to local requirements.

If applicable, the Informed Consent Form will contain separate Sections for any optional procedures. The investigator or authorized designee will explain to each patient the objectives, methods, and potential risks associated with each optional procedure. Patients will be told that they are free to refuse to participate and may withdraw their consent at any time for any reason. A separate, specific signature will be required to document a patient's agreement to participate in optional procedures. Patients who decline to participate will not provide a separate signature.

The Consent Forms must be signed and dated by the patient or the patient's legally authorized representative before his or her participation in the study. The case history or clinical records for each patient shall document the informed consent process and that written informed consent was obtained prior to participation in the study.

The Consent Forms should be revised whenever there are changes to study procedures or when new information becomes available that may affect the willingness of the patient to participate. The final revised IRB/EC-approved Consent Forms must be provided to the Sponsor for health authority submission purposes.

Patients must be re-consented to the most current version of the Consent Forms (or to a significant new information/findings addendum in accordance with applicable laws and IRB/EC policy) during their participation in the study. For any updated or revised

Consent Forms, the case history or clinical records for each patient shall document the informed consent process and that written informed consent was obtained using the updated/revised Consent Forms for continued participation in the study.

A copy of each signed Consent Form must be provided to the patient or the patient's legally authorized representative. All signed and dated Consent Forms must remain in each patient's study file or in the site file and must be available for verification by study monitors at any time.

#### 8.3 INSTITUTIONAL REVIEW BOARD OR ETHICS COMMITTEE

This protocol, the Informed Consent Forms, any information to be given to the patient, and relevant supporting information must be submitted to the IRB/EC by the Principal Investigator and reviewed and approved by the IRB/EC before the study is initiated. In addition, any patient recruitment materials must be approved by the IRB/EC.

The Principal Investigator is responsible for providing written summaries of the status of the study to the IRB/EC annually or more frequently in accordance with the requirements, policies, and procedures established by the IRB/EC. Investigators are also responsible for promptly informing the IRB/EC of any protocol amendments (see Section 9.6).

In addition to the requirements for reporting all adverse events to the Sponsor, investigators must comply with requirements for reporting serious adverse events to the local health authority and IRB/EC. Investigators may receive written IND safety reports or other safety-related communications from the Sponsor. Investigators are responsible for ensuring that such reports are reviewed and processed in accordance with health authority requirements and the policies and procedures established by their IRB/EC, and archived in the site's study file.

### 8.4 CONFIDENTIALITY

The Sponsor maintains confidentiality standards by coding each patient enrolled in the study through assignment of a unique patient identification number. This means that patient names are not included in data sets that are transmitted to any Sponsor location.

Patient medical information obtained by this study is confidential and may be disclosed to third parties only as permitted by the Informed Consent Form (or separate authorization for use and disclosure of personal health information) signed by the patient, unless permitted or required by law.

Medical information may be given to a patient's personal physician or other appropriate medical personnel responsible for the patient's welfare, for treatment purposes.

Given the complexity and exploratory nature of the analyses, data derived from will generally not be provided to study investigators or patients unless required by law. The aggregate results of any conducted research will

be available in accordance with the effective Sponsor policy on study data publication (see Section 9.5).

Data generated by this study must be available for inspection upon request by representatives of national and local health authorities, Sponsor monitors, representatives, and collaborators, and the IRB/EC for each study site, as appropriate.

#### 8.5 FINANCIAL DISCLOSURE

Investigators will provide the Sponsor with sufficient, accurate financial information in accordance with local regulations to allow the Sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate health authorities. Investigators are responsible for providing information on financial interests during the course of the study and for 1 year after completion of the study (i.e., last patient, last visit).

# 9. <u>STUDY DOCUMENTATION, MONITORING, AND ADMINISTRATION</u>

#### 9.1 STUDY DOCUMENTATION

The investigator must maintain adequate and accurate records to enable the conduct of the study to be fully documented, including, but not limited to, the protocol, protocol amendments, Informed Consent Forms, and documentation of IRB/EC and governmental approval. In addition, at the end of the study, the investigator will receive the patient data, including an audit trail containing a complete record of all changes to data.

#### 9.2 PROTOCOL DEVIATIONS

The investigator should document and explain any protocol deviations. The investigator should promptly report any deviations that might have an impact on patient safety and data integrity to the Sponsor and to the IRB/EC in accordance with established IRB/EC policies and procedures. The Sponsor will review all protocol deviations and assess whether any represent a serious breach of Good Clinical Practice guidelines and require reporting to health authorities. As per the Sponsor's standard operating procedures, prospective requests to deviate from the protocol, including requests to waive protocol eligibility criteria, are not allowed.

#### 9.3 SITE INSPECTIONS

Site visits will be conducted by the Sponsor or an authorized representative for inspection of study data, subjects' medical records, and eCRFs. The investigator will permit national and local health authorities; Sponsor monitors, representatives, and collaborators; and the IRBs/ECs to inspect facilities and records relevant to this study.

#### 9.4 ADMINISTRATIVE STRUCTURE

This trial is sponsored by Genentech. This pilot study will be conducted at study sites experienced in conducting clinical trials in CSU. Data will be recorded via an EDC system from Medidata Solutions (New York, NY) using eCRFs (see Section 7.2). The contract research organization will be responsible for submission to IRB/ECs for approval of the study protocol, patient recruitment, data collection, and reporting. An IxRS will be used to assign patients to treatment groups and to manage ongoing investigational product requests and shipments.

# 9.5 PUBLICATION OF DATA AND PROTECTION OF TRADE SECRETS

Regardless of the outcome of a trial, the Sponsor is dedicated to openly providing information on the trial to healthcare professionals and to the public, both at scientific congresses and in peer-reviewed journals. The Sponsor will comply with all requirements for publication of study results. For more information, refer to the Roche Global Policy on Sharing of Clinical Trials Data at the following Web site:

www.roche.com/roche\_global\_policy\_on\_sharing\_of\_clinical\_study\_information.pdf

The results of this study may be published or presented at scientific congresses. For all clinical trials in patients involving an IMP for which a marketing authorization application has been filed or approved in any country, the Sponsor aims to submit a journal manuscript reporting primary clinical trial results within 6 months after the availability of the respective Clinical Study Report. In addition, for all clinical trials in patients involving an IMP for which a marketing authorization application has been filed or approved in any country, the Sponsor aims to publish results from analyses of additional endpoints and exploratory data that are clinically meaningful and statistically sound.

The investigator must agree to submit all manuscripts or abstracts to the Sponsor prior to submission for publication or presentation. This allows the Sponsor to protect proprietary information and to provide comments based on information from other studies that may not yet be available to the investigator.

In accordance with standard editorial and ethical practice, the Sponsor will generally support publication of multicenter trials only in their entirety and not as individual center data. In this case, a coordinating investigator will be designated by mutual agreement.

Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements. Any formal publication of the study in which contribution of Sponsor personnel exceeded that of conventional monitoring will be considered as a joint publication by the investigator and the appropriate Sponsor personnel.

Any inventions and resulting patents, improvements, and/or know-how originating from the use of data from this study will become and remain the exclusive and unburdened property of the Sponsor, except where agreed otherwise.

#### 9.6 PROTOCOL AMENDMENTS

Any protocol amendments will be prepared by the Sponsor. Protocol amendments will be submitted to the IRB/EC and to regulatory authorities in accordance with local regulatory requirements.

Approval must be obtained from the IRB/EC and regulatory authorities (as locally required) before implementation of any changes, except for changes necessary to eliminate an immediate hazard to patients or changes that involve logistical or administrative aspects only (e.g., change in Medical Monitor or contact information).

### 10. <u>REFERENCES</u>

- Altrichter S, Peter HJ, Pisarevskaja D, et al. IgE mediated autoallergy against thyroid peroxidase–a novel pathomechanism of chronic spontaneous urticaria? PLoS ONE 2011;6:e14794.
- Broides A, Yang W, Conley ME. Genotype/phenotype correlations in X-linked agammaglobulinemia. Clin Immunol 2006;118:195–200.
- Bruton OC. Agammaglobulinemia. Pediatrics 1952;9:722–8.
- Bugatti S, Vitolo B, Caporali R, et al. B cells in rheumatoid arthritis: from pathogenic players to disease biomarkers. Biomed Res Int 2014;2014:681678. doi: 10.1155/2014/681678
- Conley ME, Broides A, Hernandez-Trujillo V, et al. Genetic analysis of patients with defects in early B-cell development. Immunol Rev 2005;203:216–34.
- Di Paolo JA, Huang T, Balazs M, et al. Specific BTK Inhibition suppresses B cell and myeloid cell-mediated arthritis. Nat Chem Biol 2011;7:41–50.
- [FDA] U.S. Food and Drug Administration. Pharmacology review of Incivek (telaprevir). 2011. Available from: http://www.accessdata.fda.gov/drugsatfda\_docs/nda/2011/201917Orig1s000TOC. cfm
- Ferrer M. Immunological events in chronic spontaneous urticaria. Clin Transl Allergy 2015;5:360. doi: 10.1186/s13601-015-0074-7
- Fiebiger E, Maurer D, Holub H, et al. Serum IgG autoantibodies directed against the α chain of FcεRI: a selective marker and pathogenetic factor for a distinct subset of chronic urticaria patients? J Clin Invest 1995;96:2606–12. doi: 10.1172/JCI118325
- Greaves M. Chronic urticaria. J Allergy Clin Immunol 2000;105:664–72.
- Greaves M. Chronic idiopathic urticaria. Curr Opin Allergy Clin Immunol 2003;3:363–8.
- Hata D, Kawakami Y, Inagaki N, et al. Involvement of Bruton's tyrosine kinase in FcεRI-dependent mast cell degranulation and cytokine production. J Exp Med. 1998 Apr 20;187:1235–47.
- Inman WH, Vessey MP, Westerholm B, et al. Thromboembolic disease and the steroidal content of oral contraceptives. A report to the Committee on Safety of Drugs. Br Med J 1970;2:203–9.
- Iyer AS, Morales JL, Huang W, et al. Absence of Tec family kinases interleukin-2 inducible T cell kinase (Itk) and Bruton's tyrosine kinase (Btk) severely impairs FcεRI-dependent mast cell responses. J Bio Chem 2011;286:9503–13. doi: 10.1074/jbc.M110.1656131
- Kaplan AP. Chronic urticaria and angioedema. N Engl J Med 2002;346:175–9.

- Kaveri SV, Maddur MS, Hegde P, et al. Intravenous immunoglobulins in immunodeficiences: more that mere replacement therapy. Clin Exp Immunol 2011;164(Suppl 2):2–5. doi: 10.1111/j.1365-2249.2011.04387.x
- Kay AB, Ying S, Ardelean E, et al. Elevations in vascular markers and eosinophils in chronic spontaneous urticarial weals with low-level persistence in uninvolved skin. Br J Dermatol 2014;171:505–11. doi: 10.1111/bjd.12991
- Kellick KA, Bottorff M, Toth PP, et al. A clinician's guide to statin drug-drug interactions. J Clin Lipidol 2014 May-Jun;8(3 Suppl):S30-46.
- Kern F, Lichtenstein LM. Defective histamine release in chronic urticaria. J Clin Invest 1976;57:1369–77.
- Kozel MA, Sabroe RA. Chronic urticaria, aetiology, management and current and future treatment options. Drugs 2004;64:2515–36.
- Lederman HM, Winkelstein JA. X-linked agammaglobulinema: an analysis of 96 patients. Medicine (Baltimore) 1985;64:145–56.
- Liu L, Di Paolo J, Barbosa J, et al. Antiarthritis effect of a novel Bruton's tyrosine kinase (BTK) inhibitor in rat collagen-induced arthritis and mechanism-based pharmacokinetic/pharmacodynamic modeling: relationships between inhibition of BTK phosphorylation and efficacy. J Pharmacol Exp Ther 2011;338:154–63.
- Luquin E, Kaplan AP, Ferrer M. Increased responsiveness of basophils of patients with chronic urticaria to sera but hypo-responsiveness to other stimuli. Clin Exp Allergy 2005;35:456–60. doi: 10.1111/j.1365-2222.2005.02212.x
- Mathias SD, Crosby RD, Zazzali JL, et al. Evaluating the minimally important difference of the urticaria activity score and other measures of disease activity in patients with chronic idiopathic urticaria. Ann Allergy Asthma Immunol 2012;108:20–4. doi: 10.1016/j.anai.2011.09.008
- Maurer M, Weller K, Bindslev-Jensen C, et al. Unmet clinical needs in chronic spontaneous urticaria. A GA2LEN task force report. Allergy 2011;66:317–30.
- McGirt LY, Vasagar K, Gober LM, et al. Successful treatment of recalcitrant chronic idiopathic urticaria with sulfasalazine. Arch Dermatol 2006;142:1337–42.
- Medicinal Products Act in the version published on 12 December 2005 (Federal Law Gazette [BGBI.]) Part I p. 3394, last amended by Article 2a of the Law of 27 March 2014 (Federal Law Gazette I p. 261).
- Misbah SA, Spickett GP, Ryba PC, et al. Chronic enteroviral meningoencephalitis in agammaglobulinemia: case report and literature review. J Clin Immunol 1992;12:266–70.

- Niiro H, Clark EA. Regulation of B-cell fate by antigen-receptor signals. Nat Rev Immunol 2002;2:945–56.
- O'Kelly M, Ratitch B. Clinical trials with missing data: a guide for practitioners. Chichester, UK: John Wiley & Sons, 2014.
- Powell RJ, Leech SC, Till S, et al. BSACI guideline for the management of chronic urticaria and angioedema. Clin Exp Allergy 2015;45:547–65. doi: 10.1111/cea.12494
- Puri K, Di Paolo J, Gold M. B-cell receptor signaling inhibitors for treatment of autoimmune inflammatory diseases and B-cell malignancies. Int Rev Immunol 2013;32:397–427.
- Reth M, Nielsen P. Signaling circuits in early B-cell development. Adv Immunol 2014;122:129–75. doi: 10.1016/B978-0-12-800267-4.00004-3
- Saini SS. Chronic spontaneuos urticaria: etiology and pathogensis. Immunol Allergy Clin North Am 2014;34:33–52. doi: 10.1016/j.iac.2013.09.012
- Sochorová K, Horvath R, Rozkova D, et al. Impaired toll-like receptor 8-mediated IL-6 and TNF-α production in antigen-presenting cells from patients with X-linked agammaglobulinemia. Blood 2007;109:2553–6.
- Snyder PW, Kazacos EA, Scott-Moncrieff JC, et al. Pathologic features of naturally occurring juvenile polyarteritis in beagle dogs. Vet Pathol 1995;32:337–45.
- Tilles SA. Approach to therapy in chronic urticaria: when Benadryl is not enough. Allergy Asthma Proc 2005;26:9–12.
- Tong LJ, Balakrishnan G, Kochan J. et al. Assessment of autoimmunity in patients with chronic urticaria. J Allergy Clin Immunol 1997;99:461–5.
- Tsukada S, Saffran DC, Rawlings DJ, et al. Deficient expression of a B cell cytoplasmic tyrosine kinase in human X-linked agammaglobulinemia. Cell 1993;72:279–90. doi:10.1016/0092-8674(93)90667-F
- van den Bruele T, Mourad-Baars PE, Claas EC, et al. Campylobacter jejuni bacteremia and Helicobacter pylori in a patient with X-linked agammaglobulinemia. Eur J Clin Microbiol Infect Dis 2010;29:1315–9.
- Vetrie D, Vořechovský I, Sideras P, et al. The gene involved in X-linked agammaglobulinaemia is a member of the src family of protein-tyrosine kinases. Nature 1993;361:226–33. doi:10.1038/361226a0
- Wang B, Sanchez RI, Franklin RB, et al. The involvement of CYP3A4 and CYP2C9 in the metabolism of 17 alpha-ethinylestradiol. Drug Metab Dispos 2004;32:1209–12.
- Whang JA, Chang BY. Bruton's tyrosine kinase inhibitors for the treatment of rheumatoid arthritis. Drug Discov Today 2014;19:1200–4. doi: 10.1016/j.drudis.2014.03.028

- Winkelstein JA, Marino MC, Lederman HM, et al. X-linked agammaglobulinema: report on a United States registry of 201 patients. Medicine (Baltimore) 2006;85:193–202.
- Ying S, Kikuchi Y, Meng Q, et al. TH1/TH2 cytokines and inflammatory cells in skin biopsy specimens from patients with chronic idiopathic urticaria: comparison with the allergen-induced late-phase cutaneous reaction. J Allergy Clin Immunol 2002;109:694–700.
- Zhang H, Cui D, Wang B, et al. Pharmacokinetic drug interactions involving 17alphaethinylestradiol: a new look at an old drug. Clin Pharmacokinet 2007;46:133–57.
- Ziegner UH, Kobayashi RH, Cunningham-Rundles C, et al. Progressive neurodegeneration in patients with primary immunodeficiency disease on IVIG treatment. Clin Immunol 2002;102:19–24.
- Zweiman B, Valenzano M, Atkins PC. Modulation of serum histamine releasing activity in chronic idiopathic urticaria. Immunopharmacology 1998;39:225–34.

# Appendix 1 Schedule of Activities (Cohorts 1 and 2)

| | | | | Tı | eatmen | : Period | | | Safety<br>Follow Up | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Week | Screer | ning a | 0 | 1 | 2 | 4 | 6 c | 8 | 12 | | |
| Day (± days) | -14<br>(-4/+2) | -7 | <b>1</b> b, d | 8 <sup>d</sup> (±1) | 15<br>(±1) | 29 <sup>d</sup> (±2) | 43<br>(±2) | 57 <sup>d,e</sup> (±2) | 85 <sup>d</sup> (±2) | Early<br>Term. | Unscheduled<br>Visit |
| Informed consent | x | - | - | (- ') | (= - / | () | () | (/ | (/ | | |
| Demographic data | х | | | | | | | | | | |
| General medical history and baseline conditions | х | | | | | | | | | | |
| Inclusion/exclusion criteria | х | Х | х | | | | | | | | |
| Randomization | | | Х | | | | | | | | |
| Train patient to complete Urticaria Patient Daily eDiary (including UAS) <sup>f</sup> | х | х | | | | | | | | | |
| Distribute eDiary to patient <sup>g</sup> | х | | | | | | | | | | |
| Urticaria Patient Daily eDiary <sup>g</sup> | | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| Concomitant medications <sup>i</sup> | Х | Х | Х | Х | х | х | х | Х | х | Х | х |
| Adverse events | | | Х | х | Х | Х | Х | Х | Х | Х | Х |
| Vital signs <sup>j</sup> | Х | Х | Х | х | х | х | | Х | Х | Х | <b>X</b> <sup>k</sup> |
| Height | х | | | | | | | | | | |
| Weight | Х | | Х | | | х | | Х | х | Х | X <sup>k</sup> |
| Complete physical examination <sup>1</sup> | Х | | | | | | | | х | | |
| Limited physical examination <sup>m</sup> | | Х | Х | х | Х | Х | | Х | | Х | X <sup>k</sup> |
| ECG <sup>n</sup> | х | | Х | х | | | | | х | Х | X <sup>k</sup> |
| Hepatitis Screening <sup>o</sup> | х | | | | | | | | | | |
| QFT (PPD if QFT not available) | х | | | | | | | | | | |

**Fenebrutinib (GDC-0853)—Genentech, Inc.** 101/Protocol GS39684, Version 4

Appendix 1
Schedule of Activities (Cohorts 1 and 2) (cont.)

| | ledule of Activ | | , | | eatment | | - , | | Safety<br>Follow Up | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Week | Screen | ing <sup>a</sup> | 0 | 1 | 2 | 4 | 6 c | 8 | 12 | | |
| Day (± days) | -14<br>(-4/+2) | -7 | <b>1</b> b, d | 8 <sup>d</sup><br>(±1) | 15<br>(±1) | 29 <sup>d</sup><br>(±2) | 43<br>(±2) | 57 <sup>d,e</sup> (±2) | 85 <sup>d</sup> (±2) | Early<br>Term. | Unscheduled<br>Visit |
| Chest X-ray <sup>p</sup> | х | | | | | | | | | | |
| Fenebrutinib/placebo administration in clinic q, r | | | Х | х | х | Х | | | | | |
| Drug Dispensing | | | Х | | | Х | | | | | |
| Hematologys | х | Х | Х | х | х | х | | Х | Х | Х | <b>X</b> <sup>k</sup> |
| Chemistry <sup>t</sup> | х | Х | Х | х | х | х | | Х | Х | Х | X <sup>k</sup> |
| Fasting Lipid Panel | | | Х | | | х | | Х | х | | |
| Coagulation studies <sup>u</sup> | х | | | | | | | | | Х | X <sup>k</sup> |
| Pregnancy test <sup>v</sup> | х | | Х | х | х | х | | Х | Х | Х | |
| Urinalysis <sup>w</sup> | х | | Х | | | | | Х | Х | Х | |
| FricTest (for patients with dermographism only) | х | | х | | | | | Х | х | х | |
| Plasma PK assessment <sup>y</sup> | | | х | Х | | | | Х | | Х | X <sup>k</sup> |
| Phone call bb | | | | | | | Х | | | | |

# Appendix 1 Schedule of Activities (Cohorts 1 and 2) (cont.)

BID=twice a day; eCRF=electronic case report form; eDiary=electronic diary (patient reported outcomes); HBcAb=hepatitis B core antibody; HBsAb=hepatitis B surface antibody; HBsAb=hepatitis B surface antigen; HCV Ab=hepatitis C antibody; OLE =open-label extension; PD=pharmacodynamic; PK=pharmacokinetic; PPD= purified protein derivative: PPI=proton pump inhibitor: QFT= QuantiFERON-TB Gold®; QTcF=QT interval corrected using Fridericia's formula; TB=tuberculosis; Term.=Termination; UAS=Urticaria Activity Score; UAS7=Urticaria Activity Score over 7 days;

- <sup>a</sup> Laboratory tests prior to randomization and dosing may be performed locally on Day 0, if central laboratory tests are not available due to sampling handling problems, breakage, or lab error.
- b Safety follow-up visit 4 weeks after the last dose of study drug if the patient discontinues the study and/or study treatment (per Sections 4.6.1 and 4.6.2) prior to Day 85 visit or do not enter the OLE.
- c Phone call instead of a clinic visit.
- d Morning clinic visit is required for visits on Days 1, 8, 29, 57, and 85; for other study visits, morning visits are recommended. For mandatory morning visits, the patient should be fasting (overnight, > 8 hours) prior to the first PK blood draw and/or fasting lipid panel.
- e Day 57 visit is the last day of the study treatment period; however, no study drug will be taken at the Day 57 visit. The last dose of blinded study drug will be the p.m. dose on Day 56 or the day before the Day 57 visit if it does not occur on Day 57. If eligible, patients may enroll into the OLE study to receive their first open-label dose of fenebrutinib on Day 1 of Study GS40868 or they will proceed and return for the safety follow-up visit 4 weeks after the last dose of study drug. For patients enrolling into the OLE study, Day 1 of Study GS40868 may be the same day as the Day 57 visit in Study GS39684.
- f Patients should be trained to use the eDiary at Day –14. At Day –7, staff should query patients for any questions they may have concerning the use of the eDiary and ensure patients understand correct usage before randomization.
- <sup>g</sup> Patient is to complete the eDiary twice daily, approximately every 12 hours (a.m./p.m.), every day for the duration of the study. The eDiary includes the UAS7 (itch score, number of hives) and other patient reported outcomes.
- Includes any medication (e.g., prescription drugs, over-the-counter drugs, vaccines, herbal or homeopathic remedies, vitamins, and nutritional or dietary supplements) used by a patient from 12 weeks prior to initiation of study drug until 4 weeks after the last dose of study drug. In addition, at each clinic visit, any use of PPIs, H2 receptor antagonists, and/or other antacids (e.g., Pepto-Bismol®, Rolaids®) should be recorded as concomitant medications, including the date, dose, and time of last administration.
- Includes respiratory rate, pulse rate, temperature, and systolic and diastolic blood pressures while the patient is in a seated position for at least 5 minutes.
- <sup>k</sup> This procedure is optional per the investigator's discretion.

# Appendix 1

# Schedule of Activities (Cohorts 1 and 2) (cont.)

- A complete physical examination should include an evaluation of the head, eyes, ears, nose, and throat and the cardiovascular, dermatological, musculoskeletal, respiratory, gastrointestinal, and neurological systems. Patients should be screened for dermographism. Any abnormality identified at baseline should be recorded on the General Medical History and Baseline Condition eCRF.
- <sup>m</sup> Perform a limited, symptom-directed examination at specified timepoints or as clinically indicated. Record new or worsened clinically significant abnormalities on the Adverse Event eCRF.
- Interpretable digital ECG recording (e.g., without artifacts) will be obtained. The ECG intervals (e.g., PR, QRS, QT, QTcF, and RR) and heart rate from the ECGs will be entered into the eCRF; ECGs for each patient should be obtained from the same machine whenever possible. ECGs can be performed without specific restrictions (e.g., can be any time of day, before or after dosing, fasting or fed) but are to be obtained prior to other procedures scheduled at that same time (e.g., vital sign measurements, blood draws). ECGs must be performed after the patient has been resting in a supine position for at least 10 minutes prior to beginning the ECG recording. Environmental distractions (e.g., television, radio, conversation) should be avoided during the pre-ECG resting period and during ECG recording.
- HBsAg, HBsAb, HBcAb, and HCV Ab.
- Performed only if required by local guidelines to rule out active TB infection.
- <sup>q</sup> On mandatory morning clinic visit days *during the treatment period* (Days 1, *8*, *29*, *and 57*), patients should be instructed that the morning dose of study drug will be taken in the clinic. On other clinic visit days, if the visit occurs in the morning, the patient should be instructed that the morning dose of study drug will be taken in the clinic. The morning dose should be taken after all pre-dose assessments are complete (i.e., ECG, questionnaires, and PK and
- e Patients will take fenebrutinib/placebo BID approximately every 12 hours starting on Day 1 and ending on Day 56 (pm) or the day before (pm) the Day 57 visit if it does not occur on Day 57. One dose (a total of 4 tablets) of fenebrutinib/placebo should be taken with water by mouth BID (a total of 8 tablets each day). The dates and times of the most recent prior meal, last dose of oral study drug (prior to clinic visit), and timing of study drug administration in clinic should be recorded at each clinic visit.
- s Includes WBC count, RBC count, hemoglobin, hematocrit, platelet count, and WBC differential (i.e., neutrophils, eosinophils, basophils, monocytes, lymphocytes, and other cells if present).
- <sup>t</sup> Includes sodium, potassium, chloride, bicarbonate, glucose, BUN or urea, creatinine, total protein, albumin, phosphorus, calcium, total and direct bilirubin, alkaline phosphatase, ALT, AST, uric acid, LDH, CRP, and lipase.
- <sup>u</sup> Includes PT, PTT, INR, and fibrinogen.
- All women of childbearing potential, including those who have had a tubal ligation, will have a serum pregnancy test at screening. Urine pregnancy tests will be performed locally at specified subsequent visits. If a urine pregnancy test result is positive, it must be confirmed by a serum pregnancy test (performed locally).
- w Includes dipstick, including pH, specific gravity, glucose, protein, ketones, blood, and microscopic examination (e.g., sediment, RBCs, WBCs, casts, crystals, epithelial cells, bacteria if present).

# Fenebrutinib (GDC-0853)—Genentech, Inc.

# Appendix 1 Schedule of Activities (Cohorts 1 and 2) (cont.)

y Collect PK samples prior to drug administration, and the patient should be fasting overnight for > 8 hours.

bb Site staff to remind patients to take the study drug and to complete their eDiaries.

# Appendix 2 Childbearing Potential, Pregnancy Testing, and Contraception

#### For Women

All women of childbearing potential (including those who have had a tubal ligation) will have a serum pregnancy test at screening and a urine pregnancy test on Study Day 1 prior to administration of study drug and monthly at appropriate clinic visits. If a urine pregnancy test result is positive, study drug will not be administered until pregnancy is ruled out. The result must be confirmed by a serum pregnancy test (conducted by the local laboratory). Refer to Section 5.4.3 of the protocol for management of a patient with a confirmed pregnancy.

All female patients are considered to be of childbearing potential unless they meet one of the following criteria:

- The patient has been postmenopausal (non-therapy-induced amenorrhea) for at least 12 continuous months with no other identified cause.
- The patient had a surgical bilateral oophorectomy (with or without hysterectomy) more than 6 weeks prior to enrollment.
- The patient had a hysterectomy.

Female patients of reproductive or childbearing potential who are unwilling to use a method of contraception that results in a failure rate of <1 % per year or remain abstinent (refrain from heterosexual intercourse), and refrain from donating eggs during the treatment period and for at least 4 weeks after the last dose of study drug will be excluded from study participation.

Abstinence is acceptable only if it is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Examples of contraceptive methods with a failure rate of < 1% per year include the following:

- Sterilization, bilateral surgical tubal ligation
- Intrauterine device
- Combined oral contraceptive pill <sup>1</sup>
- Contraceptive transdermal patch (estrogen and progestin containing)<sup>1</sup>
- Hormonal vaginal device
- Progestogen-only hormonal contraception associated with inhibition of ovulation
- Implants for contraception
- Injections for contraception (with prolonged release)

# Appendix 2 Childbearing Potential, Pregnancy Testing, and Contraception (cont.)

- Sole sexual partner consisting of surgically sterilized male partner with appropriate
  postsurgical verification of the absence of spermatozoa in the ejaculate. Patients
  may provide verbal confirmation that the partner completed appropriate follow-up
  after vasectomy. Sites are not required to obtain partner medical records.
- Women using estrogen-containing hormonal contraceptives as a method of contraception <u>must</u> also use a barrier such as a male condom in conjunction with the hormonal contraceptives.

#### For Men:

- All men must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:
- With female partners of childbearing potential or pregnant female partners, men
  must remain abstinent or use a condom during the treatment period and for at least
  4 weeks after the last dose of fenebrutinib to avoid exposing the embryo. Men must
  refrain from donating sperm during this same period.

#### For Men and Women

The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, and post-ovulation methods) and withdrawal are not acceptable methods of contraception.

# **General Instructions**

Please answer each question to the best of your ability.

There are no right or wrong answers.

For each question, please choose the response that describes your experience.

Please pay close attention to the timeframe of interest. Some questions ask about the **past 12 hours**, while others ask about the **past 24 hours**.

# Instructions for Counting the Number of Hives and Measuring the Size of the Largest Hive

**Count each hive separately** even if you have more than one hive grouped together with other hives.

Please use the ruler that you have been given to measure the size of your largest hive. If you need help, please have someone else take this measurement for you. Please do not measure a group of hives as one hive.

# **Today's Date**



Please complete this Section <u>every morning</u> throughout the duration of the study. (Please circle only one response.)

 Thinking about the <u>past 12 hours</u>, please record the severity of itch and the number of hives you may have had associated with your skin condition. <u>Please count each hive separately</u> even if you have more than one hive grouped together with other hives.

| Itch (severity) | Hives (number) |
|-----------------|--------------------------|
| 0=none | 0=none |
| 1 = mild | 1=between 1 and 6 hives |
| 2=moderate | 2=between 7 and 12 hives |
| 3=severe | 3=greater than 12 hives |

This next question asks you to estimate the size of your largest hive in centimeters (cm). Please use the ruler that you have been provided with to make this measurement. If your largest hive is located on your back or in a place that is hard to reach, please have someone else take this measurement for you. When measuring the largest hive size, please do not measure a group of hives as one hive.

| Largest Hive (size) |
|---------------------------------------------------------|
| 0=none |
| 1=less than 1.25 centimeter (cm) |
| 2=between 1.25 centimeter (cm) and 2.5 centimeters (cm) |
| 3=greater than 2.5 centimeters (cm) |

# **Today's Date**



Please complete this Section <u>every evening</u> throughout the duration of the study. (Please circle only one response.)

 Thinking about the <u>past 12 hours</u>, please record the severity of itch and the number of hives you may have had associated with your skin condition. <u>Please count each hive separately</u> even if you have more one than one hive grouped together with other hives.

| Itch (severity) | Hives (number) |
|-----------------|--------------------------|
| 0=none | 0=none |
| 1 = mild | 1=between 1 and 6 hives |
| 2=moderate | 2=between 7 and 12 hives |
| 3=severe | 3=greater than 12 hives |

This next question asks you to estimate the size of your largest hive in centimeters (cm). Please use the ruler that you have been provided with to make this measurement. If your largest hive is located on your back or in a place that is hard to reach, please have someone else take this measurement for you. When measuring the largest hive size, please do not measure a group of hives as one hive.

| Largest Hive (size) |
|---------------------------------------------------------|
| 0=none |
| 1=less than 1.25 centimeter (cm) |
| 2=between 1.25 centimeter (cm) and 2.5 centimeters (cm) |
| 3=greater than 2.5 centimeters (cm) |

# **Today's Date**



Please complete this Section twice each day (a.m. and p.m.) throughout the duration of the study (preferably at the same time each day).

# (Please circle only one response.)

- 3. Please rate how much your hives or itch interfered with your sleep during the past 24 hours.
  - 0 No interference
  - 1 Mild, little interference with sleep
  - 2 Moderate, awoke occasionally, some interference with sleep
  - 3 Substantial, woke up often, severe interference with sleep
- 4. Please rate how much your hives or itch interfered with your daily activities during **the past 24 hours**. This could include work, school, sports, hobbies, and activities with friends and family.
  - 0 No interference
  - 1 Mild, little interference with daily activities
  - 2 Moderate, some interference with daily activities
  - 3 Substantial, severe interference with daily activities

These next questions are about your symptoms and how you managed them during the past 24 hours.

| 5. | During the <b>past 24 hours</b> , did you use loratadine or cetirizine in order to |
|---|---|
| | control symptoms of your skin condition such as itch or hives? |
| | 0 = No |

1=Yes

6a. During the **past 24 hours**, did you have any rapid swelling on your face, (especially your eyelids or lips), inside your mouth (including your throat or tongue), or elsewhere on your body? This rapid swelling, also called angioedema, is at a deeper level <u>under</u> your skin than hives.

0 = No (GO TO Question 7) 1 = Yes

6b. If Yes, how did you treat this rapid swelling? (Circle all that apply.)

- 0 Did nothing (GO TO Question 7)
- 1 Took some prescription or non-prescription medication
- 2 Called my doctor, nurse or nurse practitioner
- 3 Went to see my doctor, nurse, or nurse practitioner
- 4 Went to the emergency room at the hospital
- 5 Was hospitalized
- 7. During the **past 24 hours**, did you or someone else call your doctor, nurse or nurse practitioner because of your skin condition?

0 = No 1 = Yes



# Appendix 5 Concomitant Medications (Including Foods and Herbal Products)

| Class | Expected Interaction | Recommendation | Examples of Drugs in this Class <sup>a</sup> |
|---|---|---|---|
| Antacids | Decreased<br>fenebrutinib<br>absorption due to<br>increased gastric pH | Take fenebrutinib 2 hours before or 2 hours after antacid | Pepto-Bismol, Rolaids |
| Moderate<br>or strong<br>CYP3A<br>inhibitors | Increased<br>fenebrutinib plasma<br>concentrations due<br>to inhibition of<br>metabolism | Avoid for 7 days or 5 half-lives (whichever is longer) prior to first dose of study drug and during the treatment period | <ul> <li>Antimicrobials (clarithromycin, erythromycin, itraconazole, ketoconazole, telithromycin, troleandamycin, voriconazole, posaconazole)</li> <li>Antidepressants (nefazodone)</li> <li>Antihypertensive/cardiac (verapamil, diltiazem)</li> <li>Other (grapefruit juice, Seville orange juice, pomegranate, star fruit)</li> </ul> |
| CYP3A<br>inducers | Decreased<br>fenebrutinib plasma<br>concentrations due<br>to increased<br>metabolism | Avoid for 7 days or 5 half-lives (whichever is longer) prior to first dose of study drug and during the treatment period | <ul> <li>Antimicrobials (rifampin, rifapentine, rifabutin)</li> <li>Antidepressants (St. John's wort, hyperforin)</li> <li>Antiepileptics (carbamazepine, phenytoin, phenobarbital, hyperforin)</li> <li>Diabetes (pioglitazone, troglitazone)</li> <li>Other (modafinil, bosentan)</li> </ul> |

# Appendix 5 Concomitant Medications (Including Foods and Herbal Products) (cont.)

| Class | Expected Interaction | Recommendation | Examples of Drugs in this Class <sup>a</sup> |
|---|---|---|---|
| Sensitive<br>and narrow<br>therapeutic<br>window<br>CYP3A<br>substrates | Potential for increased plasma concentrations of CYP3A substrates due to inhibition of metabolism by fenebrutinib | Use with caution and monitor for adverse events related to CYP3A substrates as directed by product labeling; consult with the Medical Monitor as needed | <ul> <li>Antiemetic/prokinetic (aprepitant, cisapride)</li> <li>Antihistamine (astemizole, terfenadine)</li> <li>Antihypertensive/cardiac (dronedarone, eplerenone, felodipine, nisoldipine, quinidine, ticagrelor, vardenafil)</li> <li>Benzodiazepines (alprazolam, diazepam, midazolam)</li> <li>Lipid-lowering (simvastatin [recommended maximum dose: 10 mg/day], lovastatin [recommended maximum dose: 20 mg/day])</li> <li>Migraine (eletriptan, ergotamine)</li> <li>Steroids (budesonide, fluticasone)</li> <li>Other (alfentanil, buspirone, conivaptan, darifenacin, dasatinib, dihydroergotamine, fentanyl, lurasidone, pimozide, quetiapine, sildenafil, tolvaptan, triazolam)</li> </ul> |
| BCRP<br>substrates<br>with a<br>narrow<br>therapeutic<br>index | Potential for increased plasma concentrations of BCRP substrates due to inhibition of transport by fenebrutinib | Use with caution and monitor for adverse events related to BCRP substrates as directed by product labeling; consult with the Medical Monitor as needed | <ul> <li>Antihypertensive (prazosin)</li> <li>Anti-inflammatory (sulfasalazine)</li> <li>Lipid-lowering (rosuvastatin [recommended maximum dose: 10 mg/day], atorvastatin [recommended maximum dose: 20 mg/day]</li> <li>Muscle relaxants (dantrolene)</li> <li>Steroids (estrone-3-sulfate)</li> </ul> |

<sup>&</sup>lt;sup>a</sup> The following list is not comprehensive. Please refer to the following websites for additional information and consult the Medical Monitor if necessary:

U.S. FDA Table of Substrates, Inhibitors, and Inducers (Tables 3-1, 3-2, 3-3, and 5-1) (http://www.fda.gov/Drugs/DevelopmentApprovalProcess/DevelopmentResources/DrugInteract ionsLabeling/ucm093664.htm)

Indiana University Department of Medicine P450 Interaction Table (http://medicine.iupui.edu/clinpharm/ddis/clinical-table)